CLINICAL TRIAL: NCT03602859
Title: A Randomized, Double-blind, Phase 3 Comparison of Platinum-based Therapy With TSR-042 and Niraparib Versus Standard of Care Platinum-based Therapy as First-line Treatment of Stage III or IV Nonmucinous Epithelial Ovarian Cancer
Brief Title: A Comparison of Platinum-based Therapy With TSR-042 and Niraparib Versus Standard of Care (SOC) Platinum-based Therapy as First-line Treatment of Stage III or IV Nonmucinous Epithelial Ovarian Cancer
Acronym: FIRST
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tesaro, Inc. (Industry)
Collaborators: European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 213350; 2024-510605-28 (Registry Identifier: CTIS)
Record Dates: First submitted 2018-06-28; First posted 2018-07-27 (Actual); Results first posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Ovarian Neoplasms; Ovarian, Fallopian Tube and Primary Peritoneal Carcinoma
Keywords: FIRST; FIRST trial; Niraparib; Dostarlimab (TSR-042); Ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — niraparib; dostarlimab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Participants receiving SOC+placebo (Placebo Comparator): Participants in this arm will receive SOC (carboplatin+paclitaxel+/-bevacizumab) in cycle 1 (each cycle is of 21 days) followed by SOC with chemotherapy treatment with dostarlimab placebo from cycles 2 to 6 and maintenance treatment of +/-bevacizumab along with niraparib placebo and dostarlimab placebo
  Interventions: Drug: Standard of care; Drug: Dostarlimab-Placebo; Drug: Niraparib-Placebo
- Participants receiving SOC+niraparib (Active Comparator): Participants in this arm will receive SOC in cycle 1 (each cycle is of 21 days) followed by SOC with chemotherapy treatment dostarlimab placebo from cycles 2 to 6 and maintenance treatment of +/- bevacizumab with niraparib and dostarlimab placebo
  Interventions: Drug: Niraparib; Drug: Standard of care; Drug: Dostarlimab-Placebo
- Participants receiving SOC+dostarlimab+niraparib (Experimental): Participants in this arm will receive SOC in cycle 1 (each cycle is of 21 days) followed by SOC with chemotherapy treatment dostarlimab, and maintenance treatment of +/-bevacizumab with niraparib and dostarlimab
  Interventions: Drug: Niraparib; Drug: Dostarlimab (TSR-042); Drug: Standard of care

INTERVENTIONS:
Drug: Niraparib — Participants will receive oral capsules of niraparib as a unit dosage strength of 100 milligrams (mg)
  Other Names: ZEJULA
  Arms: Participants receiving SOC+dostarlimab+niraparib; Participants receiving SOC+niraparib
Drug: Dostarlimab (TSR-042) — Participants will receive 500 mg dostarlimab on day 1 every 3 weeks from cycle 2 to 6 followed by 1000mg of dostarlimab on day 1 every 6 weeks to continue up to 3 years in the absence of disease progression, unacceptable toxicity, participant withdrawal, or investigator decision
  Arms: Participants receiving SOC+dostarlimab+niraparib
Drug: Standard of care — Participants will receive SOC that includes paclitaxel 175 milligrams per square meter (mg/m^2) on day 1 every 21 days + carboplatin area under the curve (AUC) of 5 to 6 milligrams per milliliter per minute (mg/mL/min) on day 1 every 21 days +/- bevacizumab 7.5 milligrams per kilograms (mg/kg) every 21 days or 15 mg/kg every 21 days for a total of 15 months.
Drug: Dostarlimab-Placebo — Participants will receive 500 mg of dostarlimab-placebo on day 1 every 3 weeks from cycle 2 to 6 followed by 1000 mg of dostarlimab-placebo on day 1 every 6 weeks to continue up to 3 years in the absence of disease progression, unacceptable toxicity, participant withdrawal, or investigator decision
  Arms: Participants receiving SOC+niraparib; Participants receiving SOC+placebo
Drug: Niraparib-Placebo — Participants will receive oral capsules of niraparib-placebo as a unit dosage strength of 100 mg.
  Arms: Participants receiving SOC+placebo

SUMMARY:
Ovarian cancer is a heterogeneous disease, characterized by complex molecular and genetic changes. The high expression of vascular endothelial growth factor (VEGF) receptor, programmed death receptor ligands 1 (PD-L1) expression, and deoxyribonucleic acid (DNA) damage in ovarian tumors provide several targets for treatment and maintenance of disease response. Given the unmet medical need of participants with advanced or metastatic ovarian cancer, this study design will enable investigators to provide participants with current SOC for ovarian cancer for the duration of the study. This is a global, multicenter, randomized, double-blind, controlled Phase 3 study that will primarily compare the progression-free survival (PFS) for participants receiving dostarlimab with SOC chemotherapy +/- bevacizumab followed by niraparib and dostarlimab maintenance +/- bevacizumab versus participants receiving SOC with chemotherapy followed by niraparib maintenance. This comparison will be investigated in participants of newly diagnosed stage III or IV advanced non-mucinous epithelial ovarian cancer participants and also to compare PFS of all participants with Stage III or IV high-grade non-mucinous epithelial ovarian cancer treated with platinum-based combination therapy, dostarlimab (TSR-042), and niraparib to SOC platinum-based combination therapy. The currently recommended SOC therapy for the first line treatment of Stage III or IV ovarian cancer is the combination of paclitaxel and carboplatin, with or without concurrent and maintenance bevacizumab. Participants will receive SOC during the chemotherapy Run-In period (cycle 1) before randomization to study treatment (cycle 2). Concurrent bevacizumab use must be determined prior to randomization at cycle 2.

ELIGIBILITY:
Inclusion criteria:

* Participants must be female, >=18 years of age, able to understand the study procedures, and agree to participate in the study by providing written informed consent.
* Participants with a histologically confirmed diagnosis of high-grade nonmucinous epithelial ovarian (serous, endometrioid, clear cell, carcinosarcoma, and mixed pathologies), fallopian tube, or peritoneal cancer that is Stage III or IV according to the International Federation of Gynecology and Obstetrics (FIGO) or tumor, node and metastasis staging criteria.
* All participants with Stage IV disease are eligible. This includes those with inoperable disease, those who undergo primary debulking surgery (PDS) (R0 or macroscopic disease), or those for whom neoadjuvant chemotherapy (NACT) is planned.
* Participants with Stage III are eligible if they meet protocol defined criteria.
* Participants must provide a blood sample for circulating tumor deoxyribonucleic acid (ctDNA) homologous recombinant repair (HRR) testing at pre-screening or screening.
* Participant must provide a minimum of 1 formalin-fixed paraffin embedded (FFPE) block slide at pre-screening or screening for PD-L1, homologous recombinant deficiency (HRD) testing.
* Participants of childbearing potential must have a negative serum or urine pregnancy test (beta human chorionic gonadotropin) within 3 days prior to receiving the first dose of study treatment.
* Participants must be postmenopausal, free from menses for >1 year, surgically sterilized, or willing to use highly effective contraception to prevent pregnancy or must agree to abstain from activities that could result in pregnancy throughout the study, starting with enrollment through 180 days after the last dose of study treatment.
* Participants must have adequate organ function: Absolute neutrophil count (ANC) >=1500/micro liter (μL;) Platelet count >=100000/μL; Hemoglobin >=9 grams per deciliter (g/dL); Serum creatinine <=1.5 × upper limit of normal (ULN) or calculated creatinine clearance >=60 milliliters per minute (mL/min) using the Cockcroft-Gault equation; total bilirubin <=1.5 × ULN or direct bilirubin <=1.5 × ULN; AST and ALT <=2.5 × ULN unless liver metastases are present, in which case they must be <=5 × ULN.
* Participants must have an ECOG score of 0 or 1.
* Participants must have normal blood pressure (BP) or adequately treated and controlled hypertension (systolic BP <=140 millimeters of mercury (mmHg) and/or diastolic BP <=90 mmHg).
* Participants must agree to complete health related quality of life (HRQoL) questionnaires throughout the study.
* Participants must be able to take oral medication.

Exclusion Criteria:

* Participant has mucinous, germ cell, transitional cell, or undifferentiated tumor.
* Participant has low-grade or Grade 1 epithelial ovarian cancer.
* Participant has not adequately recovered from prior major surgery.
* Participant is pregnant or is expecting to conceive children while receiving study drug or for up to 180 days after the last dose of study drug. Participant is breastfeeding or is expecting to breastfeed within 30 days of receiving the final dose of study drug (women should not breastfeed or store breastmilk for use, during niraparib treatment and for 30 days after receiving the final dose of study treatment).
* Participant has known active central nervous system metastases, carcinomatous meningitis, or both.
* Participant has clinically significant cardiovascular disease.
* Participant has a bowel obstruction by clinical symptoms or computed tomography (CT) scan, subocclusive mesenteric disease, abdominal or gastrointestinal fistula, gastrointestinal perforation, or intra-abdominal abscess.
* Participant has any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML).
* Participant has been diagnosed and/or treated with any therapy for invasive cancer <5 years from study enrollment, completed adjuvant chemotherapy and/or targeted therapy (example, trastuzumab) less than 3 years from enrollment, or completed adjuvant hormonal therapy less than 4 weeks from enrollment.
* Participants with definitively treated non-invasive malignancies such as cervical carcinoma in situ, ductal carcinoma in situ, Grade 1 or 2, Stage I endometrial cancer, or non-melanomatous skin cancer are allowed.
* Participant is at increased bleeding risk due to concurrent conditions (example, major injuries or major surgery within the past 28 days prior to start of study treatment and/or history of hemorrhagic stroke, transient ischemic attack, subarachnoid hemorrhage, or clinically significant hemorrhage within the past 3 months).
* Participant is immunocompromised.
* Participant has known active hepatitis B (example, hepatitis B surface antigen reactive) or hepatitis C (example, hepatitis C virus ribonucleic acid [qualitative] is detected).
* Participant is considered a poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or uncontrolled infection.
* Participant has had investigational therapy administered within 4 weeks or within a time interval less than at least 5 half-lives of the investigational agent, whichever is longer, prior to the first scheduled day of dosing in this study.
* Participant has received a live vaccine within 14 days of planned start of study therapy. Seasonal influenza vaccines that do not contain live viruses are allowed.
* Participant has a known contraindication or uncontrolled hypersensitivity to the components of paclitaxel, carboplatin, niraparib, bevacizumab, dostarlimab, or their excipients.
* Prior treatment for high-grade nonmucinous epithelial ovarian, fallopian tube, or peritoneal cancer (immunotherapy, anti-cancer therapy, radiation therapy).
* Participant has an active autoimmune disease that has required systemic treatment in the past 2 years. Replacement therapy is not considered a form of systemic therapy (example, thyroid hormone or insulin).
* Participant has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of systemic immunosuppressive therapy within 7 days prior to the first dose of study treatment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1400 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2029-04-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (160):
- United States (58):
  - GSK Investigational Site, Anchorage, Alaska
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Tucson, Arizona
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Newport Beach, California
  - GSK Investigational Site, Farmington, Connecticut
  - GSK Investigational Site, Hartford, Connecticut
  - GSK Investigational Site, Gainesville, Florida
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Geneva, Illinois
  - GSK Investigational Site, Warrenville, Illinois
  - GSK Investigational Site, Zion, Illinois
  - GSK Investigational Site, Covington, Louisiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Shreveport, Louisiana
  - GSK Investigational Site, Scarborough, Maine
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Silver Spring, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Springfield, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Billings, Montana
  - GSK Investigational Site, Neptune City, New Jersey
  - GSK Investigational Site, Teaneck, New Jersey
  - GSK Investigational Site, Hawthorne, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Stony Brook, New York
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Canton, Ohio
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Eugene, Oregon
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Paoli, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Pittsburgh, Pennsylvania
  - GSK Investigational Site, Willow Grove, Pennsylvania
  - GSK Investigational Site, Wynnewood, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Sioux Falls, South Dakota
  - GSK Investigational Site, Knoxville, Tennessee
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, The Woodlands, Texas
  - GSK Investigational Site, Tyler, Texas
  - GSK Investigational Site, Ogden, Utah
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Norfolk, Virginia
  - GSK Investigational Site, Kennewick, Washington
  - GSK Investigational Site, Seattle, Washington
- GSK Investigational Site, Minsk, Belarus
- Belgium (2):
  - GSK Investigational Site, Brasschaat
  - GSK Investigational Site, Bruges
- Canada (6):
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
  - GSK Investigational Site, Windsor
- GSK Investigational Site, Prague, Czechia
- Denmark (3):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Herlev
  - GSK Investigational Site, Roskilde
- Finland (4):
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- France (31):
  - GSK Investigational Site, Angers
  - GSK Investigational Site, Avignon
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Bordeaux
  - GSK Investigational Site, Bron
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Cholet
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Le Mans
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nancy
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Nîmes
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pierre-Bénite
  - GSK Investigational Site, Plerin-sur-mer
  - GSK Investigational Site, Poitiers
  - GSK Investigational Site, Reims
  - GSK Investigational Site, Rennes
  - GSK Investigational Site, Saint-Cloud
  - GSK Investigational Site, Saint-Priest-en-Jarez
  - GSK Investigational Site, Strasbourg
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
  - GSK Investigational Site, Villejuif
- Germany (6):
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Hamburg
  - GSK Investigational Site, Kiel
  - GSK Investigational Site, Münster
  - GSK Investigational Site, Ravensburg
  - GSK Investigational Site, Wolfsburg
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Haidari - Athens
  - GSK Investigational Site, Marousi
- Israel (5):
  - GSK Investigational Site, Beersheba
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Rehovot
- Italy (5):
  - GSK Investigational Site, Bologna
  - GSK Investigational Site, Faenza
  - GSK Investigational Site, Lugo RA
  - GSK Investigational Site, Meldola FC
  - GSK Investigational Site, Napoli
- Netherlands (6):
  - GSK Investigational Site, Amsterdam
  - GSK Investigational Site, Groningen
  - GSK Investigational Site, Maastricht
  - GSK Investigational Site, Nijmegen
  - GSK Investigational Site, Rotterdam
  - GSK Investigational Site, Utrecht
- Norway (3):
  - GSK Investigational Site, Kristiansand
  - GSK Investigational Site, Oslo
  - GSK Investigational Site, Tromsø
- Poland (3):
  - GSK Investigational Site, Olsztyn
  - GSK Investigational Site, Szczecin
  - GSK Investigational Site, Warsaw
- Romania (5):
  - GSK Investigational Site, Bucharest
  - GSK Investigational Site, Cluj-Napoca
  - GSK Investigational Site, Constanța
  - GSK Investigational Site, Craiova
  - GSK Investigational Site, Timișoara
- Spain (10):
  - GSK Investigational Site, Ávila
  - GSK Investigational Site, Badalona
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Jaén
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Toledo
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Zaragoza
- Ukraine (3):
  - GSK Investigational Site, Chernihiv
  - GSK Investigational Site, Kharkiv
  - GSK Investigational Site, Lviv
- United Kingdom (5):
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Metropolitan Borough of Wirral
  - GSK Investigational Site, Portsmouth
  - GSK Investigational Site, Sutton
  - GSK Investigational Site, Truro

IPD SHARING:
Plan to Share IPD: No
GSK will assess requests from qualified researchers for anonymized individual patient-level data and related study documents. Data sharing is subject to certain criteria, conditions, and exceptions. For further information, refer to https://www.gsk-studyregister.com/About_GSK_Patient_Level_Data_Sharing_Final_13July2023.pdf.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results presented are based on primary completion date. Safety data collection is still ongoing, and additional results will be provided within a year of study completion.
Groups:
- All Enrolled Participants: Eligible participants with ovarian cancer received standard of care (SOC) chemotherapy as combination of 175 milligram (mg)/meter^2(m^2) Paclitaxel, area under the curve (AUC) of 5 to 6 mg/millilitre (mL)/minute Carboplatin and optional 7.5 mg/kilogram (kg) or 15 mg/kg Bevacizumab as intravenous (IV) infusion on Day 1 of Cycle 1 in Chemotherapy Run-In Period.
- Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib Pbo+Dostarlimab Pbo +/-Bev (Arm1): Participants received intravenous (IV) infusion of Carboplatin+Paclitaxel along with Dostarlimab placebo (Pbo) on Day 1 of each 21-day (Q21D) cycle for up to 5 cycles starting with Cycle 2, with optional Bevacizumab (Bev) as part of Chemotherapy.
  Following this, as part of Maintenance, participants received IV infusion of 1000 mg Dostarlimab Placebo on Day 1 every 6 weeks in combination with/without 7.5 mg/kg or 15 mg/kg Bevacizumab Q21D along with oral niraparib placebo Q21D until disease progression, unacceptable toxicity, participant withdrawal, or Investigator decision
- Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2): Participants received intravenous (IV) infusion of Carboplatin+Paclitaxel along with Dostarlimab placebo on Day 1 of each 21-day (Q21D) cycle for up to 5 cycles, starting with Cycle 2 with optional Bevacizumab as part of Chemotherapy.
  Following this, as part of Maintenance, participants received IV infusion of 1000 mg Dostarlimab Placebo on Day 1 every 6 weeks in combination with/without 7.5 mg/kg or 15 mg/kg Bevacizumab Q21D along with oral niraparib Q21D until disease progression, unacceptable toxicity, participant withdrawal, or Investigator decision
- Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3): Participants received intravenous (IV) infusion of Carboplatin + Paclitaxel along with Dostarlimab on Day 1 of each 21-day (Q21D) cycle for up to 5 cycles, starting with Cycle 2 with optional Bevacizumab as part of Chemotherapy.
  Following this, as part of Maintenance, participants received IV infusion of 1000 mg Dostarlimab on Day 1 every 6 weeks in combination with/without 7.5 mg/kg or 15 mg/kg Bevacizumab Q21D along with oral niraparib Q21D until disease progression, unacceptable toxicity, participant withdrawal, or Investigator decision
Period: Chemotherapy Run-In Period (Cycle 1)
Arm/Group | All Enrolled Participants | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib Pbo+Dostarlimab Pbo +/-Bev (Arm1) | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Started | 1400 | 0 | 0 | 0
Completed | 1321 | 0 | 0 | 0
Not Completed | 79 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 0 | 0 | 0
Not completed — Disease Progression per Clinical Criteria by Investigator | 2 | 0 | 0 | 0
Not completed — Risk to Patient | 3 | 0 | 0 | 0
Not completed — Severe Noncompliance to Protocol | 6 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 10 | 0 | 0 | 0
Not completed — Death | 10 | 0 | 0 | 0
Not completed — Other | 27 | 0 | 0 | 0
Not completed — Missing | 1 | 0 | 0 | 0
Not completed — Randomized but not treated | 10 | 0 | 0 | 0
Period: Chemo Treatment Period (Cycle 2 to 6)
Arm/Group | All Enrolled Participants | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib Pbo+Dostarlimab Pbo +/-Bev (Arm1) | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Started (Safety Population included all randomized participants who received at least 1 dose of study treatment after randomization.) | 0 | 159 | 417 | 745
ITT Population (Included all randomized participants.) | 0 | 193 | 385 | 753
Completed | 0 | 129 | 371 | 645
Not Completed | 0 | 30 | 46 | 100
Not completed — Investigator decision | 0 | 1 | 5 | 3
Not completed — Adverse Event | 0 | 7 | 11 | 25
Not completed — Progression/clinical progression | 0 | 7 | 14 | 15
Not completed — Risk to Patient | 0 | 2 | 1 | 5
Not completed — Severe Noncompliance to Protocol | 0 | 2 | 2 | 8
Not completed — Withdrawal by Subject | 0 | 9 | 11 | 29
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Death | 0 | 1 | 1 | 5
Not completed — Other | 0 | 1 | 1 | 9
Period: Maintenance Period (Cycle 7 to 89)
Arm/Group | All Enrolled Participants | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib Pbo+Dostarlimab Pbo +/-Bev (Arm1) | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Started | 0 | 129 | 371 | 645
Completed | 0 | 5 | 41 | 77
Not Completed | 0 | 124 | 330 | 568
Not completed — Ongoing | 0 | 3 | 23 | 42
Not completed — Adverse Event | 0 | 6 | 24 | 91
Not completed — Thrombocytopenia Platelet Count not Returned to >=100000 cells/uL w/in | 0 | 0 | 1 | 2
Not completed — Progression/clinical progression | 0 | 83 | 251 | 356
Not completed — Risk to Patient | 0 | 2 | 1 | 2
Not completed — Severe Noncompliance to Protocol | 0 | 3 | 3 | 5
Not completed — Withdrawal by Subject | 0 | 7 | 22 | 48
Not completed — Lost to Follow-up | 0 | 0 | 2 | 2
Not completed — Death | 0 | 0 | 1 | 7
Not completed — Unblinded due to being randomized to Arm 1 | 0 | 18 | 0 | 0
Not completed — Investigator decision | 0 | 0 | 0 | 1
Not completed — Other | 0 | 2 | 2 | 12

BASELINE CHARACTERISTICS:
Population: All eligible enrolled participants received SOC during the Cycle 1 Chemotherapy Run-In Period before randomization.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1400
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 62.0 (10.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1400
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1245
  Black or African American | 30
  Asian | 29
  American Indian or Alaska Native | 8
  Unknown | 80
  Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Progression Free Survival (PFS) is defined as the time from the date of randomization to the date of first documented progressive disease (PD) or death due to any cause, whichever occurs first by the Investigator assessment according to Response Evaluation Criteria in Solid Tumors Criteria (RECIST) version 1.1. Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 millimeter (mm).
Time Frame: Up to approximately 316 weeks
Population: The Intent-to-Treat (ITT) population included all randomized participants. As pre-specified in the protocol, the comparison of data was performed only between Arm 2 and Arm 3.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2): Participants received intravenous (IV) infusion of Carboplatin + Paclitaxel along with Dostarlimab placebo on Day 1 of each 21-day (Q21D) cycle for up to 5 cycles, starting with Cycle 2 with optional Bevacizumab as part of Chemotherapy.
  Following this, as part of Maintenance, participants received IV infusion of 1000 mg Dostarlimab Placebo on Day 1 every 6 weeks in combination with/without 7.5 mg/kg or 15 mg/kg Bevacizumab Q21D along with oral niraparib Q21D until disease progression, unacceptable toxicity, participant withdrawal, or Investigator decision
- Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3): Participants received intravenous (IV) infusion of Carboplatin+Paclitaxel along with Dostarlimab on Day 1 of each 21-day (Q21D) cycle for up to 5 cycles, starting with Cycle 2 with optional Bevacizumab as part of Chemotherapy.
  Following this, as part of Maintenance, participants received IV infusion of 1000 mg Dostarlimab on Day 1 every 6 weeks in combination with/without 7.5 mg/kg or 15 mg/kg Bevacizumab Q21D along with oral niraparib Q21D until disease progression, unacceptable toxicity, participant withdrawal, or Investigator decision
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 385 | 753
Months | 19.19 [16.59 to 20.99] | 20.63 [19.22 to 22.77]
Statistical Analysis 1: Comparison: Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) vs Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3); Test type: Other; p = 0.0351, Stratified log-rank test; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.73 to 0.99] — Hazard ratio and p-value from the stratified Cox proportional hazards model and log-rank test (2-sided) are adjusted for the randomization stratification factors: concurrent bevacizumab use and homologous recombinant repair (HRR) mutation status

2. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) is defined as the time from the date of randomization to the date of death by any cause.
Time Frame: Up to approximately 316 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 385 | 753
Months | 45.37 [40.28 to 52.21] | 44.39 [41.17 to 47.54]

3. Secondary Outcome: PFS Determined by Blinded Independent Central Review (BICR) Per RECIST v1.1 Criteria
Description: Progression Free Survival (PFS) is defined as the time from the date of randomization to the date of first documented progressive disease (PD) or death due to any cause, whichever occurs first determined by the BICR according to RECIST version 1.1. Progressive Disease was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5mm.
Time Frame: Up to approximately 316 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 385 | 753
Months | 23.56 [20.14 to 27.40] | 25.89 [23.36 to 32.49]

4. Secondary Outcome: Time to First Subsequent Therapy (TFST)
Description: Time to First Subsequent Therapy (TFST) is defined as the time from randomization until the start date of the first subsequent anticancer therapy or death by any cause, whichever occurs first. First subsequent anticancer therapy is defined as the earliest anticancer therapy on the follow-up anticancer therapy form.
Time Frame: Up to approximately 316 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 385 | 753
Months | 20.93 [17.58 to 22.67] | 20.86 [19.15 to 23.92]

5. Secondary Outcome: Time to Second Subsequent Therapy (TSST)
Description: Time to Second Subsequent Therapy (TSST) is defined as the time from the date of randomization to the start date of the second subsequent anticancer therapy or death of any cause, whichever occurs first. Second subsequent anticancer therapy is defined as an anticancer therapy with a start date after the first subsequent anticancer therapy and a recorded PD on first subsequent anticancer therapy, as captured on the follow-up anticancer therapy eCRF form.
Time Frame: Up to approximately 316 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 385 | 753
Months | 33.97 [30.06 to 37.49] | 35.32 [32.46 to 38.31]

6. Secondary Outcome: Time to Second Progression (PFS2)
Description: PFS2 is defined as the time from the date of randomization to the date of first Progressive Disease per Investigator's assessment after initiation of subsequent anticancer therapy or death due to any cause, whichever occurs first.
  Progressive Disease is defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 millimeter (mm).
Time Frame: Up to approximately 316 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 385 | 753
Months | 31.84 [28.65 to 35.09] | 32.69 [30.42 to 35.38]

7. Secondary Outcome: Objective Response Rate (ORR)
Description: Objective Response Rate (ORR) is defined as the percentage of participants with measurable disease at baseline achieving a best overall response (BOR) of complete response (CR) or partial response (PR) by Investigator assessment per RECIST v1.1 criteria for participants with measurable disease at baseline. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR is defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm.
Time Frame: Up to approximately 316 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 385 | 753
Percentage of participants | 88 [83.7 to 91.6] | 88.4 [85.5 to 90.9]

8. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from the first documented response (complete response (CR) OR partial response (PR) ) to the first documented disease progression per Investigator assessed RECIST v1.1 or death by any cause in participants with measurable disease at baseline who responded to treatment. PR was defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR was defined as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PD was defined as at least a 20% increase in the sum of the diameters of target lesions, taking as a reference, the smallest sum of diameters recorded since the treatment started (e.g. percent change from nadir, where nadir is defined as the smallest sum of diameters recorded since treatment start). In addition, the sum must have an absolute increase from nadir of 5 mm.
Time Frame: Up to approximately 316 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 250 | 496
Months | 16.07 [13.86 to 18.40] | 18.27 [16.36 to 20.53]

9. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease Control Rate (DCR) is defined as the percentage of participants with measurable disease at baseline achieving a best overall response (BOR) of complete response (CR), partial response (PR) or stable disease (SD) by Investigator assessment per RECIST v1.1 criteria for participants with measurable disease at baseline. PR is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. CR is defined as the disappearance of all target lesions. SD defined as any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<)10 mm.
Time Frame: Up to approximately 316 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 385 | 753
Percentage of participants | 93.7 [90.2 to 96.2] | 93.6 [91.2 to 95.5]

10. Secondary Outcome: Number of Participants With Treatment Emergent Positive Antidrug Antibodies (ADAs) of Dostarlimab
Description: Serum samples were collected for the analysis of Anti-drug antibody (ADAs) of dostarlimab.
Time Frame: Up to approximately 316 weeks
Population: Anti-drug antibody (ADA) population included all participants from Arm 3 only who received at least one dose of dostarlimab and who had at least 1 ADA sample with an assay result.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 745
Participants | 17

11. Secondary Outcome: Change From Baseline (CFB) for the Visual Analogue Score (VAS) and Health Utility Index (HUI) of European Quality of Life 5-Dimension 5-Level Scale (EQ-5D-5L) Questionnaire
Description: EQ-5D-5L is a standardized, participant-rated health outcomes questionnaire covering five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. For each of dimensions, participant self-assigned score: 1 (no problems); 2 (slight problems); 3 (moderate problems); 4 (severe problems); 5 (extreme problems). VAS is collected separately and recorded from 0 (Worst imaginable health state) to 100 (Best imaginable health state). HUI values summarize how good or bad each health state is on a scale of 1 (full health) to 0 (worse health/dead). High HUI value indicates a good HRQoL. Baseline is defined as the latest, non-missing collected value, excluding end of treatment, safety follow-up, long term follow-up visits records and unscheduled visits after end of treatment (EOT).
Time Frame: Day1 of Chemo Cycles 2(baseline), 4&6; Day1 of Maintenance Cycles 1,2,3,6,9,12,15,17,23,29,35,41,47,53,59,65,71,77,83,89; EOT visit up to a maximum of 63 months; LTFU visit up to a maximum of 69 months(including SFU visit up to a maximum of 61 months)
Population: ITT Population.Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified timepoints. As pre-specified in the protocol, the comparison of data was performed only between Arm 2 and Arm 3.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 330 | 655
Scores on a scale
  EQ-VAS, Cycle 4 Chemotherapy: number analyzed (Participants) | 277 | 534
  EQ-VAS, Cycle 4 Chemotherapy | 1.2 (18.33) | 0.1 (18.00)
  EQ-VAS, Cycle 6 Chemotherapy: number analyzed (Participants) | 266 | 534
  EQ-VAS, Cycle 6 Chemotherapy | 4.6 (18.84) | 2.0 (18.69)
  EQ-VAS, Cycle 1 Maintenance: number analyzed (Participants) | 263 | 493
  EQ-VAS, Cycle 1 Maintenance | 5.9 (19.99) | 3.2 (18.25)
  EQ-VAS, Cycle 2 Maintenance: number analyzed (Participants) | 226 | 429
  EQ-VAS, Cycle 2 Maintenance | 6.9 (19.03) | 2.9 (19.52)
  EQ-VAS, Cycle 3 Maintenance: number analyzed (Participants) | 233 | 441
  EQ-VAS, Cycle 3 Maintenance | 4.9 (20.42) | 4.9 (19.32)
  EQ-VAS, Cycle 6 Maintenance: number analyzed (Participants) | 196 | 397
  EQ-VAS, Cycle 6 Maintenance | 5.1 (17.81) | 5.3 (18.80)
  EQ-VAS, Cycle 9 Maintenance: number analyzed (Participants) | 187 | 359
  EQ-VAS, Cycle 9 Maintenance | 7.6 (19.74) | 6.6 (18.09)
  EQ-VAS, Cycle 12 Maintenance: number analyzed (Participants) | 159 | 307
  EQ-VAS, Cycle 12 Maintenance | 9.6 (20.58) | 6.6 (17.59)
  EQ-VAS, Cycle 15 Maintenance: number analyzed (Participants) | 151 | 283
  EQ-VAS, Cycle 15 Maintenance | 8.1 (23.56) | 6.6 (17.72)
  EQ-VAS, Cycle 17 Maintenance: number analyzed (Participants) | 39 | 85
  EQ-VAS, Cycle 17 Maintenance | 14.8 (26.29) | 11.5 (19.81)
  EQ-VAS, Cycle 23 Maintenance: number analyzed (Participants) | 56 | 100
  EQ-VAS, Cycle 23 Maintenance | 13.3 (22.95) | 10.4 (20.89)
  EQ-VAS, Cycle 29 Maintenance: number analyzed (Participants) | 51 | 93
  EQ-VAS, Cycle 29 Maintenance | 12.5 (22.27) | 10.3 (19.06)
  EQ-VAS, Cycle 35 Maintenance: number analyzed (Participants) | 45 | 87
  EQ-VAS, Cycle 35 Maintenance | 9.9 (19.00) | 10.4 (16.55)
  EQ-VAS, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 103
  EQ-VAS, Cycle 41 Maintenance | 9.8 (22.91) | 10.1 (18.96)
  EQ-VAS, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 86
  EQ-VAS, Cycle 47 Maintenance | 8.8 (21.16) | 10.9 (18.39)
  EQ-VAS, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  EQ-VAS, Cycle 53 Maintenance | 8.5 (25.94) | 11.4 (18.65)
  EQ-VAS, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  EQ-VAS, Cycle 59 Maintenance | 7.3 (25.15) | 10.7 (18.14)
  EQ-VAS, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 26
  EQ-VAS, Cycle 65 Maintenance | 2.5 (11.10) | 14.9 (19.55)
  EQ-VAS, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 13
  EQ-VAS, Cycle 71 Maintenance | 5.9 (10.78) | 13.0 (17.09)
  EQ-VAS, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  EQ-VAS, Cycle 77 Maintenance | 9.3 (9.84) | 15.9 (18.65)
  EQ-VAS, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  EQ-VAS, Cycle 83 Maintenance | 9.7 (6.35) | 19.3 (21.45)
  EQ-VAS, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 1
  EQ-VAS, Cycle 89 Maintenance |  | -5.0 (NA) — Standard deviation is not applicable as only a single participant was analyzed.
  EQ-VAS, End of Treatment: number analyzed (Participants) | 179 | 337
  EQ-VAS, End of Treatment | 0.7 (21.93) | -0.1 (22.51)
  EQ-VAS, Safety Follow-up: number analyzed (Participants) | 144 | 287
  EQ-VAS, Safety Follow-up | 3.5 (21.89) | -0.1 (21.45)
  EQ-VAS, Long term Follow-up (LTFU) EOT + 3 months: number analyzed (Participants) | 132 | 248
  EQ-VAS, Long term Follow-up (LTFU) EOT + 3 months | 3.0 (21.47) | 2.7 (20.06)
  EQ-VAS, LTFU-EOT + 9 months: number analyzed (Participants) | 107 | 179
  EQ-VAS, LTFU-EOT + 9 months | 1.1 (18.14) | 2.4 (21.53)
  EQ-VAS, LTFU-EOT + 15 months: number analyzed (Participants) | 76 | 150
  EQ-VAS, LTFU-EOT + 15 months | 2.3 (21.57) | 4.3 (19.29)
  EQ-VAS, LTFU-EOT + 21 months: number analyzed (Participants) | 46 | 97
  EQ-VAS, LTFU-EOT + 21 months | 1.8 (19.39) | 1.8 (24.79)
  EQ-VAS, LTFU-EOT + 27 months: number analyzed (Participants) | 35 | 69
  EQ-VAS, LTFU-EOT + 27 months | 5.5 (15.87) | 5.0 (21.42)
  EQ-VAS, LTFU-EOT + 33 months: number analyzed (Participants) | 16 | 39
  EQ-VAS, LTFU-EOT + 33 months | 4.6 (21.75) | 9.2 (17.02)
  EQ-VAS, LTFU-EOT + 39 months: number analyzed (Participants) | 11 | 27
  EQ-VAS, LTFU-EOT + 39 months | 5.9 (22.38) | -1.9 (13.89)
  EQ-VAS, LTFU-EOT + 45 months: number analyzed (Participants) | 4 | 16
  EQ-VAS, LTFU-EOT + 45 months | 5.5 (19.23) | -4.7 (16.00)
  EQ-VAS, LTFU-EOT + 51 months: number analyzed (Participants) | 2 | 5
  EQ-VAS, LTFU-EOT + 51 months | 0.0 (0.0) | 3.6 (11.50)
  EQ-VAS, LTFU-EOT + 57 months: number analyzed (Participants) | 2 | 1
  EQ-VAS, LTFU-EOT + 57 months | 2.5 (3.54) | -12.0 (NA) — Standard deviation is not applicable as only a single participant was analyzed.
  EQ-VAS, LTFU-EOT + 63 months: number analyzed (Participants) | 1 | 0
  EQ-VAS, LTFU-EOT + 63 months | 0.0 (NA) — Standard deviation is not applicable as only a single participant was analyzed. |
  HUI, Cycle 4 Chemotherapy: number analyzed (Participants) | 275 | 537
  HUI, Cycle 4 Chemotherapy | -0.0033 (0.16847) | -0.0035 (0.19281)
  HUI, Cycle 6 Chemotherapy: number analyzed (Participants) | 266 | 536
  HUI, Cycle 6 Chemotherapy | -0.0049 (0.18207) | -0.0065 (0.19647)
  HUI, Cycle 1 Maintenance: number analyzed (Participants) | 262 | 494
  HUI, Cycle 1 Maintenance | 0.0034 (0.19324) | -0.0043 (0.20270)
  HUI, Cycle 2 Maintenance: number analyzed (Participants) | 226 | 433
  HUI, Cycle 2 Maintenance | 0.0118 (0.18781) | 0.0036 (0.20052)
  HUI, Cycle 3 Maintenance: number analyzed (Participants) | 234 | 443
  HUI, Cycle 3 Maintenance | -0.0015 (0.21441) | -0.0073 (0.21785)
  HUI, Cycle 6 Maintenance: number analyzed (Participants) | 196 | 399
  HUI, Cycle 6 Maintenance | 0.0184 (0.21704) | 0.0029 (0.19389)
  HUI, Cycle 9 Maintenance: number analyzed (Participants) | 184 | 358
  HUI, Cycle 9 Maintenance | 0.0281 (0.19001) | 0.0181 (0.20597)
  HUI, Cycle 12 Maintenance: number analyzed (Participants) | 159 | 308
  HUI, Cycle 12 Maintenance | 0.0326 (0.21333) | 0.0177 (0.19577)
  HUI, Cycle 15 Maintenance: number analyzed (Participants) | 149 | 281
  HUI, Cycle 15 Maintenance | 0.0379 (0.21060) | 0.0136 (0.18809)
  HUI, Cycle 17 Maintenance: number analyzed (Participants) | 39 | 85
  HUI, Cycle 17 Maintenance | 0.0777 (0.23603) | 0.0545 (0.19913)
  HUI, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 100
  HUI, Cycle 23 Maintenance | 0.0353 (0.16562) | 0.0012 (0.22021)
  HUI, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 94
  HUI, Cycle 29 Maintenance | 0.0610 (0.23268) | 0.0058 (0.18551)
  HUI, Cycle 35 Maintenance: number analyzed (Participants) | 45 | 85
  HUI, Cycle 35 Maintenance | 0.0295 (0.20956) | 0.0175 (0.19186)
  HUI, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 102
  HUI, Cycle 41 Maintenance | 0.0247 (0.23996) | 0.0084 (0.22003)
  HUI, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 85
  HUI, Cycle 47 Maintenance | 0.0251 (0.20478) | 0.0263 (0.19109)
  HUI, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  HUI, Cycle 53 Maintenance | 0.0285 (0.17721) | -0.0270 (0.20412)
  HUI, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  HUI, Cycle 59 Maintenance | 0.0156 (0.11589) | -0.0210 (0.19579)
  HUI, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 25
  HUI, Cycle 65 Maintenance | 0.0358 (0.10770) | -0.0302 (0.20843)
  HUI, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 13
  HUI, Cycle 71 Maintenance | 0.0604 (0.08941) | 0.0165 (0.11503)
  HUI, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  HUI, Cycle 77 Maintenance | 0.0783 (0.06087) | 0.0193 (0.20537)
  HUI, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  HUI, Cycle 83 Maintenance | 0.0200 (0.09952) | 0.0720 (0.08398)
  HUI, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  HUI, Cycle 89 Maintenance |  | 0.0640 (0.09051)
  HUI, End of Treatment: number analyzed (Participants) | 179 | 337
  HUI, End of Treatment | -0.0251 (0.22757) | -0.0310 (0.24320)
  HUI, Safety Follow-up: number analyzed (Participants) | 143 | 285
  HUI, Safety Follow-up | -0.0326 (0.22131) | -0.0460 (0.23927)
  HUI, LTFU- EOT + 3 months: number analyzed (Participants) | 132 | 249
  HUI, LTFU- EOT + 3 months | -0.0439 (0.22896) | -0.0222 (0.22768)
  HUI, LTFU-EOT + 9 months: number analyzed (Participants) | 107 | 180
  HUI, LTFU-EOT + 9 months | -0.0723 (0.20713) | -0.0400 (0.23756)
  HUI, LTFU-EOT + 15 months: number analyzed (Participants) | 75 | 150
  HUI, LTFU-EOT + 15 months | -0.0323 (0.20492) | -0.0386 (0.22117)
  HUI, LTFU-EOT + 21 months: number analyzed (Participants) | 45 | 96
  HUI, LTFU-EOT + 21 months | -0.0370 (0.16768) | -0.0457 (0.26270)
  HUI, LTFU-EOT + 27 months: number analyzed (Participants) | 35 | 68
  HUI, LTFU-EOT + 27 months | -0.0407 (0.17664) | -0.0635 (0.23835)
  HUI, LTFU-EOT + 33 months: number analyzed (Participants) | 15 | 39
  HUI, LTFU-EOT + 33 months | -0.0547 (0.15663) | -0.0114 (0.23974)
  HUI, LTFU-EOT + 39 months: number analyzed (Participants) | 11 | 27
  HUI, LTFU-EOT + 39 months | -0.0374 (0.11831) | -0.0993 (0.24071)
  HUI, LTFU-EOT + 45 months: number analyzed (Participants) | 4 | 16
  HUI, LTFU-EOT + 45 months | -0.0568 (0.14026) | -0.0648 (0.23505)
  HUI, LTFU-EOT + 51 months: number analyzed (Participants) | 1 | 5
  HUI, LTFU-EOT + 51 months | 0.0000 (NA) — Standard deviation is not applicable as only a single participant was analyzed. | 0.0028 (0.18532)
  HUI, LTFU-EOT + 57 months: number analyzed (Participants) | 2 | 1
  HUI, LTFU-EOT + 57 months | -0.0780 (0.11031) | 0.0000 (NA) — Standard deviation is not applicable as only a single participant was analyzed.
  HUI, LTFU-EOT + 63 months: number analyzed (Participants) | 1 | 0
  HUI, LTFU-EOT + 63 months | 0.0000 (NA) — Standard deviation is not applicable as only a single participant was analyzed. |

12. Secondary Outcome: Number of Participants With Improvement and Worsening in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTC-QLQ-C30)
Description: The EORTC QLQ-C30 includes 30-items with single and multi-item scales. These included five functional scales (physical functioning [PF], role functioning [RF], cognitive functioning [CF], emotional functioning [EF] and social functioning [SF]), three symptom scales (fatigue, pain and nausea/vomiting [N/V]), a global health status (GHS)/ Quality-of-Life (QoL) scale, and six single items (constipation, diarrhoea, insomnia, dyspnoea, appetite loss [AL] and financial difficulties [FD]). Response options are 1 to 4. Scores were averaged and transformed to 0 to 100, a high score for functional scales/ GHS/QoL represent better functioning ability or health-related quality-of-life (HRQoL), whereas a high score for symptom scales/ single items represent significant symptomatology.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 336 | 666
Participants
  GHS/QoL, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 547
  GHS/QoL, Cycle 4 Chemotherapy: Worsened | 70 | 148
  GHS/QoL, Cycle 4 Chemotherapy: Stable | 142 | 283
  GHS/QoL, Cycle 4 Chemotherapy: Improved | 71 | 116
  PF, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  PF, Cycle 4 Chemotherapy: Worsened | 77 | 150
  PF, Cycle 4 Chemotherapy: Stable | 146 | 290
  PF, Cycle 4 Chemotherapy: Improved | 60 | 108
  RF, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 547
  RF, Cycle 4 Chemotherapy: Worsened | 95 | 183
  RF, Cycle 4 Chemotherapy: Stable | 104 | 207
  RF, Cycle 4 Chemotherapy: Improved | 84 | 157
  EF, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  EF, Cycle 4 Chemotherapy: Worsened | 46 | 128
  EF, Cycle 4 Chemotherapy: Stable | 179 | 317
  EF, Cycle 4 Chemotherapy: Improved | 58 | 103
  CF, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  CF, Cycle 4 Chemotherapy: Worsened | 93 | 174
  CF, Cycle 4 Chemotherapy: Stable | 149 | 272
  CF, Cycle 4 Chemotherapy: Improved | 41 | 102
  SF, Cycle 4 Chemotherapy: number analyzed (Participants) | 282 | 548
  SF, Cycle 4 Chemotherapy: Worsened | 95 | 201
  SF, Cycle 4 Chemotherapy: Stable | 120 | 220
  SF, Cycle 4 Chemotherapy: Improved | 67 | 127
  Fatigue, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  Fatigue, Cycle 4 Chemotherapy: Worsened | 121 | 223
  Fatigue, Cycle 4 Chemotherapy: Stable | 79 | 155
  Fatigue, Cycle 4 Chemotherapy: Improved | 83 | 170
  N/V, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  N/V, Cycle 4 Chemotherapy: Worsened | 47 | 91
  N/V, Cycle 4 Chemotherapy: Stable | 191 | 363
  N/V, Cycle 4 Chemotherapy: Improved | 45 | 94
  Pain, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  Pain, Cycle 4 Chemotherapy: Worsened | 88 | 170
  Pain, Cycle 4 Chemotherapy: Stable | 107 | 224
  Pain, Cycle 4 Chemotherapy: Improved | 88 | 154
  Dyspnoea, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  Dyspnoea, Cycle 4 Chemotherapy: Worsened | 59 | 103
  Dyspnoea, Cycle 4 Chemotherapy: Stable | 179 | 346
  Dyspnoea, Cycle 4 Chemotherapy: Improved | 45 | 99
  Insomnia, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  Insomnia, Cycle 4 Chemotherapy: Worsened | 58 | 96
  Insomnia, Cycle 4 Chemotherapy: Stable | 147 | 319
  Insomnia, Cycle 4 Chemotherapy: Improved | 78 | 133
  AL, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  AL, Cycle 4 Chemotherapy: Worsened | 53 | 111
  AL, Cycle 4 Chemotherapy: Stable | 163 | 322
  AL, Cycle 4 Chemotherapy: Improved | 67 | 115
  Constipation, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  Constipation, Cycle 4 Chemotherapy: Worsened | 67 | 104
  Constipation, Cycle 4 Chemotherapy: Stable | 153 | 299
  Constipation, Cycle 4 Chemotherapy: Improved | 63 | 145
  Diarrhoea, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 548
  Diarrhoea, Cycle 4 Chemotherapy: Worsened | 41 | 82
  Diarrhoea, Cycle 4 Chemotherapy: Stable | 196 | 373
  Diarrhoea, Cycle 4 Chemotherapy: Improved | 46 | 93
  FD, Cycle 4 Chemotherapy: number analyzed (Participants) | 283 | 546
  FD, Cycle 4 Chemotherapy: Worsened | 28 | 98
  FD, Cycle 4 Chemotherapy: Stable | 214 | 380
  FD, Cycle 4 Chemotherapy: Improved | 41 | 68
  GHS/QoL, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 554
  GHS/QoL, Cycle 6 Chemotherapy: Worsened | 66 | 147
  GHS/QoL, Cycle 6 Chemotherapy: Stable | 133 | 260
  GHS/QoL, Cycle 6 Chemotherapy: Improved | 74 | 147
  PF, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 554
  PF, Cycle 6 Chemotherapy: Worsened | 80 | 163
  PF, Cycle 6 Chemotherapy: Stable | 131 | 274
  PF, Cycle 6 Chemotherapy: Improved | 62 | 117
  RF, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 553
  RF, Cycle 6 Chemotherapy: Worsened | 78 | 195
  RF, Cycle 6 Chemotherapy: Stable | 104 | 189
  RF, Cycle 6 Chemotherapy: Improved | 91 | 169
  EF, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 553
  EF, Cycle 6 Chemotherapy: Worsened | 48 | 123
  EF, Cycle 6 Chemotherapy: Stable | 162 | 316
  EF, Cycle 6 Chemotherapy: Improved | 63 | 114
  CF, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 553
  CF, Cycle 6 Chemotherapy: Worsened | 92 | 199
  CF, Cycle 6 Chemotherapy: Stable | 144 | 260
  CF, Cycle 6 Chemotherapy: Improved | 37 | 94
  SF, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 553
  SF, Cycle 6 Chemotherapy: Worsened | 79 | 185
  SF, Cycle 6 Chemotherapy: Stable | 116 | 222
  SF, Cycle 6 Chemotherapy: Improved | 78 | 146
  Fatigue, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 554
  Fatigue, Cycle 6 Chemotherapy: Worsened | 110 | 221
  Fatigue, Cycle 6 Chemotherapy: Stable | 71 | 163
  Fatigue, Cycle 6 Chemotherapy: Improved | 92 | 170
  N/V, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 554
  N/V, Cycle 6 Chemotherapy: Worsened | 43 | 116
  N/V, Cycle 6 Chemotherapy: Stable | 182 | 340
  N/V, Cycle 6 Chemotherapy: Improved | 48 | 98
  Pain, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 554
  Pain, Cycle 6 Chemotherapy: Worsened | 76 | 150
  Pain, Cycle 6 Chemotherapy: Stable | 99 | 220
  Pain, Cycle 6 Chemotherapy: Improved | 98 | 184
  Dyspnoea, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 553
  Dyspnoea, Cycle 6 Chemotherapy: Worsened | 56 | 150
  Dyspnoea, Cycle 6 Chemotherapy: Stable | 174 | 316
  Dyspnoea, Cycle 6 Chemotherapy: Improved | 43 | 87
  Insomnia, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 553
  Insomnia, Cycle 6 Chemotherapy: Worsened | 54 | 110
  Insomnia, Cycle 6 Chemotherapy: Stable | 135 | 301
  Insomnia, Cycle 6 Chemotherapy: Improved | 84 | 142
  AL, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 554
  AL, Cycle 6 Chemotherapy: Worsened | 44 | 113
  AL, Cycle 6 Chemotherapy: Stable | 162 | 288
  AL, Cycle 6 Chemotherapy: Improved | 67 | 153
  Constipation, Cycle 6 Chemotherapy: number analyzed (Participants) | 272 | 553
  Constipation, Cycle 6 Chemotherapy: Worsened | 51 | 117
  Constipation, Cycle 6 Chemotherapy: Stable | 148 | 300
  Constipation, Cycle 6 Chemotherapy: Improved | 73 | 136
  Diarrhoea, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 554
  Diarrhoea, Cycle 6 Chemotherapy: Worsened | 34 | 78
  Diarrhoea, Cycle 6 Chemotherapy: Stable | 193 | 388
  Diarrhoea, Cycle 6 Chemotherapy: Improved | 46 | 88
  FD, Cycle 6 Chemotherapy: number analyzed (Participants) | 273 | 552
  FD, Cycle 6 Chemotherapy: Worsened | 35 | 91
  FD, Cycle 6 Chemotherapy: Stable | 203 | 395
  FD, Cycle 6 Chemotherapy: Improved | 35 | 66
  GHS/QoL, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 502
  GHS/QoL, Cycle 1 Maintenance: Worsened | 50 | 135
  GHS/QoL, Cycle 1 Maintenance: Stable | 138 | 241
  GHS/QoL, Cycle 1 Maintenance: Improved | 78 | 126
  PF, Cycle 1 Maintenance: number analyzed (Participants) | 265 | 504
  PF, Cycle 1 Maintenance: Worsened | 62 | 130
  PF, Cycle 1 Maintenance: Stable | 127 | 255
  PF, Cycle 1 Maintenance: Improved | 76 | 119
  RF, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 502
  RF, Cycle 1 Maintenance: Worsened | 73 | 144
  RF, Cycle 1 Maintenance: Stable | 100 | 186
  RF, Cycle 1 Maintenance: Improved | 93 | 172
  EF, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 504
  EF, Cycle 1 Maintenance: Worsened | 55 | 127
  EF, Cycle 1 Maintenance: Stable | 150 | 283
  EF, Cycle 1 Maintenance: Improved | 61 | 94
  CF, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 504
  CF, Cycle 1 Maintenance: Worsened | 96 | 181
  CF, Cycle 1 Maintenance: Stable | 132 | 246
  CF, Cycle 1 Maintenance: Improved | 38 | 77
  SF, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 504
  SF, Cycle 1 Maintenance: Worsened | 83 | 154
  SF, Cycle 1 Maintenance: Stable | 109 | 224
  SF, Cycle 1 Maintenance: Improved | 74 | 126
  Fatigue, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 504
  Fatigue, Cycle 1 Maintenance: Worsened | 89 | 180
  Fatigue, Cycle 1 Maintenance: Stable | 71 | 145
  Fatigue, Cycle 1 Maintenance: Improved | 106 | 179
  N/V, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 504
  N/V, Cycle 1 Maintenance: Worsened | 35 | 90
  N/V, Cycle 1 Maintenance: Stable | 178 | 317
  N/V, Cycle 1 Maintenance: Improved | 53 | 97
  Pain, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 504
  Pain, Cycle 1 Maintenance: Worsened | 58 | 127
  Pain, Cycle 1 Maintenance: Stable | 104 | 186
  Pain, Cycle 1 Maintenance: Improved | 104 | 191
  Dyspnoea, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 501
  Dyspnoea, Cycle 1 Maintenance: Worsened | 64 | 109
  Dyspnoea, Cycle 1 Maintenance: Stable | 159 | 297
  Dyspnoea, Cycle 1 Maintenance: Improved | 43 | 95
  Insomnia, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 504
  Insomnia, Cycle 1 Maintenance: Worsened | 49 | 98
  Insomnia, Cycle 1 Maintenance: Stable | 143 | 253
  Insomnia, Cycle 1 Maintenance: Improved | 74 | 153
  AL, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 503
  AL, Cycle 1 Maintenance: Worsened | 40 | 86
  AL, Cycle 1 Maintenance: Stable | 154 | 285
  AL, Cycle 1 Maintenance: Improved | 72 | 132
  Constipation, Cycle 1 Maintenance: number analyzed (Participants) | 265 | 503
  Constipation, Cycle 1 Maintenance: Worsened | 54 | 88
  Constipation, Cycle 1 Maintenance: Stable | 143 | 270
  Constipation, Cycle 1 Maintenance: Improved | 68 | 145
  Diarrhoea, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 501
  Diarrhoea, Cycle 1 Maintenance: Worsened | 28 | 87
  Diarrhoea, Cycle 1 Maintenance: Stable | 189 | 338
  Diarrhoea, Cycle 1 Maintenance: Improved | 49 | 76
  FD, Cycle 1 Maintenance: number analyzed (Participants) | 266 | 503
  FD, Cycle 1 Maintenance: Worsened | 33 | 74
  FD, Cycle 1 Maintenance: Stable | 195 | 361
  FD, Cycle 1 Maintenance: Improved | 38 | 68
  GHS/QoL, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 446
  GHS/QoL, Cycle 2 Maintenance: Worsened | 47 | 118
  GHS/QoL, Cycle 2 Maintenance: Stable | 110 | 211
  GHS/QoL, Cycle 2 Maintenance: Improved | 74 | 117
  PF, Cycle 2 Maintenance: number analyzed (Participants) | 230 | 446
  PF, Cycle 2 Maintenance: Worsened | 43 | 107
  PF, Cycle 2 Maintenance: Stable | 115 | 236
  PF, Cycle 2 Maintenance: Improved | 72 | 103
  RF, Cycle 2 Maintenance: number analyzed (Participants) | 230 | 445
  RF, Cycle 2 Maintenance: Worsened | 58 | 139
  RF, Cycle 2 Maintenance: Stable | 83 | 151
  RF, Cycle 2 Maintenance: Improved | 89 | 155
  EF, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 446
  EF, Cycle 2 Maintenance: Worsened | 37 | 103
  EF, Cycle 2 Maintenance: Stable | 134 | 253
  EF, Cycle 2 Maintenance: Improved | 60 | 90
  CF, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 446
  CF, Cycle 2 Maintenance: Worsened | 78 | 160
  CF, Cycle 2 Maintenance: Stable | 117 | 208
  CF, Cycle 2 Maintenance: Improved | 36 | 78
  SF, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 446
  SF, Cycle 2 Maintenance: Worsened | 63 | 137
  SF, Cycle 2 Maintenance: Stable | 91 | 177
  SF, Cycle 2 Maintenance: Improved | 77 | 132
  Fatigue, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 445
  Fatigue, Cycle 2 Maintenance: Worsened | 55 | 146
  Fatigue, Cycle 2 Maintenance: Stable | 68 | 138
  Fatigue, Cycle 2 Maintenance: Improved | 108 | 161
  N/V, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 445
  N/V, Cycle 2 Maintenance: Worsened | 42 | 94
  N/V, Cycle 2 Maintenance: Stable | 144 | 266
  N/V, Cycle 2 Maintenance: Improved | 45 | 85
  Pain, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 446
  Pain, Cycle 2 Maintenance: Worsened | 48 | 128
  Pain, Cycle 2 Maintenance: Stable | 88 | 159
  Pain, Cycle 2 Maintenance: Improved | 95 | 159
  Dyspnoea, Cycle 2 Maintenance: number analyzed (Participants) | 230 | 445
  Dyspnoea, Cycle 2 Maintenance: Worsened | 34 | 91
  Dyspnoea, Cycle 2 Maintenance: Stable | 155 | 277
  Dyspnoea, Cycle 2 Maintenance: Improved | 41 | 77
  Insomnia, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 445
  Insomnia, Cycle 2 Maintenance: Worsened | 41 | 90
  Insomnia, Cycle 2 Maintenance: Stable | 115 | 220
  Insomnia, Cycle 2 Maintenance: Improved | 75 | 135
  AL, Cycle 2 Maintenance: number analyzed (Participants) | 230 | 445
  AL, Cycle 2 Maintenance: Worsened | 29 | 90
  AL, Cycle 2 Maintenance: Stable | 134 | 250
  AL, Cycle 2 Maintenance: Improved | 67 | 105
  Constipation, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 444
  Constipation, Cycle 2 Maintenance: Worsened | 42 | 85
  Constipation, Cycle 2 Maintenance: Stable | 118 | 249
  Constipation, Cycle 2 Maintenance: Improved | 71 | 110
  Diarrhoea, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 446
  Diarrhoea, Cycle 2 Maintenance: Worsened | 22 | 52
  Diarrhoea, Cycle 2 Maintenance: Stable | 160 | 315
  Diarrhoea, Cycle 2 Maintenance: Improved | 49 | 79
  FD, Cycle 2 Maintenance: number analyzed (Participants) | 231 | 446
  FD, Cycle 2 Maintenance: Worsened | 26 | 71
  FD, Cycle 2 Maintenance: Stable | 175 | 316
  FD, Cycle 2 Maintenance: Improved | 30 | 59
  GHS/QoL, Cycle 3 Maintenance: number analyzed (Participants) | 242 | 457
  GHS/QoL, Cycle 3 Maintenance: Worsened | 56 | 146
  GHS/QoL, Cycle 3 Maintenance: Stable | 110 | 199
  GHS/QoL, Cycle 3 Maintenance: Improved | 76 | 112
  PF, Cycle 3 Maintenance: number analyzed (Participants) | 241 | 455
  PF, Cycle 3 Maintenance: Worsened | 49 | 130
  PF, Cycle 3 Maintenance: Stable | 113 | 216
  PF, Cycle 3 Maintenance: Improved | 79 | 109
  RF, Cycle 3 Maintenance: number analyzed (Participants) | 241 | 456
  RF, Cycle 3 Maintenance: Worsened | 68 | 146
  RF, Cycle 3 Maintenance: Stable | 85 | 163
  RF, Cycle 3 Maintenance: Improved | 88 | 147
  EF, Cycle 3 Maintenance: number analyzed (Participants) | 242 | 457
  EF, Cycle 3 Maintenance: Worsened | 60 | 122
  EF, Cycle 3 Maintenance: Stable | 126 | 255
  EF, Cycle 3 Maintenance: Improved | 56 | 80
  CF, Cycle 3 Maintenance: number analyzed (Participants) | 242 | 457
  CF, Cycle 3 Maintenance: Worsened | 83 | 183
  CF, Cycle 3 Maintenance: Stable | 120 | 193
  CF, Cycle 3 Maintenance: Improved | 39 | 81
  SF, Cycle 3 Maintenance: number analyzed (Participants) | 242 | 456
  SF, Cycle 3 Maintenance: Worsened | 63 | 152
  SF, Cycle 3 Maintenance: Stable | 101 | 185
  SF, Cycle 3 Maintenance: Improved | 78 | 119
  Fatigue, Cycle 3 Maintenance: number analyzed (Participants) | 241 | 457
  Fatigue, Cycle 3 Maintenance: Worsened | 84 | 182
  Fatigue, Cycle 3 Maintenance: Stable | 51 | 119
  Fatigue, Cycle 3 Maintenance: Improved | 106 | 156
  N/V, Cycle 3 Maintenance: number analyzed (Participants) | 241 | 456
  N/V, Cycle 3 Maintenance: Worsened | 70 | 147
  N/V, Cycle 3 Maintenance: Stable | 122 | 241
  N/V, Cycle 3 Maintenance: Improved | 49 | 68
  Pain, Cycle 3 Maintenance: number analyzed (Participants) | 242 | 457
  Pain, Cycle 3 Maintenance: Worsened | 58 | 133
  Pain, Cycle 3 Maintenance: Stable | 95 | 167
  Pain, Cycle 3 Maintenance: Improved | 89 | 157
  Dyspnoea, Cycle 3 Maintenance: number analyzed (Participants) | 240 | 456
  Dyspnoea, Cycle 3 Maintenance: Worsened | 65 | 121
  Dyspnoea, Cycle 3 Maintenance: Stable | 136 | 258
  Dyspnoea, Cycle 3 Maintenance: Improved | 39 | 77
  Insomnia, Cycle 3 Maintenance: number analyzed (Participants) | 241 | 457
  Insomnia, Cycle 3 Maintenance: Worsened | 55 | 115
  Insomnia, Cycle 3 Maintenance: Stable | 117 | 221
  Insomnia, Cycle 3 Maintenance: Improved | 69 | 121
  AL, Cycle 3 Maintenance: number analyzed (Participants) | 240 | 457
  AL, Cycle 3 Maintenance: Worsened | 45 | 124
  AL, Cycle 3 Maintenance: Stable | 129 | 229
  AL, Cycle 3 Maintenance: Improved | 66 | 104
  Constipation, Cycle 3 Maintenance: number analyzed (Participants) | 241 | 457
  Constipation, Cycle 3 Maintenance: Worsened | 73 | 125
  Constipation, Cycle 3 Maintenance: Stable | 110 | 221
  Constipation, Cycle 3 Maintenance: Improved | 58 | 111
  Diarrhoea, Cycle 3 Maintenance: number analyzed (Participants) | 242 | 457
  Diarrhoea, Cycle 3 Maintenance: Worsened | 15 | 38
  Diarrhoea, Cycle 3 Maintenance: Stable | 177 | 329
  Diarrhoea, Cycle 3 Maintenance: Improved | 50 | 90
  FD, Cycle 3 Maintenance: number analyzed (Participants) | 242 | 455
  FD, Cycle 3 Maintenance: Worsened | 31 | 68
  FD, Cycle 3 Maintenance: Stable | 171 | 327
  FD, Cycle 3 Maintenance: Improved | 40 | 60
  GHS/QoL, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 410
  GHS/QoL, Cycle 6 Maintenance: Worsened | 30 | 89
  GHS/QoL, Cycle 6 Maintenance: Stable | 101 | 192
  GHS/QoL, Cycle 6 Maintenance: Improved | 70 | 129
  PF, Cycle 6 Maintenance: number analyzed (Participants) | 200 | 409
  PF, Cycle 6 Maintenance: Worsened | 39 | 86
  PF, Cycle 6 Maintenance: Stable | 96 | 222
  PF, Cycle 6 Maintenance: Improved | 65 | 101
  RF, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 410
  RF, Cycle 6 Maintenance: Worsened | 52 | 100
  RF, Cycle 6 Maintenance: Stable | 75 | 171
  RF, Cycle 6 Maintenance: Improved | 74 | 139
  EF, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 410
  EF, Cycle 6 Maintenance: Worsened | 36 | 86
  EF, Cycle 6 Maintenance: Stable | 113 | 246
  EF, Cycle 6 Maintenance: Improved | 52 | 78
  CF, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 410
  CF, Cycle 6 Maintenance: Worsened | 68 | 134
  CF, Cycle 6 Maintenance: Stable | 95 | 201
  CF, Cycle 6 Maintenance: Improved | 38 | 75
  SF, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 410
  SF, Cycle 6 Maintenance: Worsened | 43 | 106
  SF, Cycle 6 Maintenance: Stable | 91 | 162
  SF, Cycle 6 Maintenance: Improved | 67 | 142
  Fatigue, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 409
  Fatigue, Cycle 6 Maintenance: Worsened | 49 | 132
  Fatigue, Cycle 6 Maintenance: Stable | 59 | 110
  Fatigue, Cycle 6 Maintenance: Improved | 93 | 167
  N/V, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 409
  N/V, Cycle 6 Maintenance: Worsened | 36 | 91
  N/V, Cycle 6 Maintenance: Stable | 126 | 247
  N/V, Cycle 6 Maintenance: Improved | 39 | 71
  Pain, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 410
  Pain, Cycle 6 Maintenance: Worsened | 44 | 96
  Pain, Cycle 6 Maintenance: Stable | 85 | 161
  Pain, Cycle 6 Maintenance: Improved | 72 | 153
  Dyspnoea, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 408
  Dyspnoea, Cycle 6 Maintenance: Worsened | 43 | 105
  Dyspnoea, Cycle 6 Maintenance: Stable | 125 | 240
  Dyspnoea, Cycle 6 Maintenance: Improved | 33 | 63
  Insomnia, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 409
  Insomnia, Cycle 6 Maintenance: Worsened | 43 | 88
  Insomnia, Cycle 6 Maintenance: Stable | 99 | 211
  Insomnia, Cycle 6 Maintenance: Improved | 59 | 110
  AL, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 408
  AL, Cycle 6 Maintenance: Worsened | 29 | 68
  AL, Cycle 6 Maintenance: Stable | 111 | 232
  AL, Cycle 6 Maintenance: Improved | 61 | 108
  Constipation, Cycle 6 Maintenance: number analyzed (Participants) | 200 | 406
  Constipation, Cycle 6 Maintenance: Worsened | 62 | 106
  Constipation, Cycle 6 Maintenance: Stable | 89 | 207
  Constipation, Cycle 6 Maintenance: Improved | 49 | 93
  Diarrhoea, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 409
  Diarrhoea, Cycle 6 Maintenance: Worsened | 8 | 45
  Diarrhoea, Cycle 6 Maintenance: Stable | 152 | 293
  Diarrhoea, Cycle 6 Maintenance: Improved | 41 | 71
  FD, Cycle 6 Maintenance: number analyzed (Participants) | 201 | 409
  FD, Cycle 6 Maintenance: Worsened | 21 | 50
  FD, Cycle 6 Maintenance: Stable | 145 | 299
  FD, Cycle 6 Maintenance: Improved | 35 | 60
  GHS/QoL, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  GHS/QoL, Cycle 9 Maintenance: Worsened | 22 | 76
  GHS/QoL, Cycle 9 Maintenance: Stable | 100 | 167
  GHS/QoL, Cycle 9 Maintenance: Improved | 68 | 127
  PF, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 368
  PF, Cycle 9 Maintenance: Worsened | 30 | 80
  PF, Cycle 9 Maintenance: Stable | 91 | 192
  PF, Cycle 9 Maintenance: Improved | 69 | 96
  RF, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 369
  RF, Cycle 9 Maintenance: Worsened | 41 | 84
  RF, Cycle 9 Maintenance: Stable | 71 | 140
  RF, Cycle 9 Maintenance: Improved | 78 | 145
  EF, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  EF, Cycle 9 Maintenance: Worsened | 29 | 70
  EF, Cycle 9 Maintenance: Stable | 105 | 220
  EF, Cycle 9 Maintenance: Improved | 56 | 80
  CF, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  CF, Cycle 9 Maintenance: Worsened | 57 | 113
  CF, Cycle 9 Maintenance: Stable | 102 | 183
  CF, Cycle 9 Maintenance: Improved | 31 | 74
  SF, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  SF, Cycle 9 Maintenance: Worsened | 37 | 82
  SF, Cycle 9 Maintenance: Stable | 88 | 168
  SF, Cycle 9 Maintenance: Improved | 65 | 120
  Fatigue, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  Fatigue, Cycle 9 Maintenance: Worsened | 52 | 101
  Fatigue, Cycle 9 Maintenance: Stable | 47 | 105
  Fatigue, Cycle 9 Maintenance: Improved | 91 | 164
  N/V, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  N/V, Cycle 9 Maintenance: Worsened | 35 | 65
  N/V, Cycle 9 Maintenance: Stable | 114 | 234
  N/V, Cycle 9 Maintenance: Improved | 41 | 71
  Pain, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  Pain, Cycle 9 Maintenance: Worsened | 36 | 99
  Pain, Cycle 9 Maintenance: Stable | 77 | 145
  Pain, Cycle 9 Maintenance: Improved | 77 | 126
  Dyspnoea, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  Dyspnoea, Cycle 9 Maintenance: Worsened | 37 | 73
  Dyspnoea, Cycle 9 Maintenance: Stable | 119 | 223
  Dyspnoea, Cycle 9 Maintenance: Improved | 34 | 74
  Insomnia, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 369
  Insomnia, Cycle 9 Maintenance: Worsened | 46 | 73
  Insomnia, Cycle 9 Maintenance: Stable | 81 | 184
  Insomnia, Cycle 9 Maintenance: Improved | 63 | 112
  AL, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 370
  AL, Cycle 9 Maintenance: Worsened | 14 | 58
  AL, Cycle 9 Maintenance: Stable | 121 | 199
  AL, Cycle 9 Maintenance: Improved | 55 | 113
  Constipation, Cycle 9 Maintenance: number analyzed (Participants) | 189 | 369
  Constipation, Cycle 9 Maintenance: Worsened | 62 | 89
  Constipation, Cycle 9 Maintenance: Stable | 83 | 189
  Constipation, Cycle 9 Maintenance: Improved | 44 | 91
  Diarrhoea, Cycle 9 Maintenance: number analyzed (Participants) | 189 | 369
  Diarrhoea, Cycle 9 Maintenance: Worsened | 15 | 36
  Diarrhoea, Cycle 9 Maintenance: Stable | 138 | 264
  Diarrhoea, Cycle 9 Maintenance: Improved | 36 | 69
  FD, Cycle 9 Maintenance: number analyzed (Participants) | 190 | 369
  FD, Cycle 9 Maintenance: Worsened | 18 | 42
  FD, Cycle 9 Maintenance: Stable | 145 | 276
  FD, Cycle 9 Maintenance: Improved | 27 | 51
  GHS/QoL, Cycle 12 Maintenance: number analyzed (Participants) | 162 | 316
  GHS/QoL, Cycle 12 Maintenance: Worsened | 23 | 64
  GHS/QoL, Cycle 12 Maintenance: Stable | 69 | 141
  GHS/QoL, Cycle 12 Maintenance: Improved | 70 | 111
  PF, Cycle 12 Maintenance: number analyzed (Participants) | 161 | 314
  PF, Cycle 12 Maintenance: Worsened | 22 | 60
  PF, Cycle 12 Maintenance: Stable | 82 | 167
  PF, Cycle 12 Maintenance: Improved | 57 | 87
  RF, Cycle 12 Maintenance: number analyzed (Participants) | 161 | 313
  RF, Cycle 12 Maintenance: Worsened | 29 | 57
  RF, Cycle 12 Maintenance: Stable | 68 | 127
  RF, Cycle 12 Maintenance: Improved | 64 | 129
  EF, Cycle 12 Maintenance: number analyzed (Participants) | 162 | 315
  EF, Cycle 12 Maintenance: Worsened | 31 | 69
  EF, Cycle 12 Maintenance: Stable | 82 | 181
  EF, Cycle 12 Maintenance: Improved | 49 | 65
  CF, Cycle 12 Maintenance: number analyzed (Participants) | 162 | 315
  CF, Cycle 12 Maintenance: Worsened | 50 | 106
  CF, Cycle 12 Maintenance: Stable | 86 | 154
  CF, Cycle 12 Maintenance: Improved | 26 | 55
  SF, Cycle 12 Maintenance: number analyzed (Participants) | 162 | 314
  SF, Cycle 12 Maintenance: Worsened | 27 | 74
  SF, Cycle 12 Maintenance: Stable | 69 | 123
  SF, Cycle 12 Maintenance: Improved | 66 | 117
  Fatigue, Cycle 12 Maintenance: number analyzed (Participants) | 161 | 315
  Fatigue, Cycle 12 Maintenance: Worsened | 39 | 87
  Fatigue, Cycle 12 Maintenance: Stable | 42 | 88
  Fatigue, Cycle 12 Maintenance: Improved | 80 | 140
  N/V, Cycle 12 Maintenance: number analyzed (Participants) | 161 | 314
  N/V, Cycle 12 Maintenance: Worsened | 21 | 62
  N/V, Cycle 12 Maintenance: Stable | 105 | 190
  N/V, Cycle 12 Maintenance: Improved | 35 | 62
  Pain, Cycle 12 Maintenance: number analyzed (Participants) | 162 | 316
  Pain, Cycle 12 Maintenance: Worsened | 33 | 100
  Pain, Cycle 12 Maintenance: Stable | 71 | 97
  Pain, Cycle 12 Maintenance: Improved | 58 | 119
  Dyspnoea, Cycle 12 Maintenance: number analyzed (Participants) | 160 | 314
  Dyspnoea, Cycle 12 Maintenance: Worsened | 27 | 57
  Dyspnoea, Cycle 12 Maintenance: Stable | 107 | 197
  Dyspnoea, Cycle 12 Maintenance: Improved | 26 | 60
  Insomnia, Cycle 12 Maintenance: number analyzed (Participants) | 161 | 314
  Insomnia, Cycle 12 Maintenance: Worsened | 28 | 69
  Insomnia, Cycle 12 Maintenance: Stable | 80 | 161
  Insomnia, Cycle 12 Maintenance: Improved | 53 | 84
  AL, Cycle 12 Maintenance: number analyzed (Participants) | 161 | 314
  AL, Cycle 12 Maintenance: Worsened | 12 | 49
  AL, Cycle 12 Maintenance: Stable | 99 | 173
  AL, Cycle 12 Maintenance: Improved | 50 | 92
  Constipation, Cycle 12 Maintenance: number analyzed (Participants) | 161 | 314
  Constipation, Cycle 12 Maintenance: Worsened | 38 | 90
  Constipation, Cycle 12 Maintenance: Stable | 79 | 150
  Constipation, Cycle 12 Maintenance: Improved | 44 | 74
  Diarrhoea, Cycle 12 Maintenance: number analyzed (Participants) | 162 | 316
  Diarrhoea, Cycle 12 Maintenance: Worsened | 12 | 42
  Diarrhoea, Cycle 12 Maintenance: Stable | 119 | 221
  Diarrhoea, Cycle 12 Maintenance: Improved | 31 | 53
  FD, Cycle 12 Maintenance: number analyzed (Participants) | 162 | 313
  FD, Cycle 12 Maintenance: Worsened | 17 | 41
  FD, Cycle 12 Maintenance: Stable | 126 | 222
  FD, Cycle 12 Maintenance: Improved | 19 | 50
  GHS/QoL, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 287
  GHS/QoL, Cycle 15 Maintenance: Worsened | 26 | 60
  GHS/QoL, Cycle 15 Maintenance: Stable | 67 | 142
  GHS/QoL, Cycle 15 Maintenance: Improved | 60 | 85
  PF, Cycle 15 Maintenance: number analyzed (Participants) | 151 | 285
  PF, Cycle 15 Maintenance: Worsened | 24 | 63
  PF, Cycle 15 Maintenance: Stable | 67 | 137
  PF, Cycle 15 Maintenance: Improved | 60 | 85
  RF, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 286
  RF, Cycle 15 Maintenance: Worsened | 25 | 60
  RF, Cycle 15 Maintenance: Stable | 60 | 108
  RF, Cycle 15 Maintenance: Improved | 68 | 118
  EF, Cycle 15 Maintenance: number analyzed (Participants) | 152 | 287
  EF, Cycle 15 Maintenance: Worsened | 37 | 59
  EF, Cycle 15 Maintenance: Stable | 78 | 160
  EF, Cycle 15 Maintenance: Improved | 37 | 68
  CF, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 287
  CF, Cycle 15 Maintenance: Worsened | 54 | 111
  CF, Cycle 15 Maintenance: Stable | 78 | 120
  CF, Cycle 15 Maintenance: Improved | 21 | 56
  SF, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 287
  SF, Cycle 15 Maintenance: Worsened | 27 | 61
  SF, Cycle 15 Maintenance: Stable | 70 | 121
  SF, Cycle 15 Maintenance: Improved | 56 | 105
  Fatigue, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 287
  Fatigue, Cycle 15 Maintenance: Worsened | 38 | 81
  Fatigue, Cycle 15 Maintenance: Stable | 40 | 74
  Fatigue, Cycle 15 Maintenance: Improved | 75 | 132
  N/V, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 285
  N/V, Cycle 15 Maintenance: Worsened | 29 | 47
  N/V, Cycle 15 Maintenance: Stable | 92 | 179
  N/V, Cycle 15 Maintenance: Improved | 32 | 59
  Pain, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 287
  Pain, Cycle 15 Maintenance: Worsened | 38 | 71
  Pain, Cycle 15 Maintenance: Stable | 58 | 102
  Pain, Cycle 15 Maintenance: Improved | 57 | 114
  Dyspnoea, Cycle 15 Maintenance: number analyzed (Participants) | 152 | 287
  Dyspnoea, Cycle 15 Maintenance: Worsened | 28 | 59
  Dyspnoea, Cycle 15 Maintenance: Stable | 95 | 172
  Dyspnoea, Cycle 15 Maintenance: Improved | 29 | 56
  Insomnia, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 286
  Insomnia, Cycle 15 Maintenance: Worsened | 37 | 65
  Insomnia, Cycle 15 Maintenance: Stable | 73 | 128
  Insomnia, Cycle 15 Maintenance: Improved | 43 | 93
  AL, Cycle 15 Maintenance: number analyzed (Participants) | 152 | 285
  AL, Cycle 15 Maintenance: Worsened | 13 | 29
  AL, Cycle 15 Maintenance: Stable | 89 | 164
  AL, Cycle 15 Maintenance: Improved | 50 | 92
  Constipation, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 286
  Constipation, Cycle 15 Maintenance: Worsened | 38 | 66
  Constipation, Cycle 15 Maintenance: Stable | 76 | 147
  Constipation, Cycle 15 Maintenance: Improved | 39 | 73
  Diarrhoea, Cycle 15 Maintenance: number analyzed (Participants) | 153 | 287
  Diarrhoea, Cycle 15 Maintenance: Worsened | 12 | 29
  Diarrhoea, Cycle 15 Maintenance: Stable | 116 | 200
  Diarrhoea, Cycle 15 Maintenance: Improved | 25 | 58
  FD, Cycle 15 Maintenance: number analyzed (Participants) | 152 | 286
  FD, Cycle 15 Maintenance: Worsened | 16 | 47
  FD, Cycle 15 Maintenance: Stable | 116 | 195
  FD, Cycle 15 Maintenance: Improved | 20 | 44
  GHS/QoL, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  GHS/QoL, Cycle 17 Maintenance: Worsened | 4 | 13
  GHS/QoL, Cycle 17 Maintenance: Stable | 24 | 33
  GHS/QoL, Cycle 17 Maintenance: Improved | 12 | 39
  PF, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  PF, Cycle 17 Maintenance: Worsened | 7 | 13
  PF, Cycle 17 Maintenance: Stable | 20 | 38
  PF, Cycle 17 Maintenance: Improved | 13 | 34
  RF, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  RF, Cycle 17 Maintenance: Worsened | 10 | 20
  RF, Cycle 17 Maintenance: Stable | 14 | 24
  RF, Cycle 17 Maintenance: Improved | 16 | 41
  EF, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  EF, Cycle 17 Maintenance: Worsened | 4 | 15
  EF, Cycle 17 Maintenance: Stable | 20 | 50
  EF, Cycle 17 Maintenance: Improved | 16 | 20
  CF, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  CF, Cycle 17 Maintenance: Worsened | 13 | 32
  CF, Cycle 17 Maintenance: Stable | 21 | 42
  CF, Cycle 17 Maintenance: Improved | 6 | 11
  SF, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  SF, Cycle 17 Maintenance: Worsened | 6 | 22
  SF, Cycle 17 Maintenance: Stable | 20 | 29
  SF, Cycle 17 Maintenance: Improved | 14 | 34
  Fatigue, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  Fatigue, Cycle 17 Maintenance: Worsened | 6 | 20
  Fatigue, Cycle 17 Maintenance: Stable | 14 | 27
  Fatigue, Cycle 17 Maintenance: Improved | 20 | 38
  N/V, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  N/V, Cycle 17 Maintenance: Worsened | 8 | 17
  N/V, Cycle 17 Maintenance: Stable | 22 | 42
  N/V, Cycle 17 Maintenance: Improved | 10 | 26
  Pain, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  Pain, Cycle 17 Maintenance: Worsened | 8 | 23
  Pain, Cycle 17 Maintenance: Stable | 13 | 26
  Pain, Cycle 17 Maintenance: Improved | 19 | 36
  Dyspnoea, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  Dyspnoea, Cycle 17 Maintenance: Worsened | 6 | 19
  Dyspnoea, Cycle 17 Maintenance: Stable | 25 | 49
  Dyspnoea, Cycle 17 Maintenance: Improved | 9 | 17
  Insomnia, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  Insomnia, Cycle 17 Maintenance: Worsened | 8 | 18
  Insomnia, Cycle 17 Maintenance: Stable | 19 | 38
  Insomnia, Cycle 17 Maintenance: Improved | 13 | 29
  AL, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  AL, Cycle 17 Maintenance: Worsened | 6 | 6
  AL, Cycle 17 Maintenance: Stable | 27 | 51
  AL, Cycle 17 Maintenance: Improved | 7 | 28
  Constipation, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  Constipation, Cycle 17 Maintenance: Worsened | 6 | 19
  Constipation, Cycle 17 Maintenance: Stable | 22 | 39
  Constipation, Cycle 17 Maintenance: Improved | 12 | 27
  Diarrhoea, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  Diarrhoea, Cycle 17 Maintenance: Worsened | 7 | 10
  Diarrhoea, Cycle 17 Maintenance: Stable | 24 | 60
  Diarrhoea, Cycle 17 Maintenance: Improved | 9 | 15
  FD, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 85
  FD, Cycle 17 Maintenance: Worsened | 7 | 11
  FD, Cycle 17 Maintenance: Stable | 26 | 59
  FD, Cycle 17 Maintenance: Improved | 7 | 15
  GHS/QoL, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 102
  GHS/QoL, Cycle 23 Maintenance: Worsened | 9 | 16
  GHS/QoL, Cycle 23 Maintenance: Stable | 27 | 37
  GHS/QoL, Cycle 23 Maintenance: Improved | 19 | 49
  PF, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 100
  PF, Cycle 23 Maintenance: Worsened | 10 | 17
  PF, Cycle 23 Maintenance: Stable | 29 | 45
  PF, Cycle 23 Maintenance: Improved | 16 | 38
  RF, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 99
  RF, Cycle 23 Maintenance: Worsened | 12 | 21
  RF, Cycle 23 Maintenance: Stable | 23 | 33
  RF, Cycle 23 Maintenance: Improved | 20 | 45
  EF, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 101
  EF, Cycle 23 Maintenance: Worsened | 10 | 19
  EF, Cycle 23 Maintenance: Stable | 33 | 57
  EF, Cycle 23 Maintenance: Improved | 12 | 25
  CF, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 102
  CF, Cycle 23 Maintenance: Worsened | 15 | 37
  CF, Cycle 23 Maintenance: Stable | 28 | 48
  CF, Cycle 23 Maintenance: Improved | 12 | 17
  SF, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 102
  SF, Cycle 23 Maintenance: Worsened | 12 | 24
  SF, Cycle 23 Maintenance: Stable | 31 | 35
  SF, Cycle 23 Maintenance: Improved | 12 | 43
  Fatigue, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 101
  Fatigue, Cycle 23 Maintenance: Worsened | 10 | 25
  Fatigue, Cycle 23 Maintenance: Stable | 15 | 27
  Fatigue, Cycle 23 Maintenance: Improved | 30 | 49
  N/V, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 101
  N/V, Cycle 23 Maintenance: Worsened | 8 | 15
  N/V, Cycle 23 Maintenance: Stable | 36 | 63
  N/V, Cycle 23 Maintenance: Improved | 11 | 23
  Pain, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 101
  Pain, Cycle 23 Maintenance: Worsened | 13 | 22
  Pain, Cycle 23 Maintenance: Stable | 19 | 39
  Pain, Cycle 23 Maintenance: Improved | 23 | 40
  Dyspnoea, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 100
  Dyspnoea, Cycle 23 Maintenance: Worsened | 7 | 15
  Dyspnoea, Cycle 23 Maintenance: Stable | 37 | 62
  Dyspnoea, Cycle 23 Maintenance: Improved | 11 | 23
  Insomnia, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 102
  Insomnia, Cycle 23 Maintenance: Worsened | 10 | 20
  Insomnia, Cycle 23 Maintenance: Stable | 27 | 43
  Insomnia, Cycle 23 Maintenance: Improved | 18 | 39
  AL, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 100
  AL, Cycle 23 Maintenance: Worsened | 6 | 12
  AL, Cycle 23 Maintenance: Stable | 40 | 58
  AL, Cycle 23 Maintenance: Improved | 9 | 30
  Constipation, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 99
  Constipation, Cycle 23 Maintenance: Worsened | 8 | 27
  Constipation, Cycle 23 Maintenance: Stable | 34 | 49
  Constipation, Cycle 23 Maintenance: Improved | 13 | 23
  Diarrhoea, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 101
  Diarrhoea, Cycle 23 Maintenance: Worsened | 4 | 9
  Diarrhoea, Cycle 23 Maintenance: Stable | 41 | 70
  Diarrhoea, Cycle 23 Maintenance: Improved | 10 | 22
  FD, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 101
  FD, Cycle 23 Maintenance: Worsened | 7 | 18
  FD, Cycle 23 Maintenance: Stable | 42 | 65
  FD, Cycle 23 Maintenance: Improved | 6 | 18
  GHS/QoL, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 98
  GHS/QoL, Cycle 29 Maintenance: Worsened | 5 | 21
  GHS/QoL, Cycle 29 Maintenance: Stable | 27 | 37
  GHS/QoL, Cycle 29 Maintenance: Improved | 20 | 40
  PF, Cycle 29 Maintenance 20: number analyzed (Participants) | 52 | 97
  PF, Cycle 29 Maintenance 20: Worsened | 4 | 17
  PF, Cycle 29 Maintenance 20: Stable | 29 | 50
  PF, Cycle 29 Maintenance 20: Improved | 19 | 30
  RF, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 97
  RF, Cycle 29 Maintenance: Worsened | 5 | 20
  RF, Cycle 29 Maintenance: Stable | 22 | 40
  RF, Cycle 29 Maintenance: Improved | 25 | 37
  EF, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 98
  EF, Cycle 29 Maintenance: Worsened | 5 | 21
  EF, Cycle 29 Maintenance: Stable | 32 | 58
  EF, Cycle 29 Maintenance: Improved | 15 | 19
  CF, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 98
  CF, Cycle 29 Maintenance: Worsened | 11 | 35
  CF, Cycle 29 Maintenance: Stable | 29 | 46
  CF, Cycle 29 Maintenance: Improved | 12 | 17
  SF, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 98
  SF, Cycle 29 Maintenance: Worsened | 12 | 24
  SF, Cycle 29 Maintenance: Stable | 20 | 37
  SF, Cycle 29 Maintenance: Improved | 20 | 37
  Fatigue, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 97
  Fatigue, Cycle 29 Maintenance: Worsened | 10 | 24
  Fatigue, Cycle 29 Maintenance: Stable | 17 | 22
  Fatigue, Cycle 29 Maintenance: Improved | 25 | 51
  N/V, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 97
  N/V, Cycle 29 Maintenance: Worsened | 4 | 9
  N/V, Cycle 29 Maintenance: Stable | 37 | 64
  N/V, Cycle 29 Maintenance: Improved | 11 | 24
  Pain, Cycle 29 Maintenance: number analyzed (Participants) | 51 | 98
  Pain, Cycle 29 Maintenance: Worsened | 10 | 27
  Pain, Cycle 29 Maintenance: Stable | 20 | 43
  Pain, Cycle 29 Maintenance: Improved | 21 | 28
  Dyspnoea, Cycle 29 Maintenance: number analyzed (Participants) | 51 | 96
  Dyspnoea, Cycle 29 Maintenance: Worsened | 9 | 17
  Dyspnoea, Cycle 29 Maintenance: Stable | 30 | 66
  Dyspnoea, Cycle 29 Maintenance: Improved | 12 | 13
  Insomnia, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 97
  Insomnia, Cycle 29 Maintenance: Worsened | 14 | 24
  Insomnia, Cycle 29 Maintenance: Stable | 24 | 47
  Insomnia, Cycle 29 Maintenance: Improved | 14 | 26
  AL, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 96
  AL, Cycle 29 Maintenance: Worsened | 4 | 8
  AL, Cycle 29 Maintenance: Stable | 37 | 58
  AL, Cycle 29 Maintenance: Improved | 11 | 30
  Constipation, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 97
  Constipation, Cycle 29 Maintenance: Worsened | 5 | 19
  Constipation, Cycle 29 Maintenance: Stable | 29 | 60
  Constipation, Cycle 29 Maintenance: Improved | 18 | 18
  Diarrhoea, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 98
  Diarrhoea, Cycle 29 Maintenance: Worsened | 3 | 6
  Diarrhoea, Cycle 29 Maintenance: Stable | 39 | 76
  Diarrhoea, Cycle 29 Maintenance: Improved | 10 | 16
  FD, Cycle 29 Maintenance: number analyzed (Participants) | 52 | 98
  FD, Cycle 29 Maintenance: Worsened | 2 | 13
  FD, Cycle 29 Maintenance: Stable | 42 | 66
  FD, Cycle 29 Maintenance: Improved | 8 | 19
  GHS/QoL, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  GHS/QoL, Cycle 35 Maintenance: Worsened | 4 | 17
  GHS/QoL, Cycle 35 Maintenance: Stable | 24 | 38
  GHS/QoL, Cycle 35 Maintenance: Improved | 16 | 34
  PF, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 90
  PF, Cycle 35 Maintenance: Worsened | 9 | 19
  PF, Cycle 35 Maintenance: Stable | 19 | 45
  PF, Cycle 35 Maintenance: Improved | 16 | 26
  RF, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  RF, Cycle 35 Maintenance: Worsened | 6 | 22
  RF, Cycle 35 Maintenance: Stable | 21 | 35
  RF, Cycle 35 Maintenance: Improved | 17 | 32
  EF, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  EF, Cycle 35 Maintenance: Worsened | 8 | 16
  EF, Cycle 35 Maintenance: Stable | 24 | 51
  EF, Cycle 35 Maintenance: Improved | 12 | 22
  CF, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  CF, Cycle 35 Maintenance: Worsened | 15 | 29
  CF, Cycle 35 Maintenance: Stable | 23 | 43
  CF, Cycle 35 Maintenance: Improved | 6 | 17
  SF, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  SF, Cycle 35 Maintenance: Worsened | 11 | 18
  SF, Cycle 35 Maintenance: Stable | 21 | 29
  SF, Cycle 35 Maintenance: Improved | 12 | 42
  Fatigue, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  Fatigue, Cycle 35 Maintenance: Worsened | 10 | 25
  Fatigue, Cycle 35 Maintenance: Stable | 10 | 23
  Fatigue, Cycle 35 Maintenance: Improved | 24 | 41
  N/V, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 88
  N/V, Cycle 35 Maintenance: Worsened | 6 | 17
  N/V, Cycle 35 Maintenance: Stable | 33 | 53
  N/V, Cycle 35 Maintenance: Improved | 5 | 18
  Pain, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 90
  Pain, Cycle 35 Maintenance: Worsened | 6 | 30
  Pain, Cycle 35 Maintenance: Stable | 19 | 33
  Pain, Cycle 35 Maintenance: Improved | 19 | 27
  Dyspnoea, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  Dyspnoea, Cycle 35 Maintenance: Worsened | 8 | 21
  Dyspnoea, Cycle 35 Maintenance: Stable | 30 | 57
  Dyspnoea, Cycle 35 Maintenance: Improved | 6 | 11
  Insomnia, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  Insomnia, Cycle 35 Maintenance: Worsened | 15 | 22
  Insomnia, Cycle 35 Maintenance: Stable | 20 | 41
  Insomnia, Cycle 35 Maintenance: Improved | 9 | 26
  AL, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 87
  AL, Cycle 35 Maintenance: Worsened | 3 | 7
  AL, Cycle 35 Maintenance: Stable | 36 | 51
  AL, Cycle 35 Maintenance: Improved | 5 | 29
  Constipation, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 87
  Constipation, Cycle 35 Maintenance: Worsened | 5 | 19
  Constipation, Cycle 35 Maintenance: Stable | 27 | 48
  Constipation, Cycle 35 Maintenance: Improved | 12 | 20
  Diarrhoea, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 88
  Diarrhoea, Cycle 35 Maintenance: Worsened | 4 | 8
  Diarrhoea, Cycle 35 Maintenance: Stable | 35 | 69
  Diarrhoea, Cycle 35 Maintenance: Improved | 5 | 11
  FD, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 89
  FD, Cycle 35 Maintenance: Worsened | 6 | 15
  FD, Cycle 35 Maintenance: Stable | 30 | 53
  FD, Cycle 35 Maintenance: Improved | 8 | 21
  GHS/QoL, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  GHS/QoL, Cycle 41 Maintenance: Worsened | 10 | 22
  GHS/QoL, Cycle 41 Maintenance: Stable | 26 | 46
  GHS/QoL, Cycle 41 Maintenance: Improved | 22 | 39
  PF, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 106
  PF, Cycle 41 Maintenance: Worsened | 5 | 26
  PF, Cycle 41 Maintenance: Stable | 32 | 54
  PF, Cycle 41 Maintenance: Improved | 21 | 26
  RF, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 106
  RF, Cycle 41 Maintenance: Worsened | 9 | 29
  RF, Cycle 41 Maintenance: Stable | 25 | 38
  RF, Cycle 41 Maintenance: Improved | 24 | 39
  EF, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  EF, Cycle 41 Maintenance: Worsened | 10 | 23
  EF, Cycle 41 Maintenance: Stable | 35 | 55
  EF, Cycle 41 Maintenance: Improved | 13 | 29
  CF, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  CF, Cycle 41 Maintenance: Worsened | 23 | 42
  CF, Cycle 41 Maintenance: Stable | 25 | 46
  CF, Cycle 41 Maintenance: Improved | 10 | 19
  SF, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  SF, Cycle 41 Maintenance: Worsened | 13 | 28
  SF, Cycle 41 Maintenance: Stable | 25 | 38
  SF, Cycle 41 Maintenance: Improved | 20 | 41
  Fatigue, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 106
  Fatigue, Cycle 41 Maintenance: Worsened | 11 | 35
  Fatigue, Cycle 41 Maintenance: Stable | 17 | 27
  Fatigue, Cycle 41 Maintenance: Improved | 30 | 44
  N/V, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  N/V, Cycle 41 Maintenance: Worsened | 8 | 17
  N/V, Cycle 41 Maintenance: Stable | 39 | 66
  N/V, Cycle 41 Maintenance: Improved | 11 | 24
  Pain, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  Pain, Cycle 41 Maintenance: Worsened | 11 | 35
  Pain, Cycle 41 Maintenance: Stable | 23 | 41
  Pain, Cycle 41 Maintenance: Improved | 24 | 31
  Dyspnoea, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  Dyspnoea, Cycle 41 Maintenance: Worsened | 8 | 26
  Dyspnoea, Cycle 41 Maintenance: Stable | 39 | 71
  Dyspnoea, Cycle 41 Maintenance: Improved | 11 | 10
  Insomnia, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  Insomnia, Cycle 41 Maintenance: Worsened | 16 | 30
  Insomnia, Cycle 41 Maintenance: Stable | 25 | 52
  Insomnia, Cycle 41 Maintenance: Improved | 17 | 25
  AL, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  AL, Cycle 41 Maintenance: Worsened | 9 | 14
  AL, Cycle 41 Maintenance: Stable | 38 | 60
  AL, Cycle 41 Maintenance: Improved | 11 | 33
  Constipation, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  Constipation, Cycle 41 Maintenance: Worsened | 12 | 28
  Constipation, Cycle 41 Maintenance: Stable | 33 | 47
  Constipation, Cycle 41 Maintenance: Improved | 13 | 32
  Diarrhoea, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  Diarrhoea, Cycle 41 Maintenance: Worsened | 5 | 5
  Diarrhoea, Cycle 41 Maintenance: Stable | 44 | 85
  Diarrhoea, Cycle 41 Maintenance: Improved | 9 | 17
  FD, Cycle 41 Maintenance: number analyzed (Participants) | 58 | 107
  FD, Cycle 41 Maintenance: Worsened | 8 | 18
  FD, Cycle 41 Maintenance: Stable | 42 | 69
  FD, Cycle 41 Maintenance: Improved | 8 | 20
  GHS/QoL, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  GHS/QoL, Cycle 47 Maintenance: Worsened | 5 | 16
  GHS/QoL, Cycle 47 Maintenance: Stable | 26 | 41
  GHS/QoL, Cycle 47 Maintenance: Improved | 17 | 32
  PF, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 87
  PF, Cycle 47 Maintenance: Worsened | 4 | 17
  PF, Cycle 47 Maintenance: Stable | 30 | 49
  PF, Cycle 47 Maintenance: Improved | 14 | 21
  RF, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 87
  RF, Cycle 47 Maintenance: Worsened | 8 | 17
  RF, Cycle 47 Maintenance: Stable | 23 | 38
  RF, Cycle 47 Maintenance: Improved | 17 | 32
  EF, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  EF, Cycle 47 Maintenance: Worsened | 4 | 17
  EF, Cycle 47 Maintenance: Stable | 29 | 48
  EF, Cycle 47 Maintenance: Improved | 15 | 24
  CF, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  CF, Cycle 47 Maintenance: Worsened | 18 | 28
  CF, Cycle 47 Maintenance: Stable | 24 | 48
  CF, Cycle 47 Maintenance: Improved | 6 | 13
  SF, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  SF, Cycle 47 Maintenance: Worsened | 5 | 17
  SF, Cycle 47 Maintenance: Stable | 27 | 38
  SF, Cycle 47 Maintenance: Improved | 16 | 34
  Fatigue, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 88
  Fatigue, Cycle 47 Maintenance: Worsened | 7 | 27
  Fatigue, Cycle 47 Maintenance: Stable | 11 | 21
  Fatigue, Cycle 47 Maintenance: Improved | 30 | 40
  N/V, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  N/V, Cycle 47 Maintenance: Worsened | 9 | 14
  N/V, Cycle 47 Maintenance: Stable | 32 | 57
  N/V, Cycle 47 Maintenance: Improved | 7 | 18
  Pain, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  Pain, Cycle 47 Maintenance: Worsened | 11 | 25
  Pain, Cycle 47 Maintenance: Stable | 18 | 39
  Pain, Cycle 47 Maintenance: Improved | 19 | 25
  Dyspnoea, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  Dyspnoea, Cycle 47 Maintenance: Worsened | 6 | 20
  Dyspnoea, Cycle 47 Maintenance: Stable | 34 | 58
  Dyspnoea, Cycle 47 Maintenance: Improved | 8 | 11
  Insomnia, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  Insomnia, Cycle 47 Maintenance: Worsened | 11 | 25
  Insomnia, Cycle 47 Maintenance: Stable | 23 | 39
  Insomnia, Cycle 47 Maintenance: Improved | 14 | 25
  AL, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  AL, Cycle 47 Maintenance: Worsened | 2 | 12
  AL, Cycle 47 Maintenance: Stable | 37 | 48
  AL, Cycle 47 Maintenance: Improved | 9 | 29
  Constipation, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  Constipation, Cycle 47 Maintenance: Worsened | 13 | 21
  Constipation, Cycle 47 Maintenance: Stable | 25 | 44
  Constipation, Cycle 47 Maintenance: Improved | 10 | 24
  Diarrhoea, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  Diarrhoea, Cycle 47 Maintenance: Worsened | 6 | 8
  Diarrhoea, Cycle 47 Maintenance: Stable | 35 | 66
  Diarrhoea, Cycle 47 Maintenance: Improved | 7 | 15
  FD, Cycle 47 Maintenance: number analyzed (Participants) | 48 | 89
  FD, Cycle 47 Maintenance: Worsened | 6 | 16
  FD, Cycle 47 Maintenance: Stable | 37 | 57
  FD, Cycle 47 Maintenance: Improved | 5 | 16
  GHS/QoL, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  GHS/QoL, Cycle 53 Maintenance: Worsened | 3 | 12
  GHS/QoL, Cycle 53 Maintenance: Stable | 11 | 18
  GHS/QoL, Cycle 53 Maintenance: Improved | 12 | 24
  PF, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  PF, Cycle 53 Maintenance: Worsened | 4 | 11
  PF, Cycle 53 Maintenance: Stable | 11 | 31
  PF, Cycle 53 Maintenance: Improved | 11 | 12
  RF, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  RF, Cycle 53 Maintenance: Worsened | 5 | 16
  RF, Cycle 53 Maintenance: Stable | 11 | 22
  RF, Cycle 53 Maintenance: Improved | 10 | 16
  EF, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  EF, Cycle 53 Maintenance: Worsened | 3 | 15
  EF, Cycle 53 Maintenance: Stable | 17 | 23
  EF, Cycle 53 Maintenance: Improved | 6 | 16
  CF, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  CF, Cycle 53 Maintenance: Worsened | 10 | 19
  CF, Cycle 53 Maintenance: Stable | 13 | 25
  CF, Cycle 53 Maintenance: Improved | 3 | 10
  SF, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  SF, Cycle 53 Maintenance: Worsened | 7 | 11
  SF, Cycle 53 Maintenance: Stable | 12 | 23
  SF, Cycle 53 Maintenance: Improved | 7 | 20
  Fatigue, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  Fatigue, Cycle 53 Maintenance: Worsened | 3 | 14
  Fatigue, Cycle 53 Maintenance: Stable | 7 | 18
  Fatigue, Cycle 53 Maintenance: Improved | 16 | 22
  N/V, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  N/V, Cycle 53 Maintenance: Worsened | 3 | 7
  N/V, Cycle 53 Maintenance: Stable | 19 | 36
  N/V, Cycle 53 Maintenance: Improved | 4 | 11
  Pain, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  Pain, Cycle 53 Maintenance: Worsened | 4 | 14
  Pain, Cycle 53 Maintenance: Stable | 12 | 27
  Pain, Cycle 53 Maintenance: Improved | 10 | 13
  Dyspnoea, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  Dyspnoea, Cycle 53 Maintenance: Worsened | 3 | 12
  Dyspnoea, Cycle 53 Maintenance: Stable | 18 | 35
  Dyspnoea, Cycle 53 Maintenance: Improved | 5 | 7
  Insomnia, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  Insomnia, Cycle 53 Maintenance: Worsened | 8 | 12
  Insomnia, Cycle 53 Maintenance: Stable | 13 | 29
  Insomnia, Cycle 53 Maintenance: Improved | 5 | 13
  AL, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  AL, Cycle 53 Maintenance: Worsened | 2 | 7
  AL, Cycle 53 Maintenance: Stable | 22 | 32
  AL, Cycle 53 Maintenance: Improved | 2 | 15
  Constipation, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  Constipation, Cycle 53 Maintenance: Worsened | 7 | 9
  Constipation, Cycle 53 Maintenance: Stable | 14 | 30
  Constipation, Cycle 53 Maintenance: Improved | 5 | 15
  Diarrhoea, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  Diarrhoea, Cycle 53 Maintenance: Worsened | 2 | 5
  Diarrhoea, Cycle 53 Maintenance: Stable | 20 | 43
  Diarrhoea, Cycle 53 Maintenance: Improved | 4 | 6
  FD, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  FD, Cycle 53 Maintenance: Worsened | 6 | 10
  FD, Cycle 53 Maintenance: Stable | 16 | 36
  FD, Cycle 53 Maintenance: Improved | 4 | 8
  GHS/QoL, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  GHS/QoL, Cycle 59 Maintenance: Worsened | 1 | 3
  GHS/QoL, Cycle 59 Maintenance: Stable | 11 | 12
  GHS/QoL, Cycle 59 Maintenance: Improved | 6 | 21
  PF, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  PF, Cycle 59 Maintenance: Worsened | 3 | 9
  PF, Cycle 59 Maintenance: Stable | 8 | 18
  PF, Cycle 59 Maintenance: Improved | 7 | 9
  RF, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  RF, Cycle 59 Maintenance: Worsened | 3 | 8
  RF, Cycle 59 Maintenance: Stable | 8 | 18
  RF, Cycle 59 Maintenance: Improved | 7 | 10
  EF, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  EF, Cycle 59 Maintenance: Worsened | 4 | 6
  EF, Cycle 59 Maintenance: Stable | 11 | 18
  EF, Cycle 59 Maintenance: Improved | 3 | 12
  CF, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  CF, Cycle 59 Maintenance: Worsened | 5 | 13
  CF, Cycle 59 Maintenance: Stable | 11 | 14
  CF, Cycle 59 Maintenance: Improved | 2 | 9
  SF, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  SF, Cycle 59 Maintenance: Worsened | 4 | 6
  SF, Cycle 59 Maintenance: Stable | 10 | 12
  SF, Cycle 59 Maintenance: Improved | 4 | 18
  Fatigue, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  Fatigue, Cycle 59 Maintenance: Worsened | 4 | 7
  Fatigue, Cycle 59 Maintenance: Stable | 8 | 10
  Fatigue, Cycle 59 Maintenance: Improved | 6 | 19
  N/V, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  N/V, Cycle 59 Maintenance: Worsened | 4 | 6
  N/V, Cycle 59 Maintenance: Stable | 12 | 21
  N/V, Cycle 59 Maintenance: Improved | 2 | 9
  Pain, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  Pain, Cycle 59 Maintenance: Worsened | 1 | 6
  Pain, Cycle 59 Maintenance: Stable | 10 | 21
  Pain, Cycle 59 Maintenance: Improved | 7 | 9
  Dyspnoea, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  Dyspnoea, Cycle 59 Maintenance: Worsened | 2 | 9
  Dyspnoea, Cycle 59 Maintenance: Stable | 12 | 24
  Dyspnoea, Cycle 59 Maintenance: Improved | 4 | 3
  Insomnia, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  Insomnia, Cycle 59 Maintenance: Worsened | 6 | 6
  Insomnia, Cycle 59 Maintenance: Stable | 10 | 15
  Insomnia, Cycle 59 Maintenance: Improved | 2 | 15
  AL, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  AL, Cycle 59 Maintenance: Worsened | 1 | 3
  AL, Cycle 59 Maintenance: Stable | 16 | 21
  AL, Cycle 59 Maintenance: Improved | 1 | 12
  Constipation, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  Constipation, Cycle 59 Maintenance: Worsened | 5 | 8
  Constipation, Cycle 59 Maintenance: Stable | 12 | 20
  Constipation, Cycle 59 Maintenance: Improved | 1 | 8
  Diarrhoea, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  Diarrhoea, Cycle 59 Maintenance: Worsened | 1 | 2
  Diarrhoea, Cycle 59 Maintenance: Stable | 14 | 29
  Diarrhoea, Cycle 59 Maintenance: Improved | 3 | 5
  FD, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 36
  FD, Cycle 59 Maintenance: Worsened | 3 | 4
  FD, Cycle 59 Maintenance: Stable | 11 | 22
  FD, Cycle 59 Maintenance: Improved | 4 | 10
  GHS/QoL, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  GHS/QoL, Cycle 65 Maintenance: Worsened | 1 | 3
  GHS/QoL, Cycle 65 Maintenance: Stable | 7 | 7
  GHS/QoL, Cycle 65 Maintenance: Improved | 4 | 17
  PF, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  PF, Cycle 65 Maintenance: Worsened | 1 | 10
  PF, Cycle 65 Maintenance: Stable | 6 | 12
  PF, Cycle 65 Maintenance: Improved | 5 | 5
  RF, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  RF, Cycle 65 Maintenance: Worsened | 2 | 7
  RF, Cycle 65 Maintenance: Stable | 4 | 11
  RF, Cycle 65 Maintenance: Improved | 6 | 9
  EF, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  EF, Cycle 65 Maintenance: Worsened | 0 | 3
  EF, Cycle 65 Maintenance: Stable | 8 | 16
  EF, Cycle 65 Maintenance: Improved | 4 | 8
  CF, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  CF, Cycle 65 Maintenance: Worsened | 3 | 8
  CF, Cycle 65 Maintenance: Stable | 7 | 13
  CF, Cycle 65 Maintenance: Improved | 2 | 6
  SF, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  SF, Cycle 65 Maintenance: Worsened | 4 | 6
  SF, Cycle 65 Maintenance: Stable | 4 | 8
  SF, Cycle 65 Maintenance: Improved | 4 | 13
  Fatigue, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  Fatigue, Cycle 65 Maintenance: Worsened | 1 | 7
  Fatigue, Cycle 65 Maintenance: Stable | 5 | 8
  Fatigue, Cycle 65 Maintenance: Improved | 6 | 12
  N/V, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  N/V, Cycle 65 Maintenance: Worsened | 1 | 2
  N/V, Cycle 65 Maintenance: Stable | 9 | 19
  N/V, Cycle 65 Maintenance: Improved | 2 | 6
  Pain, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  Pain, Cycle 65 Maintenance: Worsened | 2 | 8
  Pain, Cycle 65 Maintenance: Stable | 7 | 11
  Pain, Cycle 65 Maintenance: Improved | 3 | 8
  Dyspnoea, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  Dyspnoea, Cycle 65 Maintenance: Worsened | 2 | 10
  Dyspnoea, Cycle 65 Maintenance: Stable | 9 | 15
  Dyspnoea, Cycle 65 Maintenance: Improved | 1 | 2
  Insomnia, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  Insomnia, Cycle 65 Maintenance: Worsened | 3 | 7
  Insomnia, Cycle 65 Maintenance: Stable | 7 | 15
  Insomnia, Cycle 65 Maintenance: Improved | 2 | 5
  AL, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  AL, Cycle 65 Maintenance: Worsened | 0 | 1
  AL, Cycle 65 Maintenance: Stable | 11 | 17
  AL, Cycle 65 Maintenance: Improved | 1 | 9
  Constipation, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  Constipation, Cycle 65 Maintenance: Worsened | 6 | 6
  Constipation, Cycle 65 Maintenance: Stable | 5 | 17
  Constipation, Cycle 65 Maintenance: Improved | 1 | 4
  Diarrhoea, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 27
  Diarrhoea, Cycle 65 Maintenance: Worsened | 1 | 1
  Diarrhoea, Cycle 65 Maintenance: Stable | 10 | 22
  Diarrhoea, Cycle 65 Maintenance: Improved | 1 | 4
  FD, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 26
  FD, Cycle 65 Maintenance: Worsened | 1 | 5
  FD, Cycle 65 Maintenance: Stable | 8 | 15
  FD, Cycle 65 Maintenance: Improved | 3 | 6
  GHS/QoL, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  GHS/QoL, Cycle 71 Maintenance: Worsened | 0 | 1
  GHS/QoL, Cycle 71 Maintenance: Stable | 3 | 5
  GHS/QoL, Cycle 71 Maintenance: Improved | 5 | 8
  PF, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  PF, Cycle 71 Maintenance: Worsened | 1 | 4
  PF, Cycle 71 Maintenance: Stable | 4 | 9
  PF, Cycle 71 Maintenance: Improved | 3 | 1
  RF, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  RF, Cycle 71 Maintenance: Worsened | 0 | 4
  RF, Cycle 71 Maintenance: Stable | 4 | 6
  RF, Cycle 71 Maintenance: Improved | 4 | 4
  EF, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  EF, Cycle 71 Maintenance: Worsened | 1 | 3
  EF, Cycle 71 Maintenance: Stable | 6 | 9
  EF, Cycle 71 Maintenance: Improved | 1 | 2
  CF, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  CF, Cycle 71 Maintenance: Worsened | 3 | 3
  CF, Cycle 71 Maintenance: Stable | 5 | 9
  CF, Cycle 71 Maintenance: Improved | 0 | 2
  SF, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  SF, Cycle 71 Maintenance: Worsened | 2 | 4
  SF, Cycle 71 Maintenance: Stable | 2 | 4
  SF, Cycle 71 Maintenance: Improved | 4 | 6
  Fatigue, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  Fatigue, Cycle 71 Maintenance: Worsened | 0 | 3
  Fatigue, Cycle 71 Maintenance: Stable | 3 | 4
  Fatigue, Cycle 71 Maintenance: Improved | 5 | 7
  N/V, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  N/V, Cycle 71 Maintenance: Worsened | 1 | 1
  N/V, Cycle 71 Maintenance: Stable | 5 | 10
  N/V, Cycle 71 Maintenance: Improved | 2 | 3
  Pain, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  Pain, Cycle 71 Maintenance: Worsened | 0 | 2
  Pain, Cycle 71 Maintenance: Stable | 4 | 9
  Pain, Cycle 71 Maintenance: Improved | 4 | 3
  Dyspnoea, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  Dyspnoea, Cycle 71 Maintenance: Worsened | 0 | 1
  Dyspnoea, Cycle 71 Maintenance: Stable | 7 | 12
  Dyspnoea, Cycle 71 Maintenance: Improved | 1 | 1
  Insomnia, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  Insomnia, Cycle 71 Maintenance: Worsened | 2 | 3
  Insomnia, Cycle 71 Maintenance: Stable | 4 | 8
  Insomnia, Cycle 71 Maintenance: Improved | 2 | 3
  AL, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  AL, Cycle 71 Maintenance: Worsened | 0 | 2
  AL, Cycle 71 Maintenance: Stable | 6 | 6
  AL, Cycle 71 Maintenance: Improved | 2 | 6
  Constipation, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  Constipation, Cycle 71 Maintenance: Worsened | 2 | 4
  Constipation, Cycle 71 Maintenance: Stable | 4 | 9
  Constipation, Cycle 71 Maintenance: Improved | 2 | 1
  Diarrhoea, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  Diarrhoea, Cycle 71 Maintenance: Worsened | 0 | 0
  Diarrhoea, Cycle 71 Maintenance: Stable | 7 | 11
  Diarrhoea, Cycle 71 Maintenance: Improved | 1 | 3
  FD, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 14
  FD, Cycle 71 Maintenance: Worsened | 1 | 2
  FD, Cycle 71 Maintenance: Stable | 4 | 12
  FD, Cycle 71 Maintenance: Improved | 3 | 0
  GHS/QoL, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  GHS/QoL, Cycle 77 Maintenance: Worsened | 0 | 0
  GHS/QoL, Cycle 77 Maintenance: Stable | 2 | 3
  GHS/QoL, Cycle 77 Maintenance: Improved | 2 | 8
  PF, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  PF, Cycle 77 Maintenance: Worsened | 0 | 2
  PF, Cycle 77 Maintenance: Stable | 2 | 5
  PF, Cycle 77 Maintenance: Improved | 2 | 4
  RF, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  RF, Cycle 77 Maintenance: Worsened | 0 | 2
  RF, Cycle 77 Maintenance: Stable | 1 | 4
  RF, Cycle 77 Maintenance: Improved | 3 | 5
  EF, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  EF, Cycle 77 Maintenance: Worsened | 1 | 1
  EF, Cycle 77 Maintenance: Stable | 2 | 8
  EF, Cycle 77 Maintenance: Improved | 1 | 2
  CF, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  CF, Cycle 77 Maintenance: Worsened | 2 | 2
  CF, Cycle 77 Maintenance: Stable | 1 | 3
  CF, Cycle 77 Maintenance: Improved | 1 | 6
  SF, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  SF, Cycle 77 Maintenance: Worsened | 1 | 2
  SF, Cycle 77 Maintenance: Stable | 1 | 2
  SF, Cycle 77 Maintenance: Improved | 2 | 7
  Fatigue, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  Fatigue, Cycle 77 Maintenance: Worsened | 0 | 5
  Fatigue, Cycle 77 Maintenance: Stable | 1 | 2
  Fatigue, Cycle 77 Maintenance: Improved | 3 | 4
  N/V, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  N/V, Cycle 77 Maintenance: Worsened | 0 | 2
  N/V, Cycle 77 Maintenance: Stable | 3 | 7
  N/V, Cycle 77 Maintenance: Improved | 1 | 2
  Pain, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  Pain, Cycle 77 Maintenance: Worsened | 0 | 1
  Pain, Cycle 77 Maintenance: Stable | 3 | 5
  Pain, Cycle 77 Maintenance: Improved | 1 | 5
  Dyspnoea, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  Dyspnoea, Cycle 77 Maintenance: Worsened | 0 | 3
  Dyspnoea, Cycle 77 Maintenance: Stable | 3 | 7
  Dyspnoea, Cycle 77 Maintenance: Improved | 1 | 1
  Insomnia, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  Insomnia, Cycle 77 Maintenance: Worsened | 0 | 5
  Insomnia, Cycle 77 Maintenance: Stable | 3 | 4
  Insomnia, Cycle 77 Maintenance: Improved | 1 | 2
  AL, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  AL, Cycle 77 Maintenance: Worsened | 1 | 3
  AL, Cycle 77 Maintenance: Stable | 2 | 4
  AL, Cycle 77 Maintenance: Improved | 1 | 4
  Constipation, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  Constipation, Cycle 77 Maintenance: Worsened | 1 | 1
  Constipation, Cycle 77 Maintenance: Stable | 3 | 8
  Constipation, Cycle 77 Maintenance: Improved | 0 | 2
  Diarrhoea, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  Diarrhoea, Cycle 77 Maintenance: Worsened | 0 | 0
  Diarrhoea, Cycle 77 Maintenance: Stable | 3 | 8
  Diarrhoea, Cycle 77 Maintenance: Improved | 1 | 3
  FD, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  FD, Cycle 77 Maintenance: Worsened | 1 | 1
  FD, Cycle 77 Maintenance: Stable | 2 | 10
  FD, Cycle 77 Maintenance: Improved | 1 | 0
  GHS/QoL, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  GHS/QoL, Cycle 83 Maintenance: Worsened | 0 | 0
  GHS/QoL, Cycle 83 Maintenance: Stable | 1 | 1
  GHS/QoL, Cycle 83 Maintenance: Improved | 2 | 5
  PF, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  PF, Cycle 83 Maintenance: Worsened | 1 | 2
  PF, Cycle 83 Maintenance: Stable | 1 | 1
  PF, Cycle 83 Maintenance: Improved | 1 | 3
  RF, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  RF, Cycle 83 Maintenance: Worsened | 0 | 1
  RF, Cycle 83 Maintenance: Stable | 2 | 2
  RF, Cycle 83 Maintenance: Improved | 1 | 3
  EF, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  EF, Cycle 83 Maintenance: Worsened | 0 | 2
  EF, Cycle 83 Maintenance: Stable | 3 | 3
  EF, Cycle 83 Maintenance: Improved | 0 | 1
  CF, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  CF, Cycle 83 Maintenance: Worsened | 1 | 1
  CF, Cycle 83 Maintenance: Stable | 2 | 3
  CF, Cycle 83 Maintenance: Improved | 0 | 2
  SF, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  SF, Cycle 83 Maintenance: Worsened | 1 | 1
  SF, Cycle 83 Maintenance: Stable | 1 | 1
  SF, Cycle 83 Maintenance: Improved | 1 | 4
  Fatigue, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  Fatigue, Cycle 83 Maintenance: Worsened | 0 | 1
  Fatigue, Cycle 83 Maintenance: Stable | 0 | 1
  Fatigue, Cycle 83 Maintenance: Improved | 3 | 4
  N/V, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  N/V, Cycle 83 Maintenance: Worsened | 1 | 0
  N/V, Cycle 83 Maintenance: Stable | 2 | 4
  N/V, Cycle 83 Maintenance: Improved | 0 | 2
  Pain, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  Pain, Cycle 83 Maintenance: Worsened | 0 | 1
  Pain, Cycle 83 Maintenance: Stable | 2 | 2
  Pain, Cycle 83 Maintenance: Improved | 1 | 3
  Dyspnoea, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  Dyspnoea, Cycle 83 Maintenance: Worsened | 0 | 3
  Dyspnoea, Cycle 83 Maintenance: Stable | 2 | 3
  Dyspnoea, Cycle 83 Maintenance: Improved | 1 | 0
  Insomnia, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  Insomnia, Cycle 83 Maintenance: Worsened | 0 | 2
  Insomnia, Cycle 83 Maintenance: Stable | 3 | 3
  Insomnia, Cycle 83 Maintenance: Improved | 0 | 1
  AL, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  AL, Cycle 83 Maintenance: Worsened | 0 | 1
  AL, Cycle 83 Maintenance: Stable | 3 | 2
  AL, Cycle 83 Maintenance: Improved | 0 | 3
  Constipation, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  Constipation, Cycle 83 Maintenance: Worsened | 2 | 0
  Constipation, Cycle 83 Maintenance: Stable | 0 | 6
  Constipation, Cycle 83 Maintenance: Improved | 1 | 0
  Diarrhoea, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  Diarrhoea, Cycle 83 Maintenance: Worsened | 0 | 0
  Diarrhoea, Cycle 83 Maintenance: Stable | 3 | 5
  Diarrhoea, Cycle 83 Maintenance: Improved | 0 | 1
  FD, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 6
  FD, Cycle 83 Maintenance: Worsened | 1 | 0
  FD, Cycle 83 Maintenance: Stable | 1 | 5
  FD, Cycle 83 Maintenance: Improved | 1 | 1
  GHS/QoL, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  GHS/QoL, Cycle 89 Maintenance: Worsened | 0 | 0
  GHS/QoL, Cycle 89 Maintenance: Stable | 0 | 0
  GHS/QoL, Cycle 89 Maintenance: Improved | 0 | 2
  PF, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  PF, Cycle 89 Maintenance: Worsened | 0 | 0
  PF, Cycle 89 Maintenance: Stable | 0 | 0
  PF, Cycle 89 Maintenance: Improved | 0 | 2
  RF, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  RF, Cycle 89 Maintenance: Worsened | 0 | 0
  RF, Cycle 89 Maintenance: Stable | 0 | 2
  RF, Cycle 89 Maintenance: Improved | 0 | 0
  EF, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  EF, Cycle 89 Maintenance: Worsened | 0 | 0
  EF, Cycle 89 Maintenance: Stable | 0 | 2
  EF, Cycle 89 Maintenance: Improved | 0 | 0
  CF, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  CF, Cycle 89 Maintenance: Worsened | 0 | 0
  CF, Cycle 89 Maintenance: Stable | 0 | 1
  CF, Cycle 89 Maintenance: Improved | 0 | 1
  SF, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  SF, Cycle 89 Maintenance: Worsened | 0 | 0
  SF, Cycle 89 Maintenance: Stable | 0 | 1
  SF, Cycle 89 Maintenance: Improved | 0 | 1
  Fatigue, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  Fatigue, Cycle 89 Maintenance: Worsened | 0 | 0
  Fatigue, Cycle 89 Maintenance: Stable | 0 | 0
  Fatigue, Cycle 89 Maintenance: Improved | 0 | 2
  N/V, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  N/V, Cycle 89 Maintenance: Worsened | 0 | 0
  N/V, Cycle 89 Maintenance: Stable | 0 | 1
  N/V, Cycle 89 Maintenance: Improved | 0 | 1
  Pain, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  Pain, Cycle 89 Maintenance: Worsened | 0 | 0
  Pain, Cycle 89 Maintenance: Stable | 0 | 1
  Pain, Cycle 89 Maintenance: Improved | 0 | 1
  Dyspnoea, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  Dyspnoea, Cycle 89 Maintenance: Worsened | 0 | 0
  Dyspnoea, Cycle 89 Maintenance: Stable | 0 | 2
  Dyspnoea, Cycle 89 Maintenance: Improved | 0 | 0
  Insomnia, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  Insomnia, Cycle 89 Maintenance: Worsened | 0 | 0
  Insomnia, Cycle 89 Maintenance: Stable | 0 | 2
  Insomnia, Cycle 89 Maintenance: Improved | 0 | 0
  AL, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  AL, Cycle 89 Maintenance: Worsened | 0 | 0
  AL, Cycle 89 Maintenance: Stable | 0 | 0
  AL, Cycle 89 Maintenance: Improved | 0 | 2
  Constipation, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  Constipation, Cycle 89 Maintenance: Worsened | 0 | 0
  Constipation, Cycle 89 Maintenance: Stable | 0 | 2
  Constipation, Cycle 89 Maintenance: Improved | 0 | 0
  Diarrhoea, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  Diarrhoea, Cycle 89 Maintenance: Worsened | 0 | 0
  Diarrhoea, Cycle 89 Maintenance: Stable | 0 | 2
  Diarrhoea, Cycle 89 Maintenance: Improved | 0 | 0
  FD, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  FD, Cycle 89 Maintenance: Worsened | 0 | 0
  FD, Cycle 89 Maintenance: Stable | 0 | 1
  FD, Cycle 89 Maintenance: Improved | 0 | 1
  GHS/QoL, End of treatment (EOT): number analyzed (Participants) | 184 | 345
  GHS/QoL, End of treatment (EOT): Worsened | 50 | 111
  GHS/QoL, End of treatment (EOT): Stable | 81 | 150
  GHS/QoL, End of treatment (EOT): Improved | 53 | 84
  PF, EOT: number analyzed (Participants) | 183 | 342
  PF, EOT: Worsened | 44 | 84
  PF, EOT: Stable | 80 | 161
  PF, EOT: Improved | 59 | 97
  RF, EOT: number analyzed (Participants) | 183 | 342
  RF, EOT: Worsened | 57 | 102
  RF, EOT: Stable | 64 | 115
  RF, EOT: Improved | 62 | 125
  EF, EOT: number analyzed (Participants) | 184 | 345
  EF, EOT: Worsened | 67 | 133
  EF, EOT: Stable | 92 | 161
  EF, EOT: Improved | 25 | 51
  CF, EOT: number analyzed (Participants) | 184 | 345
  CF, EOT: Worsened | 68 | 127
  CF, EOT: Stable | 92 | 155
  CF, EOT: Improved | 24 | 63
  SF, EOT: number analyzed (Participants) | 184 | 345
  SF, EOT: Worsened | 58 | 119
  SF, EOT: Stable | 68 | 118
  SF, EOT: Improved | 58 | 108
  Fatigue, EOT: number analyzed (Participants) | 184 | 344
  Fatigue, EOT: Worsened | 66 | 124
  Fatigue, EOT: Stable | 45 | 80
  Fatigue, EOT: Improved | 73 | 140
  N/V, EOT: number analyzed (Participants) | 184 | 344
  N/V, EOT: Worsened | 38 | 72
  N/V, EOT: Stable | 117 | 204
  N/V, EOT: Improved | 29 | 68
  Pain, EOT: number analyzed (Participants) | 184 | 345
  Pain, EOT: Worsened | 66 | 95
  Pain, EOT: Stable | 50 | 140
  Pain, EOT: Improved | 68 | 110
  Dyspnoea, EOT: number analyzed (Participants) | 184 | 342
  Dyspnoea, EOT: Worsened | 47 | 97
  Dyspnoea, EOT: Stable | 109 | 185
  Dyspnoea, EOT: Improved | 28 | 60
  Insomnia, EOT: number analyzed (Participants) | 184 | 344
  Insomnia, EOT: Worsened | 47 | 91
  Insomnia, EOT: Stable | 81 | 160
  Insomnia, EOT: Improved | 56 | 93
  AL, EOT: number analyzed (Participants) | 183 | 343
  AL, EOT: Worsened | 40 | 74
  AL, EOT: Stable | 94 | 188
  AL, EOT: Improved | 49 | 81
  Constipation, EOT: number analyzed (Participants) | 183 | 343
  Constipation, EOT: Worsened | 44 | 73
  Constipation, EOT: Stable | 89 | 172
  Constipation, EOT: Improved | 50 | 98
  Diarrhoea, EOT: number analyzed (Participants) | 184 | 345
  Diarrhoea, EOT: Worsened | 24 | 61
  Diarrhoea, EOT: Stable | 127 | 225
  Diarrhoea, EOT: Improved | 33 | 59
  FD, EOT: number analyzed (Participants) | 183 | 343
  FD, EOT: Worsened | 28 | 59
  FD, EOT: Stable | 130 | 239
  FD, EOT: Improved | 25 | 45
  GHS/QoL, Safety Follow-up: number analyzed (Participants) | 146 | 290
  GHS/QoL, Safety Follow-up: Worsened | 36 | 97
  GHS/QoL, Safety Follow-up: Stable | 71 | 130
  GHS/QoL, Safety Follow-up: Improved | 39 | 63
  PF, Safety Follow-up: number analyzed (Participants) | 146 | 287
  PF, Safety Follow-up: Worsened | 40 | 80
  PF, Safety Follow-up: Stable | 66 | 129
  PF, Safety Follow-up: Improved | 40 | 78
  RF, Safety Follow-up: number analyzed (Participants) | 146 | 288
  RF, Safety Follow-up: Worsened | 46 | 99
  RF, Safety Follow-up: Stable | 55 | 87
  RF, Safety Follow-up: Improved | 45 | 102
  EF, Safety Follow-up: number analyzed (Participants) | 146 | 290
  EF, Safety Follow-up: Worsened | 44 | 107
  EF, Safety Follow-up: Stable | 72 | 147
  EF, Safety Follow-up: Improved | 30 | 36
  CF, Safety Follow-up: number analyzed (Participants) | 146 | 290
  CF, Safety Follow-up: Worsened | 56 | 112
  CF, Safety Follow-up: Stable | 69 | 119
  CF, Safety Follow-up: Improved | 21 | 59
  SF, Safety Follow-up: number analyzed (Participants) | 146 | 290
  SF, Safety Follow-up: Worsened | 42 | 105
  SF, Safety Follow-up: Stable | 59 | 105
  SF, Safety Follow-up: Improved | 45 | 80
  Fatigue, Safety Follow-up: number analyzed (Participants) | 146 | 290
  Fatigue, Safety Follow-up: Worsened | 54 | 109
  Fatigue, Safety Follow-up: Stable | 31 | 75
  Fatigue, Safety Follow-up: Improved | 61 | 106
  N/V, Safety Follow-up: number analyzed (Participants) | 146 | 290
  N/V, Safety Follow-up: Worsened | 34 | 65
  N/V, Safety Follow-up: Stable | 92 | 169
  N/V, Safety Follow-up: Improved | 20 | 56
  Pain, Safety Follow-up: number analyzed (Participants) | 146 | 290
  Pain, Safety Follow-up: Worsened | 50 | 108
  Pain, Safety Follow-up: Stable | 47 | 101
  Pain, Safety Follow-up: Improved | 49 | 81
  Dyspnoea, Safety Follow-up: number analyzed (Participants) | 146 | 290
  Dyspnoea, Safety Follow-up: Worsened | 36 | 84
  Dyspnoea, Safety Follow-up: Stable | 91 | 158
  Dyspnoea, Safety Follow-up: Improved | 19 | 48
  Insomnia, Safety Follow-up: number analyzed (Participants) | 146 | 290
  Insomnia, Safety Follow-up: Worsened | 22 | 79
  Insomnia, Safety Follow-up: Stable | 75 | 132
  Insomnia, Safety Follow-up: Improved | 49 | 79
  AL, Safety Follow-up: number analyzed (Participants) | 146 | 289
  AL, Safety Follow-up: Worsened | 28 | 74
  AL, Safety Follow-up: Stable | 81 | 140
  AL, Safety Follow-up: Improved | 37 | 75
  Constipation, Safety Follow-up: number analyzed (Participants) | 145 | 290
  Constipation, Safety Follow-up: Worsened | 32 | 56
  Constipation, Safety Follow-up: Stable | 72 | 153
  Constipation, Safety Follow-up: Improved | 41 | 81
  Diarrhoea, Safety Follow-up: number analyzed (Participants) | 145 | 290
  Diarrhoea, Safety Follow-up: Worsened | 21 | 58
  Diarrhoea, Safety Follow-up: Stable | 97 | 184
  Diarrhoea, Safety Follow-up: Improved | 27 | 48
  FD, Safety Follow-up: number analyzed (Participants) | 145 | 287
  FD, Safety Follow-up: Worsened | 19 | 46
  FD, Safety Follow-up: Stable | 114 | 199
  FD, Safety Follow-up: Improved | 12 | 42
  GHS/QoL, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  GHS/QoL, LTFU (EOT + 3 months): Worsened | 39 | 84
  GHS/QoL, LTFU (EOT + 3 months): Stable | 53 | 97
  GHS/QoL, LTFU (EOT + 3 months): Improved | 43 | 69
  PF, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  PF, LTFU (EOT + 3 months): Worsened | 42 | 80
  PF, LTFU (EOT + 3 months): Stable | 66 | 100
  PF, LTFU (EOT + 3 months): Improved | 27 | 70
  RF, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 249
  RF, LTFU (EOT + 3 months): Worsened | 52 | 70
  RF, LTFU (EOT + 3 months): Stable | 42 | 84
  RF, LTFU (EOT + 3 months): Improved | 41 | 95
  EF, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  EF, LTFU (EOT + 3 months): Worsened | 30 | 76
  EF, LTFU (EOT + 3 months): Stable | 76 | 129
  EF, LTFU (EOT + 3 months): Improved | 29 | 45
  CF, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  CF, LTFU (EOT + 3 months): Worsened | 55 | 96
  CF, LTFU (EOT + 3 months): Stable | 64 | 110
  CF, LTFU (EOT + 3 months): Improved | 16 | 44
  SF, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  SF, LTFU (EOT + 3 months): Worsened | 48 | 80
  SF, LTFU (EOT + 3 months): Stable | 51 | 91
  SF, LTFU (EOT + 3 months): Improved | 36 | 79
  Fatigue, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  Fatigue, LTFU (EOT + 3 months): Worsened | 52 | 98
  Fatigue, LTFU (EOT + 3 months): Stable | 28 | 58
  Fatigue, LTFU (EOT + 3 months): Improved | 55 | 94
  N/V, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  N/V, LTFU (EOT + 3 months): Worsened | 20 | 45
  N/V, LTFU (EOT + 3 months): Stable | 88 | 155
  N/V, LTFU (EOT + 3 months): Improved | 27 | 50
  Pain, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  Pain, LTFU (EOT + 3 months): Worsened | 41 | 89
  Pain, LTFU (EOT + 3 months): Stable | 42 | 87
  Pain, LTFU (EOT + 3 months): Improved | 52 | 74
  Dyspnoea, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  Dyspnoea, LTFU (EOT + 3 months): Worsened | 33 | 71
  Dyspnoea, LTFU (EOT + 3 months): Stable | 84 | 141
  Dyspnoea, LTFU (EOT + 3 months): Improved | 18 | 38
  Insomnia, LTFU (EOT + 3 months): number analyzed (Participants) | 134 | 250
  Insomnia, LTFU (EOT + 3 months): Worsened | 28 | 58
  Insomnia, LTFU (EOT + 3 months): Stable | 66 | 111
  Insomnia, LTFU (EOT + 3 months): Improved | 40 | 81
  AL, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 249
  AL, LTFU (EOT + 3 months): Worsened | 25 | 48
  AL, LTFU (EOT + 3 months): Stable | 75 | 130
  AL, LTFU (EOT + 3 months): Improved | 35 | 71
  Constipation, LTFU (EOT + 3 months): number analyzed (Participants) | 134 | 250
  Constipation, LTFU (EOT + 3 months): Worsened | 25 | 53
  Constipation, LTFU (EOT + 3 months): Stable | 64 | 128
  Constipation, LTFU (EOT + 3 months): Improved | 45 | 69
  Diarrhoea, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  Diarrhoea, LTFU (EOT + 3 months): Worsened | 20 | 52
  Diarrhoea, LTFU (EOT + 3 months): Stable | 89 | 157
  Diarrhoea, LTFU (EOT + 3 months): Improved | 26 | 41
  FD, LTFU (EOT + 3 months): number analyzed (Participants) | 135 | 250
  FD, LTFU (EOT + 3 months): Worsened | 24 | 43
  FD, LTFU (EOT + 3 months): Stable | 90 | 169
  FD, LTFU (EOT + 3 months): Improved | 21 | 38
  GHS/QoL, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 184
  GHS/QoL, LTFU (EOT + 9 months): Worsened | 24 | 60
  GHS/QoL, LTFU (EOT + 9 months): Stable | 53 | 77
  GHS/QoL, LTFU (EOT + 9 months): Improved | 29 | 47
  PF, LTFU (EOT + 9 months): number analyzed (Participants) | 105 | 184
  PF, LTFU (EOT + 9 months): Worsened | 32 | 56
  PF, LTFU (EOT + 9 months): Stable | 59 | 83
  PF, LTFU (EOT + 9 months): Improved | 14 | 45
  RF, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 184
  RF, LTFU (EOT + 9 months): Worsened | 37 | 63
  RF, LTFU (EOT + 9 months): Stable | 37 | 59
  RF, LTFU (EOT + 9 months): Improved | 32 | 62
  EF, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 184
  EF, LTFU (EOT + 9 months): Worsened | 31 | 53
  EF, LTFU (EOT + 9 months): Stable | 57 | 97
  EF, LTFU (EOT + 9 months): Improved | 18 | 34
  CF, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 184
  CF, LTFU (EOT + 9 months): Worsened | 42 | 65
  CF, LTFU (EOT + 9 months): Stable | 55 | 89
  CF, LTFU (EOT + 9 months): Improved | 9 | 30
  SF, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 184
  SF, LTFU (EOT + 9 months): Worsened | 40 | 62
  SF, LTFU (EOT + 9 months): Stable | 37 | 69
  SF, LTFU (EOT + 9 months): Improved | 29 | 53
  Fatigue, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 183
  Fatigue, LTFU (EOT + 9 months): Worsened | 43 | 73
  Fatigue, LTFU (EOT + 9 months): Stable | 22 | 46
  Fatigue, LTFU (EOT + 9 months): Improved | 41 | 64
  N/V, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 183
  N/V, LTFU (EOT + 9 months): Worsened | 21 | 40
  N/V, LTFU (EOT + 9 months): Stable | 68 | 112
  N/V, LTFU (EOT + 9 months): Improved | 17 | 31
  Pain, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 184
  Pain, LTFU (EOT + 9 months): Worsened | 33 | 70
  Pain, LTFU (EOT + 9 months): Stable | 46 | 59
  Pain, LTFU (EOT + 9 months): Improved | 27 | 55
  Dyspnoea, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 182
  Dyspnoea, LTFU (EOT + 9 months): Worsened | 34 | 48
  Dyspnoea, LTFU (EOT + 9 months): Stable | 59 | 103
  Dyspnoea, LTFU (EOT + 9 months): Improved | 13 | 31
  Insomnia, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 183
  Insomnia, LTFU (EOT + 9 months): Worsened | 24 | 44
  Insomnia, LTFU (EOT + 9 months): Stable | 55 | 82
  Insomnia, LTFU (EOT + 9 months): Improved | 27 | 57
  AL, LTFU (EOT + 9 months): number analyzed (Participants) | 105 | 182
  AL, LTFU (EOT + 9 months): Worsened | 21 | 45
  AL, LTFU (EOT + 9 months): Stable | 59 | 93
  AL, LTFU (EOT + 9 months): Improved | 25 | 44
  Constipation, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 182
  Constipation, LTFU (EOT + 9 months): Worsened | 23 | 43
  Constipation, LTFU (EOT + 9 months): Stable | 50 | 85
  Constipation, LTFU (EOT + 9 months): Improved | 33 | 54
  Diarrhoea, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 184
  Diarrhoea, LTFU (EOT + 9 months): Worsened | 21 | 35
  Diarrhoea, LTFU (EOT + 9 months): Stable | 65 | 122
  Diarrhoea, LTFU (EOT + 9 months): Improved | 20 | 27
  FD, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 183
  FD, LTFU (EOT + 9 months): Worsened | 18 | 26
  FD, LTFU (EOT + 9 months): Stable | 67 | 129
  FD, LTFU (EOT + 9 months): Improved | 21 | 28
  GHS/QoL, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 153
  GHS/QoL, LTFU (EOT + 15 months): Worsened | 23 | 48
  GHS/QoL, LTFU (EOT + 15 months): Stable | 34 | 66
  GHS/QoL, LTFU (EOT + 15 months): Improved | 19 | 39
  PF, LTFU (EOT + 15 months): number analyzed (Participants) | 74 | 154
  PF, LTFU (EOT + 15 months): Worsened | 23 | 44
  PF, LTFU (EOT + 15 months): Stable | 38 | 71
  PF, LTFU (EOT + 15 months): Improved | 13 | 39
  RF, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  RF, LTFU (EOT + 15 months): Worsened | 29 | 46
  RF, LTFU (EOT + 15 months): Stable | 22 | 66
  RF, LTFU (EOT + 15 months): Improved | 25 | 42
  EF, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  EF, LTFU (EOT + 15 months): Worsened | 23 | 40
  EF, LTFU (EOT + 15 months): Stable | 42 | 86
  EF, LTFU (EOT + 15 months): Improved | 11 | 28
  CF, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  CF, LTFU (EOT + 15 months): Worsened | 23 | 55
  CF, LTFU (EOT + 15 months): Stable | 43 | 70
  CF, LTFU (EOT + 15 months): Improved | 10 | 29
  SF, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 153
  SF, LTFU (EOT + 15 months): Worsened | 31 | 51
  SF, LTFU (EOT + 15 months): Stable | 23 | 58
  SF, LTFU (EOT + 15 months): Improved | 22 | 44
  Fatigue, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  Fatigue, LTFU (EOT + 15 months): Worsened | 29 | 63
  Fatigue, LTFU (EOT + 15 months): Stable | 14 | 39
  Fatigue, LTFU (EOT + 15 months): Improved | 33 | 52
  N/V, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  N/V, LTFU (EOT + 15 months): Worsened | 19 | 30
  N/V, LTFU (EOT + 15 months): Stable | 49 | 101
  N/V, LTFU (EOT + 15 months): Improved | 8 | 23
  Pain, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  Pain, LTFU (EOT + 15 months): Worsened | 21 | 61
  Pain, LTFU (EOT + 15 months): Stable | 30 | 54
  Pain, LTFU (EOT + 15 months): Improved | 25 | 39
  Dyspnoea, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  Dyspnoea, LTFU (EOT + 15 months): Worsened | 24 | 47
  Dyspnoea, LTFU (EOT + 15 months): Stable | 43 | 82
  Dyspnoea, LTFU (EOT + 15 months): Improved | 9 | 25
  Insomnia, LTFU (EOT + 15 months): number analyzed (Participants) | 75 | 154
  Insomnia, LTFU (EOT + 15 months): Worsened | 19 | 35
  Insomnia, LTFU (EOT + 15 months): Stable | 32 | 71
  Insomnia, LTFU (EOT + 15 months): Improved | 24 | 48
  AL, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 153
  AL, LTFU (EOT + 15 months): Worsened | 13 | 27
  AL, LTFU (EOT + 15 months): Stable | 40 | 87
  AL, LTFU (EOT + 15 months): Improved | 23 | 39
  Constipation, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  Constipation, LTFU (EOT + 15 months): Worsened | 20 | 32
  Constipation, LTFU (EOT + 15 months): Stable | 35 | 73
  Constipation, LTFU (EOT + 15 months): Improved | 21 | 49
  Diarrhoea, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 154
  Diarrhoea, LTFU (EOT + 15 months): Worsened | 12 | 23
  Diarrhoea, LTFU (EOT + 15 months): Stable | 52 | 103
  Diarrhoea, LTFU (EOT + 15 months): Improved | 12 | 28
  FD, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 153
  FD, LTFU (EOT + 15 months): Worsened | 9 | 26
  FD, LTFU (EOT + 15 months): Stable | 54 | 105
  FD, LTFU (EOT + 15 months): Improved | 13 | 22
  GHS/QoL, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  GHS/QoL, LTFU (EOT + 21 months): Worsened | 19 | 36
  GHS/QoL, LTFU (EOT + 21 months): Stable | 14 | 37
  GHS/QoL, LTFU (EOT + 21 months): Improved | 15 | 26
  PF, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 98
  PF, LTFU (EOT + 21 months): Worsened | 15 | 33
  PF, LTFU (EOT + 21 months): Stable | 25 | 41
  PF, LTFU (EOT + 21 months): Improved | 8 | 24
  RF, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  RF, LTFU (EOT + 21 months): Worsened | 15 | 35
  RF, LTFU (EOT + 21 months): Stable | 16 | 30
  RF, LTFU (EOT + 21 months): Improved | 17 | 34
  EF, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  EF, LTFU (EOT + 21 months): Worsened | 16 | 27
  EF, LTFU (EOT + 21 months): Stable | 28 | 44
  EF, LTFU (EOT + 21 months): Improved | 4 | 28
  CF, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  CF, LTFU (EOT + 21 months): Worsened | 18 | 40
  CF, LTFU (EOT + 21 months): Stable | 24 | 39
  CF, LTFU (EOT + 21 months): Improved | 6 | 20
  SF, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  SF, LTFU (EOT + 21 months): Worsened | 13 | 43
  SF, LTFU (EOT + 21 months): Stable | 20 | 32
  SF, LTFU (EOT + 21 months): Improved | 15 | 24
  Fatigue, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  Fatigue, LTFU (EOT + 21 months): Worsened | 22 | 42
  Fatigue, LTFU (EOT + 21 months): Stable | 9 | 26
  Fatigue, LTFU (EOT + 21 months): Improved | 17 | 31
  N/V, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  N/V, LTFU (EOT + 21 months): Worsened | 13 | 23
  N/V, LTFU (EOT + 21 months): Stable | 28 | 61
  N/V, LTFU (EOT + 21 months): Improved | 7 | 15
  Pain, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  Pain, LTFU (EOT + 21 months): Worsened | 16 | 34
  Pain, LTFU (EOT + 21 months): Stable | 14 | 34
  Pain, LTFU (EOT + 21 months): Improved | 18 | 31
  Dyspnoea, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  Dyspnoea, LTFU (EOT + 21 months): Worsened | 18 | 27
  Dyspnoea, LTFU (EOT + 21 months): Stable | 24 | 58
  Dyspnoea, LTFU (EOT + 21 months): Improved | 6 | 14
  Insomnia, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  Insomnia, LTFU (EOT + 21 months): Worsened | 14 | 25
  Insomnia, LTFU (EOT + 21 months): Stable | 22 | 41
  Insomnia, LTFU (EOT + 21 months): Improved | 12 | 33
  AL, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  AL, LTFU (EOT + 21 months): Worsened | 11 | 21
  AL, LTFU (EOT + 21 months): Stable | 24 | 56
  AL, LTFU (EOT + 21 months): Improved | 13 | 22
  Constipation, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  Constipation, LTFU (EOT + 21 months): Worsened | 8 | 27
  Constipation, LTFU (EOT + 21 months): Stable | 22 | 45
  Constipation, LTFU (EOT + 21 months): Improved | 18 | 27
  Diarrhoea, LTFU (EOT + 21 months): number analyzed (Participants) | 48 | 99
  Diarrhoea, LTFU (EOT + 21 months): Worsened | 12 | 17
  Diarrhoea, LTFU (EOT + 21 months): Stable | 32 | 62
  Diarrhoea, LTFU (EOT + 21 months): Improved | 4 | 20
  FD, LTFU (EOT + 21 months): number analyzed (Participants) | 47 | 99
  FD, LTFU (EOT + 21 months): Worsened | 5 | 18
  FD, LTFU (EOT + 21 months): Stable | 33 | 68
  FD, LTFU (EOT + 21 months): Improved | 9 | 13
  GHS/QoL, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  GHS/QoL, LTFU (EOT + 27 months): Worsened | 9 | 17
  GHS/QoL, LTFU (EOT + 27 months): Stable | 15 | 32
  GHS/QoL, LTFU (EOT + 27 months): Improved | 12 | 21
  PF, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  PF, LTFU (EOT + 27 months): Worsened | 13 | 22
  PF, LTFU (EOT + 27 months): Stable | 16 | 32
  PF, LTFU (EOT + 27 months): Improved | 7 | 16
  RF, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  RF, LTFU (EOT + 27 months): Worsened | 9 | 20
  RF, LTFU (EOT + 27 months): Stable | 13 | 22
  RF, LTFU (EOT + 27 months): Improved | 14 | 28
  EF, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  EF, LTFU (EOT + 27 months): Worsened | 9 | 20
  EF, LTFU (EOT + 27 months): Stable | 21 | 31
  EF, LTFU (EOT + 27 months): Improved | 6 | 19
  CF, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  CF, LTFU (EOT + 27 months): Worsened | 12 | 27
  CF, LTFU (EOT + 27 months): Stable | 16 | 28
  CF, LTFU (EOT + 27 months): Improved | 8 | 15
  SF, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  SF, LTFU (EOT + 27 months): Worsened | 14 | 28
  SF, LTFU (EOT + 27 months): Stable | 11 | 21
  SF, LTFU (EOT + 27 months): Improved | 11 | 21
  Fatigue, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  Fatigue, LTFU (EOT + 27 months): Worsened | 14 | 25
  Fatigue, LTFU (EOT + 27 months): Stable | 7 | 18
  Fatigue, LTFU (EOT + 27 months): Improved | 15 | 27
  N/V, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  N/V, LTFU (EOT + 27 months): Worsened | 7 | 12
  N/V, LTFU (EOT + 27 months): Stable | 25 | 46
  N/V, LTFU (EOT + 27 months): Improved | 4 | 12
  Pain, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  Pain, LTFU (EOT + 27 months): Worsened | 9 | 28
  Pain, LTFU (EOT + 27 months): Stable | 13 | 18
  Pain, LTFU (EOT + 27 months): Improved | 14 | 24
  Dyspnoea, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  Dyspnoea, LTFU (EOT + 27 months): Worsened | 11 | 17
  Dyspnoea, LTFU (EOT + 27 months): Stable | 19 | 43
  Dyspnoea, LTFU (EOT + 27 months): Improved | 6 | 10
  Insomnia, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  Insomnia, LTFU (EOT + 27 months): Worsened | 8 | 16
  Insomnia, LTFU (EOT + 27 months): Stable | 18 | 31
  Insomnia, LTFU (EOT + 27 months): Improved | 10 | 23
  AL, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  AL, LTFU (EOT + 27 months): Worsened | 9 | 13
  AL, LTFU (EOT + 27 months): Stable | 16 | 44
  AL, LTFU (EOT + 27 months): Improved | 11 | 13
  Constipation, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  Constipation, LTFU (EOT + 27 months): Worsened | 5 | 15
  Constipation, LTFU (EOT + 27 months): Stable | 17 | 33
  Constipation, LTFU (EOT + 27 months): Improved | 14 | 22
  Diarrhoea, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  Diarrhoea, LTFU (EOT + 27 months): Worsened | 8 | 12
  Diarrhoea, LTFU (EOT + 27 months): Stable | 25 | 43
  Diarrhoea, LTFU (EOT + 27 months): Improved | 3 | 15
  FD, LTFU (EOT + 27 months): number analyzed (Participants) | 36 | 70
  FD, LTFU (EOT + 27 months): Worsened | 4 | 11
  FD, LTFU (EOT + 27 months): Stable | 25 | 49
  FD, LTFU (EOT + 27 months): Improved | 7 | 10
  GHS/QoL, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 38
  GHS/QoL, LTFU (EOT + 33 months): Worsened | 4 | 8
  GHS/QoL, LTFU (EOT + 33 months): Stable | 6 | 20
  GHS/QoL, LTFU (EOT + 33 months): Improved | 6 | 10
  PF, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  PF, LTFU (EOT + 33 months): Worsened | 5 | 10
  PF, LTFU (EOT + 33 months): Stable | 9 | 14
  PF, LTFU (EOT + 33 months): Improved | 2 | 15
  RF, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  RF, LTFU (EOT + 33 months): Worsened | 4 | 12
  RF, LTFU (EOT + 33 months): Stable | 8 | 13
  RF, LTFU (EOT + 33 months): Improved | 4 | 14
  EF, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 38
  EF, LTFU (EOT + 33 months): Worsened | 5 | 4
  EF, LTFU (EOT + 33 months): Stable | 8 | 24
  EF, LTFU (EOT + 33 months): Improved | 3 | 10
  CF, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 38
  CF, LTFU (EOT + 33 months): Worsened | 5 | 15
  CF, LTFU (EOT + 33 months): Stable | 9 | 15
  CF, LTFU (EOT + 33 months): Improved | 2 | 8
  SF, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 38
  SF, LTFU (EOT + 33 months): Worsened | 5 | 14
  SF, LTFU (EOT + 33 months): Stable | 6 | 15
  SF, LTFU (EOT + 33 months): Improved | 5 | 9
  Fatigue, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  Fatigue, LTFU (EOT + 33 months): Worsened | 5 | 11
  Fatigue, LTFU (EOT + 33 months): Stable | 2 | 12
  Fatigue, LTFU (EOT + 33 months): Improved | 9 | 16
  N/V, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  N/V, LTFU (EOT + 33 months): Worsened | 4 | 7
  N/V, LTFU (EOT + 33 months): Stable | 11 | 24
  N/V, LTFU (EOT + 33 months): Improved | 1 | 8
  Pain, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  Pain, LTFU (EOT + 33 months): Worsened | 2 | 16
  Pain, LTFU (EOT + 33 months): Stable | 7 | 10
  Pain, LTFU (EOT + 33 months): Improved | 7 | 13
  Dyspnoea, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  Dyspnoea, LTFU (EOT + 33 months): Worsened | 5 | 10
  Dyspnoea, LTFU (EOT + 33 months): Stable | 9 | 21
  Dyspnoea, LTFU (EOT + 33 months): Improved | 2 | 8
  Insomnia, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 38
  Insomnia, LTFU (EOT + 33 months): Worsened | 3 | 6
  Insomnia, LTFU (EOT + 33 months): Stable | 9 | 15
  Insomnia, LTFU (EOT + 33 months): Improved | 4 | 17
  AL, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  AL, LTFU (EOT + 33 months): Worsened | 6 | 3
  AL, LTFU (EOT + 33 months): Stable | 7 | 28
  AL, LTFU (EOT + 33 months): Improved | 3 | 8
  Constipation, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  Constipation, LTFU (EOT + 33 months): Worsened | 2 | 10
  Constipation, LTFU (EOT + 33 months): Stable | 7 | 19
  Constipation, LTFU (EOT + 33 months): Improved | 7 | 10
  Diarrhoea, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 38
  Diarrhoea, LTFU (EOT + 33 months): Worsened | 5 | 3
  Diarrhoea, LTFU (EOT + 33 months): Stable | 10 | 26
  Diarrhoea, LTFU (EOT + 33 months): Improved | 1 | 9
  FD, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 38
  FD, LTFU (EOT + 33 months): Worsened | 2 | 6
  FD, LTFU (EOT + 33 months): Stable | 10 | 26
  FD, LTFU (EOT + 33 months): Improved | 4 | 6
  GHS/QoL, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  GHS/QoL, LTFU (EOT + 39 months): Worsened | 3 | 7
  GHS/QoL, LTFU (EOT + 39 months): Stable | 3 | 14
  GHS/QoL, LTFU (EOT + 39 months): Improved | 5 | 6
  PF, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  PF, LTFU (EOT + 39 months): Worsened | 2 | 7
  PF, LTFU (EOT + 39 months): Stable | 6 | 12
  PF, LTFU (EOT + 39 months): Improved | 3 | 8
  RF, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  RF, LTFU (EOT + 39 months): Worsened | 0 | 6
  RF, LTFU (EOT + 39 months): Stable | 7 | 12
  RF, LTFU (EOT + 39 months): Improved | 4 | 9
  EF, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  EF, LTFU (EOT + 39 months): Worsened | 2 | 8
  EF, LTFU (EOT + 39 months): Stable | 7 | 16
  EF, LTFU (EOT + 39 months): Improved | 2 | 3
  CF, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  CF, LTFU (EOT + 39 months): Worsened | 4 | 12
  CF, LTFU (EOT + 39 months): Stable | 5 | 7
  CF, LTFU (EOT + 39 months): Improved | 2 | 8
  SF, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  SF, LTFU (EOT + 39 months): Worsened | 1 | 9
  SF, LTFU (EOT + 39 months): Stable | 4 | 12
  SF, LTFU (EOT + 39 months): Improved | 6 | 6
  Fatigue, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  Fatigue, LTFU (EOT + 39 months): Worsened | 1 | 10
  Fatigue, LTFU (EOT + 39 months): Stable | 3 | 6
  Fatigue, LTFU (EOT + 39 months): Improved | 7 | 11
  N/V, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  N/V, LTFU (EOT + 39 months): Worsened | 3 | 5
  N/V, LTFU (EOT + 39 months): Stable | 8 | 19
  N/V, LTFU (EOT + 39 months): Improved | 0 | 3
  Pain, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  Pain, LTFU (EOT + 39 months): Worsened | 4 | 10
  Pain, LTFU (EOT + 39 months): Stable | 4 | 8
  Pain, LTFU (EOT + 39 months): Improved | 3 | 9
  Dyspnoea, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  Dyspnoea, LTFU (EOT + 39 months): Worsened | 5 | 9
  Dyspnoea, LTFU (EOT + 39 months): Stable | 3 | 15
  Dyspnoea, LTFU (EOT + 39 months): Improved | 3 | 3
  Insomnia, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  Insomnia, LTFU (EOT + 39 months): Worsened | 5 | 5
  Insomnia, LTFU (EOT + 39 months): Stable | 3 | 9
  Insomnia, LTFU (EOT + 39 months): Improved | 3 | 13
  AL, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  AL, LTFU (EOT + 39 months): Worsened | 1 | 2
  AL, LTFU (EOT + 39 months): Stable | 7 | 20
  AL, LTFU (EOT + 39 months): Improved | 3 | 5
  Constipation, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  Constipation, LTFU (EOT + 39 months): Worsened | 2 | 10
  Constipation, LTFU (EOT + 39 months): Stable | 5 | 10
  Constipation, LTFU (EOT + 39 months): Improved | 4 | 7
  Diarrhoea, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  Diarrhoea, LTFU (EOT + 39 months): Worsened | 2 | 6
  Diarrhoea, LTFU (EOT + 39 months): Stable | 8 | 16
  Diarrhoea, LTFU (EOT + 39 months): Improved | 1 | 5
  FD, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  FD, LTFU (EOT + 39 months): Worsened | 3 | 5
  FD, LTFU (EOT + 39 months): Stable | 6 | 18
  FD, LTFU (EOT + 39 months): Improved | 2 | 4
  GHS/QoL, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  GHS/QoL, LTFU (EOT + 45 months): Worsened | 1 | 4
  GHS/QoL, LTFU (EOT + 45 months): Stable | 1 | 8
  GHS/QoL, LTFU (EOT + 45 months): Improved | 2 | 3
  PF, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  PF, LTFU (EOT + 45 months): Worsened | 1 | 3
  PF, LTFU (EOT + 45 months): Stable | 2 | 8
  PF, LTFU (EOT + 45 months): Improved | 1 | 4
  RF, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  RF, LTFU (EOT + 45 months): Worsened | 0 | 2
  RF, LTFU (EOT + 45 months): Stable | 4 | 8
  RF, LTFU (EOT + 45 months): Improved | 0 | 5
  EF, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  EF, LTFU (EOT + 45 months): Worsened | 0 | 4
  EF, LTFU (EOT + 45 months): Stable | 3 | 8
  EF, LTFU (EOT + 45 months): Improved | 1 | 3
  CF, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  CF, LTFU (EOT + 45 months): Worsened | 0 | 4
  CF, LTFU (EOT + 45 months): Stable | 4 | 7
  CF, LTFU (EOT + 45 months): Improved | 0 | 4
  SF, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  SF, LTFU (EOT + 45 months): Worsened | 0 | 3
  SF, LTFU (EOT + 45 months): Stable | 2 | 8
  SF, LTFU (EOT + 45 months): Improved | 2 | 4
  Fatigue, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  Fatigue, LTFU (EOT + 45 months): Worsened | 1 | 5
  Fatigue, LTFU (EOT + 45 months): Stable | 1 | 4
  Fatigue, LTFU (EOT + 45 months): Improved | 2 | 6
  N/V, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  N/V, LTFU (EOT + 45 months): Worsened | 0 | 2
  N/V, LTFU (EOT + 45 months): Stable | 4 | 11
  N/V, LTFU (EOT + 45 months): Improved | 0 | 2
  Pain, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  Pain, LTFU (EOT + 45 months): Worsened | 1 | 5
  Pain, LTFU (EOT + 45 months): Stable | 1 | 6
  Pain, LTFU (EOT + 45 months): Improved | 2 | 4
  Dyspnoea, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  Dyspnoea, LTFU (EOT + 45 months): Worsened | 1 | 3
  Dyspnoea, LTFU (EOT + 45 months): Stable | 2 | 9
  Dyspnoea, LTFU (EOT + 45 months): Improved | 1 | 3
  Insomnia, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  Insomnia, LTFU (EOT + 45 months): Worsened | 2 | 5
  Insomnia, LTFU (EOT + 45 months): Stable | 1 | 2
  Insomnia, LTFU (EOT + 45 months): Improved | 1 | 8
  AL, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  AL, LTFU (EOT + 45 months): Worsened | 0 | 1
  AL, LTFU (EOT + 45 months): Stable | 2 | 12
  AL, LTFU (EOT + 45 months): Improved | 2 | 2
  Constipation, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  Constipation, LTFU (EOT + 45 months): Worsened | 1 | 5
  Constipation, LTFU (EOT + 45 months): Stable | 1 | 7
  Constipation, LTFU (EOT + 45 months): Improved | 2 | 3
  Diarrhoea, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  Diarrhoea, LTFU (EOT + 45 months): Worsened | 0 | 5
  Diarrhoea, LTFU (EOT + 45 months): Stable | 3 | 7
  Diarrhoea, LTFU (EOT + 45 months): Improved | 1 | 3
  FD, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  FD, LTFU (EOT + 45 months): Worsened | 1 | 2
  FD, LTFU (EOT + 45 months): Stable | 1 | 11
  FD, LTFU (EOT + 45 months): Improved | 2 | 2
  GHS/QoL, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  GHS/QoL, LTFU (EOT + 51 months): Worsened | 0 | 0
  GHS/QoL, LTFU (EOT + 51 months): Stable | 2 | 4
  GHS/QoL, LTFU (EOT + 51 months): Improved | 0 | 1
  PF, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  PF, LTFU (EOT + 51 months): Worsened | 1 | 1
  PF, LTFU (EOT + 51 months): Stable | 1 | 3
  PF, LTFU (EOT + 51 months): Improved | 0 | 1
  RF, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  RF, LTFU (EOT + 51 months): Worsened | 0 | 0
  RF, LTFU (EOT + 51 months): Stable | 1 | 2
  RF, LTFU (EOT + 51 months): Improved | 1 | 3
  EF, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  EF, LTFU (EOT + 51 months): Worsened | 0 | 1
  EF, LTFU (EOT + 51 months): Stable | 1 | 2
  EF, LTFU (EOT + 51 months): Improved | 1 | 2
  CF, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  CF, LTFU (EOT + 51 months): Worsened | 0 | 1
  CF, LTFU (EOT + 51 months): Stable | 2 | 2
  CF, LTFU (EOT + 51 months): Improved | 0 | 2
  SF, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  SF, LTFU (EOT + 51 months): Worsened | 0 | 1
  SF, LTFU (EOT + 51 months): Stable | 1 | 3
  SF, LTFU (EOT + 51 months): Improved | 1 | 1
  Fatigue, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  Fatigue, LTFU (EOT + 51 months): Worsened | 0 | 1
  Fatigue, LTFU (EOT + 51 months): Stable | 1 | 0
  Fatigue, LTFU (EOT + 51 months): Improved | 1 | 4
  N/V, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  N/V, LTFU (EOT + 51 months): Worsened | 0 | 0
  N/V, LTFU (EOT + 51 months): Stable | 2 | 5
  N/V, LTFU (EOT + 51 months): Improved | 0 | 0
  Pain, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  Pain, LTFU (EOT + 51 months): Worsened | 0 | 0
  Pain, LTFU (EOT + 51 months): Stable | 1 | 2
  Pain, LTFU (EOT + 51 months): Improved | 1 | 3
  Dyspnoea, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  Dyspnoea, LTFU (EOT + 51 months): Worsened | 1 | 0
  Dyspnoea, LTFU (EOT + 51 months): Stable | 1 | 4
  Dyspnoea, LTFU (EOT + 51 months): Improved | 0 | 1
  Insomnia, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  Insomnia, LTFU (EOT + 51 months): Worsened | 0 | 1
  Insomnia, LTFU (EOT + 51 months): Stable | 1 | 3
  Insomnia, LTFU (EOT + 51 months): Improved | 1 | 1
  AL, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  AL, LTFU (EOT + 51 months): Worsened | 0 | 0
  AL, LTFU (EOT + 51 months): Stable | 1 | 4
  AL, LTFU (EOT + 51 months): Improved | 1 | 1
  Constipation, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  Constipation, LTFU (EOT + 51 months): Worsened | 0 | 2
  Constipation, LTFU (EOT + 51 months): Stable | 1 | 2
  Constipation, LTFU (EOT + 51 months): Improved | 1 | 1
  Diarrhoea, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  Diarrhoea, LTFU (EOT + 51 months): Worsened | 0 | 1
  Diarrhoea, LTFU (EOT + 51 months): Stable | 1 | 3
  Diarrhoea, LTFU (EOT + 51 months): Improved | 1 | 1
  FD, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  FD, LTFU (EOT + 51 months): Worsened | 0 | 0
  FD, LTFU (EOT + 51 months): Stable | 0 | 3
  FD, LTFU (EOT + 51 months): Improved | 2 | 2
  GHS/QoL, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  GHS/QoL, LTFU (EOT + 57 months): Worsened | 0 | 0
  GHS/QoL, LTFU (EOT + 57 months): Stable | 2 | 1
  GHS/QoL, LTFU (EOT + 57 months): Improved | 0 | 0
  PF, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  PF, LTFU (EOT + 57 months): Worsened | 1 | 0
  PF, LTFU (EOT + 57 months): Stable | 1 | 1
  PF, LTFU (EOT + 57 months): Improved | 0 | 0
  RF, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  RF, LTFU (EOT + 57 months): Worsened | 0 | 0
  RF, LTFU (EOT + 57 months): Stable | 2 | 0
  RF, LTFU (EOT + 57 months): Improved | 0 | 1
  EF, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  EF, LTFU (EOT + 57 months): Worsened | 0 | 0
  EF, LTFU (EOT + 57 months): Stable | 2 | 0
  EF, LTFU (EOT + 57 months): Improved | 0 | 1
  CF, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  CF, LTFU (EOT + 57 months): Worsened | 0 | 0
  CF, LTFU (EOT + 57 months): Stable | 2 | 1
  CF, LTFU (EOT + 57 months): Improved | 0 | 0
  SF, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  SF, LTFU (EOT + 57 months): Worsened | 0 | 0
  SF, LTFU (EOT + 57 months): Stable | 1 | 1
  SF, LTFU (EOT + 57 months): Improved | 1 | 0
  Fatigue, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  Fatigue, LTFU (EOT + 57 months): Worsened | 0 | 0
  Fatigue, LTFU (EOT + 57 months): Stable | 1 | 1
  Fatigue, LTFU (EOT + 57 months): Improved | 1 | 0
  N/V, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  N/V, LTFU (EOT + 57 months): Worsened | 0 | 0
  N/V, LTFU (EOT + 57 months): Stable | 2 | 1
  N/V, LTFU (EOT + 57 months): Improved | 0 | 0
  Pain, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  Pain, LTFU (EOT + 57 months): Worsened | 0 | 0
  Pain, LTFU (EOT + 57 months): Stable | 1 | 0
  Pain, LTFU (EOT + 57 months): Improved | 1 | 1
  Dyspnoea, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  Dyspnoea, LTFU (EOT + 57 months): Worsened | 1 | 0
  Dyspnoea, LTFU (EOT + 57 months): Stable | 1 | 1
  Dyspnoea, LTFU (EOT + 57 months): Improved | 0 | 0
  Insomnia, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  Insomnia, LTFU (EOT + 57 months): Worsened | 0 | 0
  Insomnia, LTFU (EOT + 57 months): Stable | 1 | 1
  Insomnia, LTFU (EOT + 57 months): Improved | 1 | 0
  AL, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  AL, LTFU (EOT + 57 months): Worsened | 0 | 0
  AL, LTFU (EOT + 57 months): Stable | 1 | 1
  AL, LTFU (EOT + 57 months): Improved | 1 | 0
  Constipation, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  Constipation, LTFU (EOT + 57 months): Worsened | 0 | 0
  Constipation, LTFU (EOT + 57 months): Stable | 1 | 0
  Constipation, LTFU (EOT + 57 months): Improved | 1 | 1
  Diarrhoea, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  Diarrhoea, LTFU (EOT + 57 months): Worsened | 0 | 0
  Diarrhoea, LTFU (EOT + 57 months): Stable | 1 | 0
  Diarrhoea, LTFU (EOT + 57 months): Improved | 1 | 1
  FD, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  FD, LTFU (EOT + 57 months): Worsened | 0 | 0
  FD, LTFU (EOT + 57 months): Stable | 0 | 1
  FD, LTFU (EOT + 57 months): Improved | 2 | 0
  GHS/QoL, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  GHS/QoL, LTFU (EOT + 63 months): Worsened | 0 | 0
  GHS/QoL, LTFU (EOT + 63 months): Stable | 1 | 0
  GHS/QoL, LTFU (EOT + 63 months): Improved | 0 | 0
  PF, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  PF, LTFU (EOT + 63 months): Worsened | 0 | 0
  PF, LTFU (EOT + 63 months): Stable | 1 | 0
  PF, LTFU (EOT + 63 months): Improved | 0 | 0
  RF, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  RF, LTFU (EOT + 63 months): Worsened | 0 | 0
  RF, LTFU (EOT + 63 months): Stable | 1 | 0
  RF, LTFU (EOT + 63 months): Improved | 0 | 0
  EF, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  EF, LTFU (EOT + 63 months): Worsened | 0 | 0
  EF, LTFU (EOT + 63 months): Stable | 1 | 0
  EF, LTFU (EOT + 63 months): Improved | 0 | 0
  CF, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  CF, LTFU (EOT + 63 months): Worsened | 0 | 0
  CF, LTFU (EOT + 63 months): Stable | 1 | 0
  CF, LTFU (EOT + 63 months): Improved | 0 | 0
  SF, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  SF, LTFU (EOT + 63 months): Worsened | 0 | 0
  SF, LTFU (EOT + 63 months): Stable | 1 | 0
  SF, LTFU (EOT + 63 months): Improved | 0 | 0
  Fatigue, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  Fatigue, LTFU (EOT + 63 months): Worsened | 0 | 0
  Fatigue, LTFU (EOT + 63 months): Stable | 1 | 0
  Fatigue, LTFU (EOT + 63 months): Improved | 0 | 0
  N/V, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  N/V, LTFU (EOT + 63 months): Worsened | 0 | 0
  N/V, LTFU (EOT + 63 months): Stable | 1 | 0
  N/V, LTFU (EOT + 63 months): Improved | 0 | 0
  Pain, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  Pain, LTFU (EOT + 63 months): Worsened | 0 | 0
  Pain, LTFU (EOT + 63 months): Stable | 1 | 0
  Pain, LTFU (EOT + 63 months): Improved | 0 | 0
  Dyspnoea, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  Dyspnoea, LTFU (EOT + 63 months): Worsened | 0 | 0
  Dyspnoea, LTFU (EOT + 63 months): Stable | 1 | 0
  Dyspnoea, LTFU (EOT + 63 months): Improved | 0 | 0
  Insomnia, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  Insomnia, LTFU (EOT + 63 months): Worsened | 0 | 0
  Insomnia, LTFU (EOT + 63 months): Stable | 1 | 0
  Insomnia, LTFU (EOT + 63 months): Improved | 0 | 0
  AL, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  AL, LTFU (EOT + 63 months): Worsened | 0 | 0
  AL, LTFU (EOT + 63 months): Stable | 1 | 0
  AL, LTFU (EOT + 63 months): Improved | 0 | 0
  Constipation, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  Constipation, LTFU (EOT + 63 months): Worsened | 0 | 0
  Constipation, LTFU (EOT + 63 months): Stable | 0 | 0
  Constipation, LTFU (EOT + 63 months): Improved | 1 | 0
  Diarrhoea, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  Diarrhoea, LTFU (EOT + 63 months): Worsened | 0 | 0
  Diarrhoea, LTFU (EOT + 63 months): Stable | 1 | 0
  Diarrhoea, LTFU (EOT + 63 months): Improved | 0 | 0
  FD, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  FD, LTFU (EOT + 63 months): Worsened | 0 | 0
  FD, LTFU (EOT + 63 months): Stable | 0 | 0
  FD, LTFU (EOT + 63 months): Improved | 1 | 0

13. Secondary Outcome: Number of Participants With Change in Status in EORTC-QLQ Ovarian Cancer Module (EORTC-QLQ-OV28) Questionnaire
Description: The EORTC QLQ-OV28 supplements the QLQ-C30. It includes three functional scales (body image (BI), sexuality (S), attitude to disease/treatment(ATD)) and five symptom scales/items (abdominal/GI symptoms (AS), peripheral neuropathy (PN), hormonal/menopausal symptoms (MS), other chemotherapy side effects (CSE), and hair loss (HS)). Participants responded on a scale of 1-4 (1=not at all, 2=a little, 3=quite a bit, 4=very much). Higher scores represent better functioning (better quality of life). For functional scales: improved (worsened) is defined as >=10 points increase (decrease) from baseline. For symptom scales: improved (worsened) is defined as >=10 points decrease (increase) from baseline. Baseline is defined as the latest, non-missing collected value, excluding end of treatment, safety follow-up, long term follow-up visits records and unscheduled visits after end of treatment.
Time Frame: as for outcome 11
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
Number analyzed (Participants) | 331 | 657
Participants
  BI, Cycle 4 Chemotherapy: number analyzed (Participants) | 270 | 534
  BI, Cycle 4 Chemotherapy: Worsened | 89 | 214
  BI, Cycle 4 Chemotherapy: Stable | 108 | 189
  BI, Cycle 4 Chemotherapy: Improved | 73 | 131
  S, Cycle 4 Chemotherapy: number analyzed (Participants) | 269 | 526
  S, Cycle 4 Chemotherapy: Worsened | 30 | 59
  S, Cycle 4 Chemotherapy: Stable | 188 | 390
  S, Cycle 4 Chemotherapy: Improved | 51 | 77
  ATD, Cycle 4 Chemotherapy: number analyzed (Participants) | 270 | 534
  ATD, Cycle 4 Chemotherapy: Worsened | 103 | 205
  ATD, Cycle 4 Chemotherapy: Stable | 91 | 148
  ATD, Cycle 4 Chemotherapy: Improved | 76 | 181
  AS, Cycle 4 Chemotherapy: number analyzed (Participants) | 276 | 535
  AS, Cycle 4 Chemotherapy: Worsened | 40 | 81
  AS, Cycle 4 Chemotherapy: Stable | 166 | 325
  AS, Cycle 4 Chemotherapy: Improved | 70 | 129
  PN, Cycle 4 Chemotherapy: number analyzed (Participants) | 276 | 535
  PN, Cycle 4 Chemotherapy: Worsened | 151 | 316
  PN, Cycle 4 Chemotherapy: Stable | 68 | 135
  PN, Cycle 4 Chemotherapy: Improved | 57 | 84
  MS, Cycle 4 Chemotherapy: number analyzed (Participants) | 276 | 535
  MS, Cycle 4 Chemotherapy: Worsened | 68 | 153
  MS, Cycle 4 Chemotherapy: Stable | 135 | 255
  MS, Cycle 4 Chemotherapy: Improved | 73 | 127
  CSE, Cycle 4 Chemotherapy: number analyzed (Participants) | 276 | 535
  CSE, Cycle 4 Chemotherapy: Worsened | 88 | 168
  CSE, Cycle 4 Chemotherapy: Stable | 145 | 278
  CSE, Cycle 4 Chemotherapy: Improved | 43 | 89
  HS, Cycle 4 Chemotherapy: number analyzed (Participants) | 273 | 534
  HS, Cycle 4 Chemotherapy: Worsened | 92 | 176
  HS, Cycle 4 Chemotherapy: Stable | 81 | 139
  HS, Cycle 4 Chemotherapy: Improved | 100 | 219
  BI, Cycle 6 Chemotherapy: number analyzed (Participants) | 266 | 532
  BI, Cycle 6 Chemotherapy: Worsened | 99 | 216
  BI, Cycle 6 Chemotherapy: Stable | 97 | 168
  BI, Cycle 6 Chemotherapy: Improved | 70 | 148
  S, Cycle 6 Chemotherapy: number analyzed (Participants) | 261 | 525
  S, Cycle 6 Chemotherapy: Worsened | 29 | 71
  S, Cycle 6 Chemotherapy: Stable | 184 | 368
  S, Cycle 6 Chemotherapy: Improved | 48 | 86
  ATD, Cycle 6 Chemotherapy: number analyzed (Participants) | 265 | 532
  ATD, Cycle 6 Chemotherapy: Worsened | 87 | 218
  ATD, Cycle 6 Chemotherapy: Stable | 81 | 132
  ATD, Cycle 6 Chemotherapy: Improved | 97 | 182
  AS, Cycle 6 Chemotherapy: number analyzed (Participants) | 267 | 534
  AS, Cycle 6 Chemotherapy: Worsened | 32 | 66
  AS, Cycle 6 Chemotherapy: Stable | 148 | 312
  AS, Cycle 6 Chemotherapy: Improved | 87 | 156
  PN, Cycle 6 Chemotherapy: number analyzed (Participants) | 267 | 533
  PN, Cycle 6 Chemotherapy: Worsened | 175 | 371
  PN, Cycle 6 Chemotherapy: Stable | 50 | 99
  PN, Cycle 6 Chemotherapy: Improved | 42 | 63
  MS, Cycle 6 Chemotherapy: number analyzed (Participants) | 267 | 533
  MS, Cycle 6 Chemotherapy: Worsened | 71 | 161
  MS, Cycle 6 Chemotherapy: Stable | 113 | 240
  MS, Cycle 6 Chemotherapy: Improved | 83 | 132
  CSE, Cycle 6 Chemotherapy: number analyzed (Participants) | 267 | 532
  CSE, Cycle 6 Chemotherapy: Worsened | 77 | 173
  CSE, Cycle 6 Chemotherapy: Stable | 144 | 279
  CSE, Cycle 6 Chemotherapy: Improved | 46 | 80
  HS, Cycle 6 Chemotherapy: number analyzed (Participants) | 266 | 532
  HS, Cycle 6 Chemotherapy: Worsened | 106 | 181
  HS, Cycle 6 Chemotherapy: Stable | 60 | 121
  HS, Cycle 6 Chemotherapy: Improved | 100 | 230
  BI, Cycle 1 Maintenance: number analyzed (Participants) | 262 | 494
  BI, Cycle 1 Maintenance: Worsened | 95 | 187
  BI, Cycle 1 Maintenance: Stable | 92 | 165
  BI, Cycle 1 Maintenance: Improved | 75 | 142
  S, Cycle 1 Maintenance: number analyzed (Participants) | 254 | 485
  S, Cycle 1 Maintenance: Worsened | 29 | 63
  S, Cycle 1 Maintenance: Stable | 172 | 337
  S, Cycle 1 Maintenance: Improved | 53 | 85
  ATD, Cycle 1 Maintenance: number analyzed (Participants) | 262 | 494
  ATD, Cycle 1 Maintenance: Worsened | 104 | 181
  ATD, Cycle 1 Maintenance: Stable | 73 | 143
  ATD, Cycle 1 Maintenance: Improved | 85 | 170
  AS, Cycle 1 Maintenance: number analyzed (Participants) | 262 | 496
  AS, Cycle 1 Maintenance: Worsened | 25 | 55
  AS, Cycle 1 Maintenance: Stable | 152 | 284
  AS, Cycle 1 Maintenance: Improved | 85 | 157
  PN, Cycle 1 Maintenance: number analyzed (Participants) | 262 | 495
  PN, Cycle 1 Maintenance: Worsened | 173 | 358
  PN, Cycle 1 Maintenance: Stable | 49 | 73
  PN, Cycle 1 Maintenance: Improved | 40 | 64
  MS, Cycle 1 Maintenance: number analyzed (Participants) | 262 | 496
  MS, Cycle 1 Maintenance: Worsened | 68 | 127
  MS, Cycle 1 Maintenance: Stable | 115 | 239
  MS, Cycle 1 Maintenance: Improved | 79 | 130
  CSE, Cycle 1 Maintenance: number analyzed (Participants) | 262 | 495
  CSE, Cycle 1 Maintenance: Worsened | 66 | 162
  CSE, Cycle 1 Maintenance: Stable | 151 | 235
  CSE, Cycle 1 Maintenance: Improved | 45 | 98
  HS, Cycle 1 Maintenance: number analyzed (Participants) | 260 | 494
  HS, Cycle 1 Maintenance: Worsened | 89 | 145
  HS, Cycle 1 Maintenance: Stable | 56 | 117
  HS, Cycle 1 Maintenance: Improved | 115 | 232
  BI, Cycle 2 Maintenance: number analyzed (Participants) | 227 | 429
  BI, Cycle 2 Maintenance: Worsened | 74 | 162
  BI, Cycle 2 Maintenance: Stable | 85 | 143
  BI, Cycle 2 Maintenance: Improved | 68 | 124
  S, Cycle 2 Maintenance: number analyzed (Participants) | 220 | 417
  S, Cycle 2 Maintenance: Worsened | 16 | 53
  S, Cycle 2 Maintenance: Stable | 166 | 290
  S, Cycle 2 Maintenance: Improved | 38 | 74
  ATD, Cycle 2 Maintenance: number analyzed (Participants) | 227 | 428
  ATD, Cycle 2 Maintenance: Worsened | 75 | 156
  ATD, Cycle 2 Maintenance: Stable | 54 | 103
  ATD, Cycle 2 Maintenance: Improved | 98 | 169
  AS, Cycle 2 Maintenance: number analyzed (Participants) | 228 | 431
  AS, Cycle 2 Maintenance: Worsened | 19 | 35
  AS, Cycle 2 Maintenance: Stable | 127 | 260
  AS, Cycle 2 Maintenance: Improved | 82 | 136
  PN, Cycle 2 Maintenance: number analyzed (Participants) | 228 | 430
  PN, Cycle 2 Maintenance: Worsened | 128 | 277
  PN, Cycle 2 Maintenance: Stable | 57 | 79
  PN, Cycle 2 Maintenance: Improved | 43 | 74
  MS, Cycle 2 Maintenance: number analyzed (Participants) | 228 | 430
  MS, Cycle 2 Maintenance: Worsened | 52 | 129
  MS, Cycle 2 Maintenance: Stable | 106 | 186
  MS, Cycle 2 Maintenance: Improved | 70 | 115
  CSE, Cycle 2 Maintenance: number analyzed (Participants) | 228 | 430
  CSE, Cycle 2 Maintenance: Worsened | 54 | 115
  CSE, Cycle 2 Maintenance: Stable | 125 | 229
  CSE, Cycle 2 Maintenance: Improved | 49 | 86
  HS, Cycle 2 Maintenance: number analyzed (Participants) | 224 | 428
  HS, Cycle 2 Maintenance: Worsened | 48 | 85
  HS, Cycle 2 Maintenance: Stable | 57 | 100
  HS, Cycle 2 Maintenance: Improved | 119 | 243
  BI, Cycle 3 Maintenance: number analyzed (Participants) | 232 | 441
  BI, Cycle 3 Maintenance: Worsened | 70 | 159
  BI, Cycle 3 Maintenance: Stable | 88 | 147
  BI, Cycle 3 Maintenance: Improved | 74 | 135
  S, Cycle 3 Maintenance: number analyzed (Participants) | 226 | 424
  S, Cycle 3 Maintenance: Worsened | 24 | 55
  S, Cycle 3 Maintenance: Stable | 161 | 291
  S, Cycle 3 Maintenance: Improved | 41 | 78
  ATD, Cycle 3 Maintenance: number analyzed (Participants) | 232 | 441
  ATD, Cycle 3 Maintenance: Worsened | 71 | 161
  ATD, Cycle 3 Maintenance: Stable | 55 | 109
  ATD, Cycle 3 Maintenance: Improved | 106 | 171
  AS, Cycle 3 Maintenance: number analyzed (Participants) | 233 | 442
  AS, Cycle 3 Maintenance: Worsened | 38 | 56
  AS, Cycle 3 Maintenance: Stable | 123 | 246
  AS, Cycle 3 Maintenance: Improved | 72 | 140
  PN, Cycle 3 Maintenance: number analyzed (Participants) | 232 | 442
  PN, Cycle 3 Maintenance: Worsened | 129 | 285
  PN, Cycle 3 Maintenance: Stable | 53 | 91
  PN, Cycle 3 Maintenance: Improved | 50 | 66
  MS, Cycle 3 Maintenance: number analyzed (Participants) | 232 | 442
  MS, Cycle 3 Maintenance: Worsened | 69 | 144
  MS, Cycle 3 Maintenance: Stable | 92 | 193
  MS, Cycle 3 Maintenance: Improved | 71 | 105
  CSE, Cycle 3 Maintenance: number analyzed (Participants) | 232 | 442
  CSE, Cycle 3 Maintenance: Worsened | 54 | 110
  CSE, Cycle 3 Maintenance: Stable | 118 | 242
  CSE, Cycle 3 Maintenance: Improved | 60 | 90
  HS, Cycle 3 Maintenance: number analyzed (Participants) | 232 | 440
  HS, Cycle 3 Maintenance: Worsened | 32 | 54
  HS, Cycle 3 Maintenance: Stable | 66 | 96
  HS, Cycle 3 Maintenance: Improved | 134 | 290
  BI, Cycle 6 Maintenance: number analyzed (Participants) | 195 | 397
  BI, Cycle 6 Maintenance: Worsened | 54 | 126
  BI, Cycle 6 Maintenance: Stable | 72 | 132
  BI, Cycle 6 Maintenance: Improved | 69 | 139
  S, Cycle 6 Maintenance: number analyzed (Participants) | 190 | 382
  S, Cycle 6 Maintenance: Worsened | 16 | 45
  S, Cycle 6 Maintenance: Stable | 121 | 242
  S, Cycle 6 Maintenance: Improved | 53 | 95
  ATD, Cycle 6 Maintenance9: number analyzed (Participants) | 195 | 397
  ATD, Cycle 6 Maintenance9: Worsened | 54 | 117
  ATD, Cycle 6 Maintenance9: Stable | 44 | 101
  ATD, Cycle 6 Maintenance9: Improved | 97 | 179
  AS, Cycle 6 Maintenance: number analyzed (Participants) | 198 | 399
  AS, Cycle 6 Maintenance: Worsened | 22 | 49
  AS, Cycle 6 Maintenance: Stable | 106 | 222
  AS, Cycle 6 Maintenance: Improved | 70 | 128
  PN, Cycle 6 Maintenance: number analyzed (Participants) | 198 | 398
  PN, Cycle 6 Maintenance: Worsened | 108 | 234
  PN, Cycle 6 Maintenance: Stable | 43 | 89
  PN, Cycle 6 Maintenance: Improved | 47 | 75
  MS, Cycle 6 Maintenance: number analyzed (Participants) | 198 | 398
  MS, Cycle 6 Maintenance: Worsened | 53 | 127
  MS, Cycle 6 Maintenance: Stable | 85 | 164
  MS, Cycle 6 Maintenance: Improved | 60 | 107
  CSE, Cycle 6 Maintenance: number analyzed (Participants) | 198 | 398
  CSE, Cycle 6 Maintenance: Worsened | 37 | 102
  CSE, Cycle 6 Maintenance: Stable | 111 | 200
  CSE, Cycle 6 Maintenance: Improved | 50 | 96
  HS, Cycle 6 Maintenance: number analyzed (Participants) | 196 | 397
  HS, Cycle 6 Maintenance: Worsened | 13 | 23
  HS, Cycle 6 Maintenance: Stable | 58 | 92
  HS, Cycle 6 Maintenance: Improved | 125 | 282
  BI, Cycle 9 Maintenance: number analyzed (Participants) | 185 | 359
  BI, Cycle 9 Maintenance: Worsened | 51 | 99
  BI, Cycle 9 Maintenance: Stable | 59 | 130
  BI, Cycle 9 Maintenance: Improved | 75 | 130
  S, Cycle 9 Maintenance: number analyzed (Participants) | 179 | 344
  S, Cycle 9 Maintenance: Worsened | 19 | 40
  S, Cycle 9 Maintenance: Stable | 109 | 201
  S, Cycle 9 Maintenance: Improved | 51 | 103
  ATD, Cycle 9 Maintenance: number analyzed (Participants) | 185 | 359
  ATD, Cycle 9 Maintenance: Worsened | 47 | 89
  ATD, Cycle 9 Maintenance: Stable | 39 | 86
  ATD, Cycle 9 Maintenance: Improved | 99 | 184
  AS, Cycle 9 Maintenance: number analyzed (Participants) | 186 | 361
  AS, Cycle 9 Maintenance: Worsened | 22 | 38
  AS, Cycle 9 Maintenance: Stable | 103 | 198
  AS, Cycle 9 Maintenance: Improved | 61 | 125
  PN, Cycle 9 Maintenance: number analyzed (Participants) | 186 | 360
  PN, Cycle 9 Maintenance: Worsened | 91 | 206
  PN, Cycle 9 Maintenance: Stable | 52 | 75
  PN, Cycle 9 Maintenance: Improved | 43 | 79
  MS, Cycle 9 Maintenance: number analyzed (Participants) | 186 | 360
  MS, Cycle 9 Maintenance: Worsened | 51 | 96
  MS, Cycle 9 Maintenance: Stable | 67 | 158
  MS, Cycle 9 Maintenance: Improved | 68 | 106
  CSE, Cycle 9 Maintenance: number analyzed (Participants) | 186 | 360
  CSE, Cycle 9 Maintenance: Worsened | 39 | 81
  CSE, Cycle 9 Maintenance: Stable | 101 | 193
  CSE, Cycle 9 Maintenance: Improved | 46 | 86
  HS, Cycle 9 Maintenance: number analyzed (Participants) | 185 | 359
  HS, Cycle 9 Maintenance: Worsened | 7 | 17
  HS, Cycle 9 Maintenance: Stable | 52 | 74
  HS, Cycle 9 Maintenance: Improved | 126 | 268
  BI, Cycle 12 Maintenance: number analyzed (Participants) | 156 | 308
  BI, Cycle 12 Maintenance: Worsened | 32 | 79
  BI, Cycle 12 Maintenance: Stable | 57 | 99
  BI, Cycle 12 Maintenance: Improved | 67 | 130
  S, Cycle 12 Maintenance: number analyzed (Participants) | 151 | 293
  S, Cycle 12 Maintenance: Worsened | 14 | 30
  S, Cycle 12 Maintenance: Stable | 86 | 178
  S, Cycle 12 Maintenance: Improved | 51 | 85
  ATD, Cycle 12 Maintenance: number analyzed (Participants) | 156 | 308
  ATD, Cycle 12 Maintenance: Worsened | 35 | 83
  ATD, Cycle 12 Maintenance: Stable | 39 | 59
  ATD, Cycle 12 Maintenance: Improved | 82 | 166
  AS, Cycle 12 Maintenance: number analyzed (Participants) | 158 | 308
  AS, Cycle 12 Maintenance: Worsened | 16 | 49
  AS, Cycle 12 Maintenance: Stable | 90 | 166
  AS, Cycle 12 Maintenance: Improved | 52 | 93
  PN, Cycle 12 Maintenance: number analyzed (Participants) | 158 | 308
  PN, Cycle 12 Maintenance: Worsened | 68 | 164
  PN, Cycle 12 Maintenance: Stable | 46 | 73
  PN, Cycle 12 Maintenance: Improved | 44 | 71
  MS, Cycle 12 Maintenance: number analyzed (Participants) | 158 | 308
  MS, Cycle 12 Maintenance: Worsened | 44 | 91
  MS, Cycle 12 Maintenance: Stable | 59 | 138
  MS, Cycle 12 Maintenance: Improved | 55 | 79
  CSE, Cycle 12 Maintenance: number analyzed (Participants) | 158 | 308
  CSE, Cycle 12 Maintenance: Worsened | 25 | 66
  CSE, Cycle 12 Maintenance: Stable | 95 | 164
  CSE, Cycle 12 Maintenance: Improved | 38 | 78
  HS, Cycle 12 Maintenance: number analyzed (Participants) | 157 | 305
  HS, Cycle 12 Maintenance: Worsened | 5 | 6
  HS, Cycle 12 Maintenance: Stable | 44 | 68
  HS, Cycle 12 Maintenance: Improved | 108 | 231
  BI, Cycle 15 Maintenance: number analyzed (Participants) | 149 | 279
  BI, Cycle 15 Maintenance: Worsened | 40 | 73
  BI, Cycle 15 Maintenance: Stable | 54 | 92
  BI, Cycle 15 Maintenance: Improved | 55 | 114
  S, Cycle 15 Maintenance: number analyzed (Participants) | 144 | 263
  S, Cycle 15 Maintenance: Worsened | 18 | 33
  S, Cycle 15 Maintenance: Stable | 82 | 162
  S, Cycle 15 Maintenance: Improved | 44 | 68
  ATD, Cycle 15 Maintenance: number analyzed (Participants) | 149 | 279
  ATD, Cycle 15 Maintenance: Worsened | 26 | 59
  ATD, Cycle 15 Maintenance: Stable | 35 | 69
  ATD, Cycle 15 Maintenance: Improved | 88 | 151
  AS, Cycle 15 Maintenance: number analyzed (Participants) | 150 | 281
  AS, Cycle 15 Maintenance: Worsened | 22 | 30
  AS, Cycle 15 Maintenance: Stable | 86 | 154
  AS, Cycle 15 Maintenance: Improved | 42 | 97
  PN, Cycle 15 Maintenance: number analyzed (Participants) | 150 | 278
  PN, Cycle 15 Maintenance: Worsened | 66 | 147
  PN, Cycle 15 Maintenance: Stable | 42 | 59
  PN, Cycle 15 Maintenance: Improved | 42 | 72
  MS, Cycle 15 Maintenance: number analyzed (Participants) | 150 | 279
  MS, Cycle 15 Maintenance: Worsened | 41 | 80
  MS, Cycle 15 Maintenance: Stable | 62 | 116
  MS, Cycle 15 Maintenance: Improved | 47 | 83
  CSE, Cycle 15 Maintenance: number analyzed (Participants) | 150 | 278
  CSE, Cycle 15 Maintenance: Worsened | 30 | 60
  CSE, Cycle 15 Maintenance: Stable | 80 | 144
  CSE, Cycle 15 Maintenance: Improved | 40 | 74
  HS, Cycle 15 Maintenance: number analyzed (Participants) | 147 | 278
  HS, Cycle 15 Maintenance: Worsened | 7 | 6
  HS, Cycle 15 Maintenance: Stable | 40 | 59
  HS, Cycle 15 Maintenance: Improved | 100 | 213
  BI, Cycle 17 Maintenance: number analyzed (Participants) | 39 | 82
  BI, Cycle 17 Maintenance: Worsened | 10 | 15
  BI, Cycle 17 Maintenance: Stable | 13 | 32
  BI, Cycle 17 Maintenance: Improved | 16 | 35
  S, Cycle 17 Maintenance: number analyzed (Participants) | 38 | 79
  S, Cycle 17 Maintenance: Worsened | 4 | 10
  S, Cycle 17 Maintenance: Stable | 18 | 42
  S, Cycle 17 Maintenance: Improved | 16 | 27
  ATD, Cycle 17 Maintenance: number analyzed (Participants) | 39 | 81
  ATD, Cycle 17 Maintenance: Worsened | 8 | 16
  ATD, Cycle 17 Maintenance: Stable | 6 | 17
  ATD, Cycle 17 Maintenance: Improved | 25 | 48
  AS, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 83
  AS, Cycle 17 Maintenance: Worsened | 7 | 9
  AS, Cycle 17 Maintenance: Stable | 19 | 38
  AS, Cycle 17 Maintenance: Improved | 14 | 36
  PN, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 83
  PN, Cycle 17 Maintenance: Worsened | 19 | 45
  PN, Cycle 17 Maintenance: Stable | 7 | 19
  PN, Cycle 17 Maintenance: Improved | 14 | 19
  MS, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 83
  MS, Cycle 17 Maintenance: Worsened | 10 | 25
  MS, Cycle 17 Maintenance: Stable | 11 | 31
  MS, Cycle 17 Maintenance: Improved | 19 | 27
  CSE, Cycle 17 Maintenance: number analyzed (Participants) | 40 | 83
  CSE, Cycle 17 Maintenance: Worsened | 7 | 20
  CSE, Cycle 17 Maintenance: Stable | 20 | 38
  CSE, Cycle 17 Maintenance: Improved | 13 | 25
  HS, Cycle 17 Maintenance: number analyzed (Participants) | 39 | 82
  HS, Cycle 17 Maintenance: Worsened | 1 | 2
  HS, Cycle 17 Maintenance: Stable | 10 | 14
  HS, Cycle 17 Maintenance: Improved | 28 | 66
  BI, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 99
  BI, Cycle 23 Maintenance: Worsened | 9 | 25
  BI, Cycle 23 Maintenance: Stable | 20 | 37
  BI, Cycle 23 Maintenance: Improved | 26 | 37
  S, Cycle 23 Maintenance: number analyzed (Participants) | 54 | 92
  S, Cycle 23 Maintenance: Worsened | 4 | 9
  S, Cycle 23 Maintenance: Stable | 36 | 52
  S, Cycle 23 Maintenance: Improved | 14 | 31
  ATD, Cycle 23 Maintenance: number analyzed (Participants) | 55 | 98
  ATD, Cycle 23 Maintenance: Worsened | 8 | 21
  ATD, Cycle 23 Maintenance: Stable | 15 | 20
  ATD, Cycle 23 Maintenance: Improved | 32 | 57
  AS, Cycle 23 Maintenance: number analyzed (Participants) | 56 | 99
  AS, Cycle 23 Maintenance: Worsened | 8 | 12
  AS, Cycle 23 Maintenance: Stable | 34 | 52
  AS, Cycle 23 Maintenance: Improved | 14 | 35
  PN, Cycle 23 Maintenance: number analyzed (Participants) | 56 | 99
  PN, Cycle 23 Maintenance: Worsened | 20 | 50
  PN, Cycle 23 Maintenance: Stable | 18 | 17
  PN, Cycle 23 Maintenance: Improved | 18 | 32
  MS, Cycle 23 Maintenance: number analyzed (Participants) | 56 | 100
  MS, Cycle 23 Maintenance: Worsened | 18 | 28
  MS, Cycle 23 Maintenance: Stable | 25 | 46
  MS, Cycle 23 Maintenance: Improved | 13 | 26
  CSE, Cycle 23 Maintenance: number analyzed (Participants) | 56 | 99
  CSE, Cycle 23 Maintenance: Worsened | 9 | 21
  CSE, Cycle 23 Maintenance: Stable | 28 | 48
  CSE, Cycle 23 Maintenance: Improved | 19 | 30
  HS, Cycle 23 Maintenance: number analyzed (Participants) | 56 | 97
  HS, Cycle 23 Maintenance: Worsened | 4 | 6
  HS, Cycle 23 Maintenance: Stable | 17 | 17
  HS, Cycle 23 Maintenance: Improved | 35 | 74
  BI, Cycle 29 Maintenance: number analyzed (Participants) | 51 | 93
  BI, Cycle 29 Maintenance: Worsened | 13 | 26
  BI, Cycle 29 Maintenance: Stable | 18 | 29
  BI, Cycle 29 Maintenance: Improved | 20 | 38
  S, Cycle 29 Maintenance: number analyzed (Participants) | 49 | 85
  S, Cycle 29 Maintenance: Worsened | 5 | 11
  S, Cycle 29 Maintenance: Stable | 25 | 46
  S, Cycle 29 Maintenance: Improved | 19 | 28
  ATD, Cycle 29 Maintenance: number analyzed (Participants) | 51 | 94
  ATD, Cycle 29 Maintenance: Worsened | 8 | 18
  ATD, Cycle 29 Maintenance: Stable | 11 | 21
  ATD, Cycle 29 Maintenance: Improved | 32 | 55
  AS, Cycle 29 Maintenance: number analyzed (Participants) | 51 | 94
  AS, Cycle 29 Maintenance: Worsened | 9 | 14
  AS, Cycle 29 Maintenance: Stable | 30 | 52
  AS, Cycle 29 Maintenance: Improved | 12 | 28
  PN, Cycle 29 Maintenance: number analyzed (Participants) | 50 | 94
  PN, Cycle 29 Maintenance: Worsened | 17 | 48
  PN, Cycle 29 Maintenance: Stable | 16 | 20
  PN, Cycle 29 Maintenance: Improved | 17 | 26
  MS, Cycle 29 Maintenance: number analyzed (Participants) | 50 | 94
  MS, Cycle 29 Maintenance: Worsened | 14 | 24
  MS, Cycle 29 Maintenance: Stable | 16 | 45
  MS, Cycle 29 Maintenance: Improved | 20 | 25
  CSE, Cycle 29 Maintenance: number analyzed (Participants) | 50 | 94
  CSE, Cycle 29 Maintenance: Worsened | 7 | 19
  CSE, Cycle 29 Maintenance: Stable | 30 | 54
  CSE, Cycle 29 Maintenance: Improved | 13 | 21
  HS, Cycle 29 Maintenance: number analyzed (Participants) | 50 | 93
  HS, Cycle 29 Maintenance: Worsened | 1 | 6
  HS, Cycle 29 Maintenance: Stable | 14 | 19
  HS, Cycle 29 Maintenance: Improved | 35 | 68
  BI, Cycle 35 Maintenance: number analyzed (Participants) | 45 | 85
  BI, Cycle 35 Maintenance: Worsened | 13 | 19
  BI, Cycle 35 Maintenance: Stable | 11 | 35
  BI, Cycle 35 Maintenance: Improved | 21 | 31
  S, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 80
  S, Cycle 35 Maintenance: Worsened | 5 | 12
  S, Cycle 35 Maintenance: Stable | 26 | 47
  S, Cycle 35 Maintenance: Improved | 13 | 21
  ATD, Cycle 35 Maintenance: number analyzed (Participants) | 45 | 84
  ATD, Cycle 35 Maintenance: Worsened | 9 | 20
  ATD, Cycle 35 Maintenance: Stable | 11 | 14
  ATD, Cycle 35 Maintenance: Improved | 25 | 50
  AS, Cycle 35 Maintenance: number analyzed (Participants) | 44 | 86
  AS, Cycle 35 Maintenance: Worsened | 6 | 15
  AS, Cycle 35 Maintenance: Stable | 25 | 48
  AS, Cycle 35 Maintenance: Improved | 13 | 23
  PN, Cycle 35 Maintenance: number analyzed (Participants) | 45 | 86
  PN, Cycle 35 Maintenance: Worsened | 14 | 33
  PN, Cycle 35 Maintenance: Stable | 19 | 28
  PN, Cycle 35 Maintenance: Improved | 12 | 25
  MS, Cycle 35 Maintenance: number analyzed (Participants) | 45 | 86
  MS, Cycle 35 Maintenance: Worsened | 9 | 26
  MS, Cycle 35 Maintenance: Stable | 17 | 38
  MS, Cycle 35 Maintenance: Improved | 19 | 22
  CSE, Cycle 35 Maintenance: number analyzed (Participants) | 45 | 86
  CSE, Cycle 35 Maintenance: Worsened | 10 | 18
  CSE, Cycle 35 Maintenance: Stable | 24 | 42
  CSE, Cycle 35 Maintenance: Improved | 11 | 26
  HS, Cycle 35 Maintenance: number analyzed (Participants) | 45 | 84
  HS, Cycle 35 Maintenance: Worsened | 2 | 6
  HS, Cycle 35 Maintenance: Stable | 15 | 14
  HS, Cycle 35 Maintenance: Improved | 28 | 64
  BI, Cycle 41 Maintenance: number analyzed (Participants) | 57 | 104
  BI, Cycle 41 Maintenance: Worsened | 23 | 30
  BI, Cycle 41 Maintenance: Stable | 15 | 36
  BI, Cycle 41 Maintenance: Improved | 19 | 38
  S, Cycle 41 Maintenance: number analyzed (Participants) | 57 | 101
  S, Cycle 41 Maintenance: Worsened | 6 | 14
  S, Cycle 41 Maintenance: Stable | 30 | 53
  S, Cycle 41 Maintenance: Improved | 21 | 34
  ATD, Cycle 41 Maintenance: number analyzed (Participants) | 57 | 104
  ATD, Cycle 41 Maintenance: Worsened | 10 | 26
  ATD, Cycle 41 Maintenance: Stable | 13 | 21
  ATD, Cycle 41 Maintenance: Improved | 34 | 57
  AS, Cycle 41 Maintenance: number analyzed (Participants) | 57 | 104
  AS, Cycle 41 Maintenance: Worsened | 11 | 16
  AS, Cycle 41 Maintenance: Stable | 31 | 52
  AS, Cycle 41 Maintenance: Improved | 15 | 36
  PN, Cycle 41 Maintenance: number analyzed (Participants) | 56 | 103
  PN, Cycle 41 Maintenance: Worsened | 25 | 52
  PN, Cycle 41 Maintenance: Stable | 19 | 27
  PN, Cycle 41 Maintenance: Improved | 12 | 24
  MS, Cycle 41 Maintenance: number analyzed (Participants) | 56 | 103
  MS, Cycle 41 Maintenance: Worsened | 18 | 29
  MS, Cycle 41 Maintenance: Stable | 19 | 51
  MS, Cycle 41 Maintenance: Improved | 19 | 23
  CSE, Cycle 41 Maintenance: number analyzed (Participants) | 56 | 103
  CSE, Cycle 41 Maintenance: Worsened | 15 | 20
  CSE, Cycle 41 Maintenance: Stable | 26 | 50
  CSE, Cycle 41 Maintenance: Improved | 15 | 33
  HS, Cycle 41 Maintenance: number analyzed (Participants) | 57 | 103
  HS, Cycle 41 Maintenance: Worsened | 3 | 9
  HS, Cycle 41 Maintenance: Stable | 17 | 17
  HS, Cycle 41 Maintenance: Improved | 37 | 77
  BI, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 86
  BI, Cycle 47 Maintenance: Worsened | 14 | 19
  BI, Cycle 47 Maintenance: Stable | 18 | 34
  BI, Cycle 47 Maintenance: Improved | 15 | 33
  S, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 79
  S, Cycle 47 Maintenance: Worsened | 6 | 6
  S, Cycle 47 Maintenance: Stable | 21 | 46
  S, Cycle 47 Maintenance: Improved | 20 | 27
  ATD, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 85
  ATD, Cycle 47 Maintenance: Worsened | 7 | 19
  ATD, Cycle 47 Maintenance: Stable | 9 | 19
  ATD, Cycle 47 Maintenance: Improved | 31 | 47
  AS, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 86
  AS, Cycle 47 Maintenance: Worsened | 10 | 16
  AS, Cycle 47 Maintenance: Stable | 28 | 44
  AS, Cycle 47 Maintenance: Improved | 9 | 26
  PN, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 86
  PN, Cycle 47 Maintenance: Worsened | 21 | 40
  PN, Cycle 47 Maintenance: Stable | 14 | 25
  PN, Cycle 47 Maintenance: Improved | 12 | 21
  MS, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 86
  MS, Cycle 47 Maintenance: Worsened | 12 | 24
  MS, Cycle 47 Maintenance: Stable | 19 | 43
  MS, Cycle 47 Maintenance: Improved | 16 | 19
  CSE, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 86
  CSE, Cycle 47 Maintenance: Worsened | 9 | 18
  CSE, Cycle 47 Maintenance: Stable | 29 | 44
  CSE, Cycle 47 Maintenance: Improved | 9 | 24
  HS, Cycle 47 Maintenance: number analyzed (Participants) | 47 | 82
  HS, Cycle 47 Maintenance: Worsened | 5 | 6
  HS, Cycle 47 Maintenance: Stable | 12 | 16
  HS, Cycle 47 Maintenance: Improved | 30 | 60
  BI, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  BI, Cycle 53 Maintenance: Worsened | 10 | 14
  BI, Cycle 53 Maintenance: Stable | 8 | 20
  BI, Cycle 53 Maintenance: Improved | 8 | 20
  S, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 51
  S, Cycle 53 Maintenance: Worsened | 4 | 5
  S, Cycle 53 Maintenance: Stable | 11 | 32
  S, Cycle 53 Maintenance: Improved | 11 | 14
  ATD, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  ATD, Cycle 53 Maintenance: Worsened | 3 | 12
  ATD, Cycle 53 Maintenance: Stable | 5 | 9
  ATD, Cycle 53 Maintenance: Improved | 18 | 33
  AS, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  AS, Cycle 53 Maintenance: Worsened | 5 | 11
  AS, Cycle 53 Maintenance: Stable | 15 | 33
  AS, Cycle 53 Maintenance: Improved | 6 | 10
  PN, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 53
  PN, Cycle 53 Maintenance: Worsened | 7 | 27
  PN, Cycle 53 Maintenance: Stable | 13 | 15
  PN, Cycle 53 Maintenance: Improved | 6 | 11
  MS, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 53
  MS, Cycle 53 Maintenance: Worsened | 7 | 24
  MS, Cycle 53 Maintenance: Stable | 9 | 18
  MS, Cycle 53 Maintenance: Improved | 10 | 11
  CSE, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 53
  CSE, Cycle 53 Maintenance: Worsened | 4 | 11
  CSE, Cycle 53 Maintenance: Stable | 14 | 33
  CSE, Cycle 53 Maintenance: Improved | 8 | 9
  HS, Cycle 53 Maintenance: number analyzed (Participants) | 26 | 54
  HS, Cycle 53 Maintenance: Worsened | 4 | 2
  HS, Cycle 53 Maintenance: Stable | 8 | 11
  HS, Cycle 53 Maintenance: Improved | 14 | 41
  BI, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  BI, Cycle 59 Maintenance: Worsened | 6 | 7
  BI, Cycle 59 Maintenance: Stable | 6 | 11
  BI, Cycle 59 Maintenance: Improved | 6 | 17
  S, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 34
  S, Cycle 59 Maintenance: Worsened | 1 | 3
  S, Cycle 59 Maintenance: Stable | 9 | 20
  S, Cycle 59 Maintenance: Improved | 8 | 11
  ATD, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  ATD, Cycle 59 Maintenance: Worsened | 3 | 4
  ATD, Cycle 59 Maintenance: Stable | 5 | 6
  ATD, Cycle 59 Maintenance: Improved | 10 | 25
  AS, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  AS, Cycle 59 Maintenance: Worsened | 3 | 6
  AS, Cycle 59 Maintenance: Stable | 12 | 20
  AS, Cycle 59 Maintenance: Improved | 3 | 9
  PN, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  PN, Cycle 59 Maintenance: Worsened | 7 | 15
  PN, Cycle 59 Maintenance: Stable | 6 | 12
  PN, Cycle 59 Maintenance: Improved | 5 | 8
  MS, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  MS, Cycle 59 Maintenance: Worsened | 5 | 9
  MS, Cycle 59 Maintenance: Stable | 6 | 17
  MS, Cycle 59 Maintenance: Improved | 7 | 9
  CSE, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  CSE, Cycle 59 Maintenance: Worsened | 3 | 6
  CSE, Cycle 59 Maintenance: Stable | 10 | 22
  CSE, Cycle 59 Maintenance: Improved | 5 | 7
  HS, Cycle 59 Maintenance: number analyzed (Participants) | 18 | 35
  HS, Cycle 59 Maintenance: Worsened | 4 | 3
  HS, Cycle 59 Maintenance: Stable | 4 | 6
  HS, Cycle 59 Maintenance: Improved | 10 | 26
  BI, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 25
  BI, Cycle 65 Maintenance: Worsened | 3 | 4
  BI, Cycle 65 Maintenance: Stable | 4 | 10
  BI, Cycle 65 Maintenance: Improved | 5 | 11
  S, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 24
  S, Cycle 65 Maintenance: Worsened | 2 | 3
  S, Cycle 65 Maintenance: Stable | 5 | 12
  S, Cycle 65 Maintenance: Improved | 5 | 9
  ATD, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 25
  ATD, Cycle 65 Maintenance: Worsened | 1 | 5
  ATD, Cycle 65 Maintenance: Stable | 5 | 5
  ATD, Cycle 65 Maintenance: Improved | 6 | 15
  AS, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 25
  AS, Cycle 65 Maintenance: Worsened | 2 | 4
  AS, Cycle 65 Maintenance: Stable | 9 | 17
  AS, Cycle 65 Maintenance: Improved | 1 | 4
  PN, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 25
  PN, Cycle 65 Maintenance: Worsened | 5 | 9
  PN, Cycle 65 Maintenance: Stable | 5 | 9
  PN, Cycle 65 Maintenance: Improved | 2 | 7
  MS, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 25
  MS, Cycle 65 Maintenance: Worsened | 3 | 6
  MS, Cycle 65 Maintenance: Stable | 3 | 14
  MS, Cycle 65 Maintenance: Improved | 6 | 5
  CSE, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 25
  CSE, Cycle 65 Maintenance: Worsened | 2 | 5
  CSE, Cycle 65 Maintenance: Stable | 9 | 14
  CSE, Cycle 65 Maintenance: Improved | 1 | 6
  HS, Cycle 65 Maintenance: number analyzed (Participants) | 12 | 25
  HS, Cycle 65 Maintenance: Worsened | 4 | 2
  HS, Cycle 65 Maintenance: Stable | 4 | 3
  HS, Cycle 65 Maintenance: Improved | 4 | 20
  BI, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 13
  BI, Cycle 71 Maintenance: Worsened | 1 | 3
  BI, Cycle 71 Maintenance: Stable | 1 | 6
  BI, Cycle 71 Maintenance: Improved | 6 | 4
  S, Cycle 71 Maintenance: number analyzed (Participants) | 7 | 13
  S, Cycle 71 Maintenance: Worsened | 2 | 0
  S, Cycle 71 Maintenance: Stable | 4 | 10
  S, Cycle 71 Maintenance: Improved | 1 | 3
  ATD, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 13
  ATD, Cycle 71 Maintenance: Worsened | 1 | 2
  ATD, Cycle 71 Maintenance: Stable | 1 | 4
  ATD, Cycle 71 Maintenance: Improved | 6 | 7
  AS, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 13
  AS, Cycle 71 Maintenance: Worsened | 3 | 1
  AS, Cycle 71 Maintenance: Stable | 4 | 11
  AS, Cycle 71 Maintenance: Improved | 1 | 1
  PN, Cycle 71 Maintenance: number analyzed (Participants) | 7 | 13
  PN, Cycle 71 Maintenance: Worsened | 2 | 6
  PN, Cycle 71 Maintenance: Stable | 4 | 4
  PN, Cycle 71 Maintenance: Improved | 1 | 3
  MS, Cycle 71 Maintenance: number analyzed (Participants) | 7 | 13
  MS, Cycle 71 Maintenance: Worsened | 1 | 3
  MS, Cycle 71 Maintenance: Stable | 1 | 7
  MS, Cycle 71 Maintenance: Improved | 5 | 3
  CSE, Cycle 71 Maintenance: number analyzed (Participants) | 7 | 13
  CSE, Cycle 71 Maintenance: Worsened | 1 | 1
  CSE, Cycle 71 Maintenance: Stable | 5 | 10
  CSE, Cycle 71 Maintenance: Improved | 1 | 2
  HS, Cycle 71 Maintenance: number analyzed (Participants) | 8 | 13
  HS, Cycle 71 Maintenance: Worsened | 3 | 0
  HS, Cycle 71 Maintenance: Stable | 2 | 5
  HS, Cycle 71 Maintenance: Improved | 3 | 8
  BI, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  BI, Cycle 77 Maintenance: Worsened | 1 | 3
  BI, Cycle 77 Maintenance: Stable | 1 | 2
  BI, Cycle 77 Maintenance: Improved | 2 | 6
  S, Cycle 77 Maintenance: number analyzed (Participants) | 3 | 11
  S, Cycle 77 Maintenance: Worsened | 1 | 2
  S, Cycle 77 Maintenance: Stable | 2 | 4
  S, Cycle 77 Maintenance: Improved | 0 | 5
  ATD, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  ATD, Cycle 77 Maintenance: Worsened | 0 | 2
  ATD, Cycle 77 Maintenance: Stable | 1 | 1
  ATD, Cycle 77 Maintenance: Improved | 3 | 8
  AS, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  AS, Cycle 77 Maintenance: Worsened | 0 | 2
  AS, Cycle 77 Maintenance: Stable | 2 | 6
  AS, Cycle 77 Maintenance: Improved | 2 | 3
  PN, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  PN, Cycle 77 Maintenance: Worsened | 2 | 6
  PN, Cycle 77 Maintenance: Stable | 1 | 1
  PN, Cycle 77 Maintenance: Improved | 1 | 4
  MS, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  MS, Cycle 77 Maintenance: Worsened | 0 | 5
  MS, Cycle 77 Maintenance: Stable | 0 | 4
  MS, Cycle 77 Maintenance: Improved | 4 | 2
  CSE, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  CSE, Cycle 77 Maintenance: Worsened | 1 | 1
  CSE, Cycle 77 Maintenance: Stable | 2 | 8
  CSE, Cycle 77 Maintenance: Improved | 1 | 2
  HS, Cycle 77 Maintenance: number analyzed (Participants) | 4 | 11
  HS, Cycle 77 Maintenance: Worsened | 0 | 3
  HS, Cycle 77 Maintenance: Stable | 2 | 1
  HS, Cycle 77 Maintenance: Improved | 2 | 7
  BI, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 5
  BI, Cycle 83 Maintenance: Worsened | 1 | 1
  BI, Cycle 83 Maintenance: Stable | 0 | 0
  BI, Cycle 83 Maintenance: Improved | 2 | 4
  S, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 5
  S, Cycle 83 Maintenance: Worsened | 1 | 1
  S, Cycle 83 Maintenance: Stable | 1 | 0
  S, Cycle 83 Maintenance: Improved | 1 | 4
  ATD, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 5
  ATD, Cycle 83 Maintenance: Worsened | 0 | 0
  ATD, Cycle 83 Maintenance: Stable | 1 | 0
  ATD, Cycle 83 Maintenance: Improved | 2 | 5
  AS, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 5
  AS, Cycle 83 Maintenance: Worsened | 0 | 0
  AS, Cycle 83 Maintenance: Stable | 2 | 4
  AS, Cycle 83 Maintenance: Improved | 1 | 1
  PN, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 5
  PN, Cycle 83 Maintenance: Worsened | 0 | 1
  PN, Cycle 83 Maintenance: Stable | 1 | 0
  PN, Cycle 83 Maintenance: Improved | 2 | 4
  MS, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 5
  MS, Cycle 83 Maintenance: Worsened | 0 | 1
  MS, Cycle 83 Maintenance: Stable | 0 | 4
  MS, Cycle 83 Maintenance: Improved | 3 | 0
  CSE, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 5
  CSE, Cycle 83 Maintenance: Worsened | 1 | 0
  CSE, Cycle 83 Maintenance: Stable | 1 | 2
  CSE, Cycle 83 Maintenance: Improved | 1 | 3
  HS, Cycle 83 Maintenance: number analyzed (Participants) | 3 | 5
  HS, Cycle 83 Maintenance: Worsened | 0 | 1
  HS, Cycle 83 Maintenance: Stable | 2 | 0
  HS, Cycle 83 Maintenance: Improved | 1 | 4
  BI, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  BI, Cycle 89 Maintenance: Worsened | 0 | 0
  BI, Cycle 89 Maintenance: Stable | 0 | 0
  BI, Cycle 89 Maintenance: Improved | 0 | 2
  S, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 1
  S, Cycle 89 Maintenance: Worsened | 0 | 0
  S, Cycle 89 Maintenance: Stable | 0 | 0
  S, Cycle 89 Maintenance: Improved | 0 | 1
  ATD, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  ATD, Cycle 89 Maintenance: Worsened | 0 | 0
  ATD, Cycle 89 Maintenance: Stable | 0 | 0
  ATD, Cycle 89 Maintenance: Improved | 0 | 2
  AS, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  AS, Cycle 89 Maintenance: Worsened | 0 | 0
  AS, Cycle 89 Maintenance: Stable | 0 | 0
  AS, Cycle 89 Maintenance: Improved | 0 | 2
  PN, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  PN, Cycle 89 Maintenance: Worsened | 0 | 0
  PN, Cycle 89 Maintenance: Stable | 0 | 1
  PN, Cycle 89 Maintenance: Improved | 0 | 1
  MS, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  MS, Cycle 89 Maintenance: Worsened | 0 | 0
  MS, Cycle 89 Maintenance: Stable | 0 | 2
  MS, Cycle 89 Maintenance: Improved | 0 | 0
  CSE, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  CSE, Cycle 89 Maintenance: Worsened | 0 | 0
  CSE, Cycle 89 Maintenance: Stable | 0 | 0
  CSE, Cycle 89 Maintenance: Improved | 0 | 2
  HS, Cycle 89 Maintenance: number analyzed (Participants) | 0 | 2
  HS, Cycle 89 Maintenance: Worsened | 0 | 0
  HS, Cycle 89 Maintenance: Stable | 0 | 0
  HS, Cycle 89 Maintenance: Improved | 0 | 2
  BI, End of treatment: number analyzed (Participants) | 181 | 337
  BI, End of treatment: Worsened | 45 | 94
  BI, End of treatment: Stable | 68 | 109
  BI, End of treatment: Improved | 68 | 134
  S, End of treatment: number analyzed (Participants) | 176 | 324
  S, End of treatment: Worsened | 21 | 52
  S, End of treatment: Stable | 122 | 206
  S, End of treatment: Improved | 33 | 66
  ATD, End of treatment: number analyzed (Participants) | 180 | 338
  ATD, End of treatment: Worsened | 65 | 124
  ATD, End of treatment: Stable | 43 | 72
  ATD, End of treatment: Improved | 72 | 142
  AS, End of treatment: number analyzed (Participants) | 181 | 341
  AS, End of treatment: Worsened | 45 | 59
  AS, End of treatment: Stable | 90 | 186
  AS, End of treatment: Improved | 46 | 96
  PN, End of treatment: number analyzed (Participants) | 181 | 339
  PN, End of treatment: Worsened | 79 | 171
  PN, End of treatment: Stable | 52 | 83
  PN, End of treatment: Improved | 50 | 85
  MS, End of treatment: number analyzed (Participants) | 181 | 340
  MS, End of treatment: Worsened | 42 | 97
  MS, End of treatment: Stable | 83 | 149
  MS, End of treatment: Improved | 56 | 94
  CSE, End of treatment: number analyzed (Participants) | 181 | 340
  CSE, End of treatment: Worsened | 35 | 75
  CSE, End of treatment: Stable | 94 | 180
  CSE, End of treatment: Improved | 52 | 85
  HS, End of treatment: number analyzed (Participants) | 180 | 340
  HS, End of treatment: Worsened | 13 | 24
  HS, End of treatment: Stable | 45 | 76
  HS, End of treatment: Improved | 122 | 240
  BI, Safety Follow-up: number analyzed (Participants) | 141 | 280
  BI, Safety Follow-up: Worsened | 42 | 94
  BI, Safety Follow-up: Stable | 47 | 84
  BI, Safety Follow-up: Improved | 52 | 102
  S, Safety Follow-up: number analyzed (Participants) | 134 | 272
  S, Safety Follow-up: Worsened | 16 | 42
  S, Safety Follow-up: Stable | 90 | 175
  S, Safety Follow-up: Improved | 28 | 55
  ATD, Safety Follow-up: number analyzed (Participants) | 141 | 281
  ATD, Safety Follow-up: Worsened | 50 | 111
  ATD, Safety Follow-up: Stable | 32 | 67
  ATD, Safety Follow-up: Improved | 59 | 103
  AS, Safety Follow-up: number analyzed (Participants) | 143 | 282
  AS, Safety Follow-up: Worsened | 22 | 55
  AS, Safety Follow-up: Stable | 78 | 152
  AS, Safety Follow-up: Improved | 43 | 75
  PN, Safety Follow-up: number analyzed (Participants) | 143 | 282
  PN, Safety Follow-up: Worsened | 72 | 151
  PN, Safety Follow-up: Stable | 36 | 70
  PN, Safety Follow-up: Improved | 35 | 61
  MS, Safety Follow-up: number analyzed (Participants) | 143 | 282
  MS, Safety Follow-up: Worsened | 29 | 83
  MS, Safety Follow-up: Stable | 67 | 130
  MS, Safety Follow-up: Improved | 47 | 69
  CSE, Safety Follow-up: number analyzed (Participants) | 143 | 282
  CSE, Safety Follow-up: Worsened | 29 | 66
  CSE, Safety Follow-up: Stable | 77 | 139
  CSE, Safety Follow-up: Improved | 37 | 77
  HS, Safety Follow-up: number analyzed (Participants) | 142 | 281
  HS, Safety Follow-up: Worsened | 15 | 26
  HS, Safety Follow-up: Stable | 37 | 52
  HS, Safety Follow-up: Improved | 90 | 203
  BI, LTFU (EOT + 3 months): number analyzed (Participants) | 134 | 243
  BI, LTFU (EOT + 3 months): Worsened | 47 | 79
  BI, LTFU (EOT + 3 months): Stable | 46 | 83
  BI, LTFU (EOT + 3 months): Improved | 41 | 81
  S, LTFU (EOT + 3 months): number analyzed (Participants) | 128 | 234
  S, LTFU (EOT + 3 months): Worsened | 24 | 35
  S, LTFU (EOT + 3 months): Stable | 79 | 157
  S, LTFU (EOT + 3 months): Improved | 25 | 42
  ATD, LTFU (EOT + 3 months): number analyzed (Participants) | 134 | 243
  ATD, LTFU (EOT + 3 months): Worsened | 46 | 88
  ATD, LTFU (EOT + 3 months): Stable | 33 | 47
  ATD, LTFU (EOT + 3 months): Improved | 55 | 108
  AS, LTFU (EOT + 3 months): number analyzed (Participants) | 134 | 243
  AS, LTFU (EOT + 3 months): Worsened | 23 | 44
  AS, LTFU (EOT + 3 months): Stable | 68 | 132
  AS, LTFU (EOT + 3 months): Improved | 43 | 67
  PN, LTFU (EOT + 3 months): number analyzed (Participants) | 134 | 243
  PN, LTFU (EOT + 3 months): Worsened | 63 | 135
  PN, LTFU (EOT + 3 months): Stable | 39 | 56
  PN, LTFU (EOT + 3 months): Improved | 32 | 52
  MS, LTFU (EOT + 3 months): number analyzed (Participants) | 134 | 242
  MS, LTFU (EOT + 3 months): Worsened | 27 | 56
  MS, LTFU (EOT + 3 months): Stable | 52 | 108
  MS, LTFU (EOT + 3 months): Improved | 55 | 78
  CSE, LTFU (EOT + 3 months): number analyzed (Participants) | 134 | 243
  CSE, LTFU (EOT + 3 months): Worsened | 30 | 67
  CSE, LTFU (EOT + 3 months): Stable | 79 | 116
  CSE, LTFU (EOT + 3 months): Improved | 25 | 60
  HS, LTFU (EOT + 3 months): number analyzed (Participants) | 132 | 240
  HS, LTFU (EOT + 3 months): Worsened | 17 | 25
  HS, LTFU (EOT + 3 months): Stable | 29 | 42
  HS, LTFU (EOT + 3 months): Improved | 86 | 173
  BI, LTFU (EOT + 9 months): number analyzed (Participants) | 107 | 180
  BI, LTFU (EOT + 9 months): Worsened | 36 | 56
  BI, LTFU (EOT + 9 months): Stable | 37 | 56
  BI, LTFU (EOT + 9 months): Improved | 34 | 68
  S, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 172
  S, LTFU (EOT + 9 months): Worsened | 13 | 31
  S, LTFU (EOT + 9 months): Stable | 74 | 110
  S, LTFU (EOT + 9 months): Improved | 19 | 31
  ATD, LTFU (EOT + 9 months): number analyzed (Participants) | 106 | 179
  ATD, LTFU (EOT + 9 months): Worsened | 42 | 67
  ATD, LTFU (EOT + 9 months): Stable | 17 | 28
  ATD, LTFU (EOT + 9 months): Improved | 47 | 84
  AS, LTFU (EOT + 9 months): number analyzed (Participants) | 107 | 180
  AS, LTFU (EOT + 9 months): Worsened | 18 | 35
  AS, LTFU (EOT + 9 months): Stable | 58 | 86
  AS, LTFU (EOT + 9 months): Improved | 31 | 59
  PN, LTFU (EOT + 9 months): number analyzed (Participants) | 107 | 180
  PN, LTFU (EOT + 9 months): Worsened | 60 | 92
  PN, LTFU (EOT + 9 months): Stable | 24 | 47
  PN, LTFU (EOT + 9 months): Improved | 23 | 41
  MS, LTFU (EOT + 9 months): number analyzed (Participants) | 107 | 180
  MS, LTFU (EOT + 9 months): Worsened | 22 | 38
  MS, LTFU (EOT + 9 months): Stable | 50 | 82
  MS, LTFU (EOT + 9 months): Improved | 35 | 60
  CSE, LTFU (EOT + 9 months): number analyzed (Participants) | 107 | 180
  CSE, LTFU (EOT + 9 months): Worsened | 32 | 48
  CSE, LTFU (EOT + 9 months): Stable | 54 | 88
  CSE, LTFU (EOT + 9 months): Improved | 21 | 44
  HS, LTFU (EOT + 9 months): number analyzed (Participants) | 107 | 179
  HS, LTFU (EOT + 9 months): Worsened | 12 | 16
  HS, LTFU (EOT + 9 months): Stable | 26 | 40
  HS, LTFU (EOT + 9 months): Improved | 69 | 123
  BI, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 149
  BI, LTFU (EOT + 15 months): Worsened | 22 | 42
  BI, LTFU (EOT + 15 months): Stable | 31 | 46
  BI, LTFU (EOT + 15 months): Improved | 23 | 61
  S, LTFU (EOT + 15 months): number analyzed (Participants) | 70 | 143
  S, LTFU (EOT + 15 months): Worsened | 12 | 26
  S, LTFU (EOT + 15 months): Stable | 43 | 86
  S, LTFU (EOT + 15 months): Improved | 15 | 31
  ATD, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 148
  ATD, LTFU (EOT + 15 months): Worsened | 30 | 54
  ATD, LTFU (EOT + 15 months): Stable | 16 | 33
  ATD, LTFU (EOT + 15 months): Improved | 30 | 61
  AS, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 149
  AS, LTFU (EOT + 15 months): Worsened | 19 | 23
  AS, LTFU (EOT + 15 months): Stable | 37 | 81
  AS, LTFU (EOT + 15 months): Improved | 20 | 45
  PN, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 146
  PN, LTFU (EOT + 15 months): Worsened | 43 | 79
  PN, LTFU (EOT + 15 months): Stable | 13 | 40
  PN, LTFU (EOT + 15 months): Improved | 20 | 27
  MS, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 149
  MS, LTFU (EOT + 15 months): Worsened | 17 | 37
  MS, LTFU (EOT + 15 months): Stable | 41 | 78
  MS, LTFU (EOT + 15 months): Improved | 18 | 34
  CSE, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 147
  CSE, LTFU (EOT + 15 months): Worsened | 19 | 45
  CSE, LTFU (EOT + 15 months): Stable | 41 | 73
  CSE, LTFU (EOT + 15 months): Improved | 16 | 29
  HS, LTFU (EOT + 15 months): number analyzed (Participants) | 76 | 148
  HS, LTFU (EOT + 15 months): Worsened | 7 | 13
  HS, LTFU (EOT + 15 months): Stable | 21 | 34
  HS, LTFU (EOT + 15 months): Improved | 48 | 101
  BI, LTFU (EOT + 21 months): number analyzed (Participants) | 46 | 96
  BI, LTFU (EOT + 21 months): Worsened | 12 | 26
  BI, LTFU (EOT + 21 months): Stable | 18 | 31
  BI, LTFU (EOT + 21 months): Improved | 16 | 39
  S, LTFU (EOT + 21 months): number analyzed (Participants) | 44 | 93
  S, LTFU (EOT + 21 months): Worsened | 5 | 13
  S, LTFU (EOT + 21 months): Stable | 26 | 62
  S, LTFU (EOT + 21 months): Improved | 13 | 18
  ATD, LTFU (EOT + 21 months): number analyzed (Participants) | 46 | 96
  ATD, LTFU (EOT + 21 months): Worsened | 17 | 36
  ATD, LTFU (EOT + 21 months): Stable | 11 | 18
  ATD, LTFU (EOT + 21 months): Improved | 18 | 42
  AS, LTFU (EOT + 21 months): number analyzed (Participants) | 47 | 96
  AS, LTFU (EOT + 21 months): Worsened | 12 | 19
  AS, LTFU (EOT + 21 months): Stable | 25 | 48
  AS, LTFU (EOT + 21 months): Improved | 10 | 29
  PN, LTFU (EOT + 21 months): number analyzed (Participants) | 46 | 96
  PN, LTFU (EOT + 21 months): Worsened | 18 | 53
  PN, LTFU (EOT + 21 months): Stable | 13 | 25
  PN, LTFU (EOT + 21 months): Improved | 15 | 18
  MS, LTFU (EOT + 21 months): number analyzed (Participants) | 47 | 96
  MS, LTFU (EOT + 21 months): Worsened | 12 | 25
  MS, LTFU (EOT + 21 months): Stable | 21 | 44
  MS, LTFU (EOT + 21 months): Improved | 14 | 27
  CSE, LTFU (EOT + 21 months): number analyzed (Participants) | 46 | 96
  CSE, LTFU (EOT + 21 months): Worsened | 10 | 25
  CSE, LTFU (EOT + 21 months): Stable | 27 | 50
  CSE, LTFU (EOT + 21 months): Improved | 9 | 21
  HS, LTFU (EOT + 21 months): number analyzed (Participants) | 47 | 95
  HS, LTFU (EOT + 21 months): Worsened | 4 | 11
  HS, LTFU (EOT + 21 months): Stable | 6 | 22
  HS, LTFU (EOT + 21 months): Improved | 37 | 62
  BI, LTFU (EOT + 27 months): number analyzed (Participants) | 35 | 69
  BI, LTFU (EOT + 27 months): Worsened | 10 | 21
  BI, LTFU (EOT + 27 months): Stable | 15 | 22
  BI, LTFU (EOT + 27 months): Improved | 10 | 26
  S, LTFU (EOT + 27 months): number analyzed (Participants) | 32 | 66
  S, LTFU (EOT + 27 months): Worsened | 6 | 9
  S, LTFU (EOT + 27 months): Stable | 18 | 41
  S, LTFU (EOT + 27 months): Improved | 8 | 16
  ATD, LTFU (EOT + 27 months): number analyzed (Participants) | 34 | 69
  ATD, LTFU (EOT + 27 months): Worsened | 16 | 28
  ATD, LTFU (EOT + 27 months): Stable | 7 | 14
  ATD, LTFU (EOT + 27 months): Improved | 11 | 27
  AS, LTFU (EOT + 27 months): number analyzed (Participants) | 35 | 69
  AS, LTFU (EOT + 27 months): Worsened | 5 | 15
  AS, LTFU (EOT + 27 months): Stable | 21 | 38
  AS, LTFU (EOT + 27 months): Improved | 9 | 16
  PN, LTFU (EOT + 27 months): number analyzed (Participants) | 35 | 69
  PN, LTFU (EOT + 27 months): Worsened | 19 | 36
  PN, LTFU (EOT + 27 months): Stable | 9 | 16
  PN, LTFU (EOT + 27 months): Improved | 7 | 17
  MS, LTFU (EOT + 27 months): number analyzed (Participants) | 35 | 69
  MS, LTFU (EOT + 27 months): Worsened | 8 | 17
  MS, LTFU (EOT + 27 months): Stable | 18 | 29
  MS, LTFU (EOT + 27 months): Improved | 9 | 23
  CSE, LTFU (EOT + 27 months): number analyzed (Participants) | 35 | 69
  CSE, LTFU (EOT + 27 months): Worsened | 11 | 24
  CSE, LTFU (EOT + 27 months): Stable | 18 | 31
  CSE, LTFU (EOT + 27 months): Improved | 6 | 14
  HS, LTFU (EOT + 27 months): number analyzed (Participants) | 35 | 69
  HS, LTFU (EOT + 27 months): Worsened | 6 | 8
  HS, LTFU (EOT + 27 months): Stable | 7 | 14
  HS, LTFU (EOT + 27 months): Improved | 22 | 47
  BI, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  BI, LTFU (EOT + 33 months): Worsened | 1 | 12
  BI, LTFU (EOT + 33 months): Stable | 8 | 12
  BI, LTFU (EOT + 33 months): Improved | 7 | 15
  S, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 38
  S, LTFU (EOT + 33 months): Worsened | 0 | 6
  S, LTFU (EOT + 33 months): Stable | 13 | 23
  S, LTFU (EOT + 33 months): Improved | 3 | 9
  ATD, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  ATD, LTFU (EOT + 33 months): Worsened | 9 | 15
  ATD, LTFU (EOT + 33 months): Stable | 4 | 6
  ATD, LTFU (EOT + 33 months): Improved | 3 | 18
  AS, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  AS, LTFU (EOT + 33 months): Worsened | 4 | 7
  AS, LTFU (EOT + 33 months): Stable | 7 | 25
  AS, LTFU (EOT + 33 months): Improved | 5 | 7
  PN, LTFU (EOT + 33 months): number analyzed (Participants) | 15 | 39
  PN, LTFU (EOT + 33 months): Worsened | 8 | 19
  PN, LTFU (EOT + 33 months): Stable | 5 | 12
  PN, LTFU (EOT + 33 months): Improved | 2 | 8
  MS, LTFU (EOT + 33 months): number analyzed (Participants) | 16 | 39
  MS, LTFU (EOT + 33 months): Worsened | 2 | 12
  MS, LTFU (EOT + 33 months): Stable | 8 | 17
  MS, LTFU (EOT + 33 months): Improved | 6 | 10
  CSE, LTFU (EOT + 33 months): number analyzed (Participants) | 15 | 39
  CSE, LTFU (EOT + 33 months): Worsened | 4 | 11
  CSE, LTFU (EOT + 33 months): Stable | 7 | 20
  CSE, LTFU (EOT + 33 months): Improved | 4 | 8
  HS, LTFU (EOT + 33 months): number analyzed (Participants) | 15 | 39
  HS, LTFU (EOT + 33 months): Worsened | 1 | 5
  HS, LTFU (EOT + 33 months): Stable | 3 | 11
  HS, LTFU (EOT + 33 months): Improved | 11 | 23
  BI, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  BI, LTFU (EOT + 39 months): Worsened | 3 | 11
  BI, LTFU (EOT + 39 months): Stable | 6 | 6
  BI, LTFU (EOT + 39 months): Improved | 2 | 10
  S, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  S, LTFU (EOT + 39 months): Worsened | 0 | 6
  S, LTFU (EOT + 39 months): Stable | 10 | 18
  S, LTFU (EOT + 39 months): Improved | 1 | 3
  ATD, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  ATD, LTFU (EOT + 39 months): Worsened | 3 | 12
  ATD, LTFU (EOT + 39 months): Stable | 3 | 5
  ATD, LTFU (EOT + 39 months): Improved | 5 | 10
  AS, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  AS, LTFU (EOT + 39 months): Worsened | 2 | 5
  AS, LTFU (EOT + 39 months): Stable | 6 | 18
  AS, LTFU (EOT + 39 months): Improved | 3 | 4
  PN, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  PN, LTFU (EOT + 39 months): Worsened | 5 | 14
  PN, LTFU (EOT + 39 months): Stable | 4 | 8
  PN, LTFU (EOT + 39 months): Improved | 2 | 5
  MS, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  MS, LTFU (EOT + 39 months): Worsened | 4 | 10
  MS, LTFU (EOT + 39 months): Stable | 6 | 10
  MS, LTFU (EOT + 39 months): Improved | 1 | 7
  CSE, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  CSE, LTFU (EOT + 39 months): Worsened | 3 | 8
  CSE, LTFU (EOT + 39 months): Stable | 7 | 14
  CSE, LTFU (EOT + 39 months): Improved | 1 | 5
  HS, LTFU (EOT + 39 months): number analyzed (Participants) | 11 | 27
  HS, LTFU (EOT + 39 months): Worsened | 1 | 3
  HS, LTFU (EOT + 39 months): Stable | 3 | 5
  HS, LTFU (EOT + 39 months): Improved | 7 | 19
  BI, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 16
  BI, LTFU (EOT + 45 months): Worsened | 1 | 6
  BI, LTFU (EOT + 45 months): Stable | 2 | 5
  BI, LTFU (EOT + 45 months): Improved | 1 | 5
  S, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 15
  S, LTFU (EOT + 45 months): Worsened | 1 | 1
  S, LTFU (EOT + 45 months): Stable | 3 | 11
  S, LTFU (EOT + 45 months): Improved | 0 | 3
  ATD, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 16
  ATD, LTFU (EOT + 45 months): Worsened | 3 | 5
  ATD, LTFU (EOT + 45 months): Stable | 0 | 5
  ATD, LTFU (EOT + 45 months): Improved | 1 | 6
  AS, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 16
  AS, LTFU (EOT + 45 months): Worsened | 0 | 4
  AS, LTFU (EOT + 45 months): Stable | 2 | 10
  AS, LTFU (EOT + 45 months): Improved | 2 | 2
  PN, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 16
  PN, LTFU (EOT + 45 months): Worsened | 3 | 11
  PN, LTFU (EOT + 45 months): Stable | 0 | 4
  PN, LTFU (EOT + 45 months): Improved | 1 | 1
  MS, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 16
  MS, LTFU (EOT + 45 months): Worsened | 0 | 6
  MS, LTFU (EOT + 45 months): Stable | 3 | 5
  MS, LTFU (EOT + 45 months): Improved | 1 | 5
  CSE, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 16
  CSE, LTFU (EOT + 45 months): Worsened | 1 | 5
  CSE, LTFU (EOT + 45 months): Stable | 2 | 10
  CSE, LTFU (EOT + 45 months): Improved | 1 | 1
  HS, LTFU (EOT + 45 months): number analyzed (Participants) | 4 | 16
  HS, LTFU (EOT + 45 months): Worsened | 0 | 1
  HS, LTFU (EOT + 45 months): Stable | 3 | 3
  HS, LTFU (EOT + 45 months): Improved | 1 | 12
  BI, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  BI, LTFU (EOT + 51 months): Worsened | 1 | 1
  BI, LTFU (EOT + 51 months): Stable | 1 | 1
  BI, LTFU (EOT + 51 months): Improved | 0 | 3
  S, LTFU (EOT + 51 months): number analyzed (Participants) | 1 | 5
  S, LTFU (EOT + 51 months): Worsened | 1 | 0
  S, LTFU (EOT + 51 months): Stable | 0 | 4
  S, LTFU (EOT + 51 months): Improved | 0 | 1
  ATD, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  ATD, LTFU (EOT + 51 months): Worsened | 2 | 1
  ATD, LTFU (EOT + 51 months): Stable | 0 | 2
  ATD, LTFU (EOT + 51 months): Improved | 0 | 2
  AS, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  AS, LTFU (EOT + 51 months): Worsened | 0 | 0
  AS, LTFU (EOT + 51 months): Stable | 2 | 5
  AS, LTFU (EOT + 51 months): Improved | 0 | 0
  PN, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  PN, LTFU (EOT + 51 months): Worsened | 2 | 2
  PN, LTFU (EOT + 51 months): Stable | 0 | 2
  PN, LTFU (EOT + 51 months): Improved | 0 | 1
  MS, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  MS, LTFU (EOT + 51 months): Worsened | 0 | 1
  MS, LTFU (EOT + 51 months): Stable | 2 | 3
  MS, LTFU (EOT + 51 months): Improved | 0 | 1
  CSE, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  CSE, LTFU (EOT + 51 months): Worsened | 0 | 2
  CSE, LTFU (EOT + 51 months): Stable | 1 | 3
  CSE, LTFU (EOT + 51 months): Improved | 1 | 0
  HS, LTFU (EOT + 51 months): number analyzed (Participants) | 2 | 5
  HS, LTFU (EOT + 51 months): Worsened | 0 | 0
  HS, LTFU (EOT + 51 months): Stable | 1 | 2
  HS, LTFU (EOT + 51 months): Improved | 1 | 3
  BI, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  BI, LTFU (EOT + 57 months): Worsened | 0 | 0
  BI, LTFU (EOT + 57 months): Stable | 1 | 0
  BI, LTFU (EOT + 57 months): Improved | 1 | 1
  S, LTFU (EOT + 57 months): number analyzed (Participants) | 1 | 1
  S, LTFU (EOT + 57 months): Worsened | 1 | 0
  S, LTFU (EOT + 57 months): Stable | 0 | 1
  S, LTFU (EOT + 57 months): Improved | 0 | 0
  ATD, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  ATD, LTFU (EOT + 57 months): Worsened | 0 | 0
  ATD, LTFU (EOT + 57 months): Stable | 2 | 1
  ATD, LTFU (EOT + 57 months): Improved | 0 | 0
  AS, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  AS, LTFU (EOT + 57 months): Worsened | 0 | 0
  AS, LTFU (EOT + 57 months): Stable | 2 | 1
  AS, LTFU (EOT + 57 months): Improved | 0 | 0
  PN, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  PN, LTFU (EOT + 57 months): Worsened | 2 | 1
  PN, LTFU (EOT + 57 months): Stable | 0 | 0
  PN, LTFU (EOT + 57 months): Improved | 0 | 0
  MS, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  MS, LTFU (EOT + 57 months): Worsened | 0 | 0
  MS, LTFU (EOT + 57 months): Stable | 2 | 0
  MS, LTFU (EOT + 57 months): Improved | 0 | 1
  CSE, LTFU (EOT + 57 months): number analyzed (Participants) | 2 | 1
  CSE, LTFU (EOT + 57 months): Worsened | 1 | 0
  CSE, LTFU (EOT + 57 months): Stable | 0 | 1
  CSE, LTFU (EOT + 57 months): Improved | 1 | 0
  HS, LTFU (EOT + 57 months): number analyzed (Participants) | 1 | 1
  HS, LTFU (EOT + 57 months): Worsened | 0 | 0
  HS, LTFU (EOT + 57 months): Stable | 0 | 1
  HS, LTFU (EOT + 57 months): Improved | 1 | 0
  BI, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  BI, LTFU (EOT + 63 months): Worsened | 0 | 0
  BI, LTFU (EOT + 63 months): Stable | 1 | 0
  BI, LTFU (EOT + 63 months): Improved | 0 | 0
  S, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  S, LTFU (EOT + 63 months): Worsened | 1 | 0
  S, LTFU (EOT + 63 months): Stable | 0 | 0
  S, LTFU (EOT + 63 months): Improved | 0 | 0
  ATD, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  ATD, LTFU (EOT + 63 months): Worsened | 0 | 0
  ATD, LTFU (EOT + 63 months): Stable | 1 | 0
  ATD, LTFU (EOT + 63 months): Improved | 0 | 0
  AS, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  AS, LTFU (EOT + 63 months): Worsened | 0 | 0
  AS, LTFU (EOT + 63 months): Stable | 1 | 0
  AS, LTFU (EOT + 63 months): Improved | 0 | 0
  PN, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  PN, LTFU (EOT + 63 months): Worsened | 1 | 0
  PN, LTFU (EOT + 63 months): Stable | 0 | 0
  PN, LTFU (EOT + 63 months): Improved | 0 | 0
  MS, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  MS, LTFU (EOT + 63 months): Worsened | 0 | 0
  MS, LTFU (EOT + 63 months): Stable | 1 | 0
  MS, LTFU (EOT + 63 months): Improved | 0 | 0
  CSE, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  CSE, LTFU (EOT + 63 months): Worsened | 0 | 0
  CSE, LTFU (EOT + 63 months): Stable | 0 | 0
  CSE, LTFU (EOT + 63 months): Improved | 1 | 0
  HS, LTFU (EOT + 63 months): number analyzed (Participants) | 1 | 0
  HS, LTFU (EOT + 63 months): Worsened | 0 | 0
  HS, LTFU (EOT + 63 months): Stable | 0 | 0
  HS, LTFU (EOT + 63 months): Improved | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality, non-serious adverse event (SAEs) and SAEs were collected up to approximately 316 weeks.
Description: All-cause mortality, non-serious adverse events (AEs), and serious adverse events (SAEs) were collected for all enrolled participants, including those who received only standard of care and no study intervention (not treated arm) and those who received at least one dose of a study intervention (arms 1, 2, and 3).
Groups:
- Not Treated: Eligible participants with ovarian cancer received standard of care (SOC) chemotherapy as combination of 175 milligram (mg)/meter^2(m^2) Paclitaxel, area under the curve (AUC) of 5 to 6 mg/millilitre (mL)/minute Carboplatin and optional 7.5 mg/kilogram (kg) or 15 mg/kg Bevacizumab as intravenous (IV) infusion on Day 1 of Cycle 1 in Chemotherapy Run-In Period. They were not randomized to chemotherapy treatment period and no study intervention was administered.
Arm/Group | Not Treated | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib Pbo+Dostarlimab Pbo +/-Bev (Arm1) | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3)
All-Cause Mortality (participants affected / at risk) | 33/79 | 106/159 | 235/417 | 430/745
Serious Adverse Events (participants affected / at risk) | 35/79 | 63/159 | 190/417 | 405/745
Other Adverse Events (participants affected / at risk) | 51/79 | 158/159 | 417/417 | 745/745
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Treated (N=79) | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib Pbo+Dostarlimab Pbo +/-Bev (Arm1) (N=159) | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) (N=417) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3) (N=745)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (7) | 10 (11) | 25 (28)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 4 (5) | 12 (13) | 21 (25)
Intestinal obstruction (Gastrointestinal disorders) | 3 (3) | 3 (3) | 11 (12) | 17 (20)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 9 (12)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5) | 8 (8)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 8 (10)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (5) | 6 (6)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 5 (5)
Ileus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 6 (6)
Subileus (Gastrointestinal disorders) | 2 (3) | 0 (0) | 2 (2) | 3 (4)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 3 (3)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Ascites (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Diaphragmatic hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernial eventration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intestinal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenic colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Retroperitoneal haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasculitis gastrointestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus of small bowel (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2) | 7 (7) | 11 (14)
Sepsis (Infections and infestations) | 2 (3) | 2 (2) | 2 (2) | 11 (11)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (4) | 2 (2) | 12 (15)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2) | 6 (6) | 9 (10)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 5 (6)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Septic shock (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 4 (4)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Urosepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Vascular device infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Escherichia sepsis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Pelvic abscess (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Abdominal infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Clostridial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Device related bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Enterobacter sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Klebsiella sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post procedural infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Splenic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Appendiceal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacterial sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clostridial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis intestinal perforated (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endocarditis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis shigella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemophilus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected lymphocele (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infected seroma (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Legionella infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Listeria sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meningitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meningoencephalitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neutropenic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pseudomonas infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stoma site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdiaphragmatic abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection pseudomonal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 25 (27) | 31 (35)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 19 (24) | 28 (30)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 2 (2) | 6 (6) | 20 (20)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (3) | 8 (9) | 7 (7)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 6 (6) | 6 (6)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Aplasia pure red cell (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acquired amegakaryocytic thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atypical haemolytic uraemic syndrome (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Splenic haematoma (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 7 (7) | 13 (14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 7 (7) | 10 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 10 (10)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 8 (8)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary amyloidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 4 (5) | 2 (2) | 21 (23)
Asthenia (General disorders) | 0 (0) | 1 (1) | 4 (5) | 7 (7)
General physical health deterioration (General disorders) | 0 (0) | 0 (0) | 4 (4) | 4 (5)
Mucosal inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperthermia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Inflammation (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hernia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hernia obstructive (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Performance status decreased (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 1 (1) | 1 (1) | 10 (12) | 28 (30)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 8 (8)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
General physical condition abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 6 (7) | 9 (10)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (5)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Calciphylaxis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
Postoperative ileus (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Failure to anastomose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural intestinal perforation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 6 (6)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 5 (6)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Facial paralysis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myasthenic syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Optic neuritis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parkinsonism (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIth nerve paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Embolism (Vascular disorders) | 1 (1) | 0 (0) | 4 (4) | 4 (4)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (6)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 4 (4)
Hypotension (Vascular disorders) | 2 (2) | 1 (1) | 1 (1) | 3 (4)
Lymphocele (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Acute cardiac event (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial thrombosis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated myocarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 9 (11)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Immune-mediated nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Obstructive nephropathy (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary bladder polyp (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urogenital fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vesical fistula (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 4 (4)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acute monocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myelomonocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gallbladder adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ovarian Sertoli-Leydig cell tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Autoimmune hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertransaminasaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 5 (5)
Hypophysitis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Autoimmune thyroiditis (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune-mediated hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Primary hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Degenerative bone disease (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Soft tissue necrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cytokine release syndrome (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sarcoidosis (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dermatitis exfoliative generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pelvic haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal detachment (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Blindness (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileostomy closure (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Not Treated (N=79) | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib Pbo+Dostarlimab Pbo +/-Bev (Arm1) (N=159) | Paclitaxel + Carboplatin + Dostarlimab Pbo +/- Bev, Then Niraparib+Dostarlimab Pbo +/- Bev (Arm2) (N=417) | Paclitaxel + Carboplatin + Dostarlimab +/- Bev, Then Niraparib+Dostarlimab +/- Bev (Arm3) (N=745)
Nausea (Gastrointestinal disorders) | 15 (16) | 86 (150) | 251 (485) | 443 (1010)
Constipation (Gastrointestinal disorders) | 7 (7) | 70 (106) | 193 (339) | 365 (617)
Diarrhoea (Gastrointestinal disorders) | 11 (11) | 63 (94) | 148 (282) | 296 (560)
Abdominal pain (Gastrointestinal disorders) | 8 (8) | 47 (64) | 119 (184) | 262 (410)
Vomiting (Gastrointestinal disorders) | 11 (13) | 34 (52) | 132 (197) | 240 (419)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 12 (15) | 48 (66) | 103 (167)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 8 (14) | 45 (57) | 79 (90)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 11 (16) | 33 (39) | 76 (97)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 12 (16) | 37 (44) | 60 (74)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 5 (5) | 21 (27) | 71 (86)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 15 (16) | 24 (30) | 51 (54)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 10 (12) | 21 (29) | 29 (34)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 7 (8) | 21 (25) | 25 (34)
Fatigue (General disorders) | 6 (6) | 61 (98) | 151 (306) | 346 (673)
Asthenia (General disorders) | 8 (8) | 53 (126) | 158 (365) | 254 (671)
Pyrexia (General disorders) | 3 (3) | 11 (16) | 40 (51) | 119 (152)
Oedema peripheral (General disorders) | 1 (1) | 11 (17) | 40 (48) | 76 (95)
Mucosal inflammation (General disorders) | 1 (1) | 11 (14) | 37 (47) | 70 (104)
Pain (General disorders) | 3 (3) | 10 (13) | 28 (33) | 51 (67)
Anaemia (Blood and lymphatic system disorders) | 11 (18) | 70 (167) | 269 (914) | 485 (1755)
Neutropenia (Blood and lymphatic system disorders) | 5 (5) | 50 (115) | 156 (442) | 260 (764)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (4) | 22 (40) | 164 (477) | 263 (796)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 8 (9) | 29 (98) | 63 (157)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 76 (128) | 173 (322) | 312 (551)
Headache (Nervous system disorders) | 0 (0) | 42 (57) | 106 (182) | 199 (307)
Dizziness (Nervous system disorders) | 3 (3) | 16 (21) | 63 (93) | 125 (176)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 25 (45) | 59 (95) | 118 (193)
Dysgeusia (Nervous system disorders) | 0 (0) | 16 (18) | 34 (43) | 85 (104)
Paraesthesia (Nervous system disorders) | 2 (2) | 9 (15) | 40 (53) | 55 (74)
Neurotoxicity (Nervous system disorders) | 0 (0) | 9 (12) | 13 (28) | 25 (46)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4) | 66 (79) | 193 (258) | 328 (411)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 20 (30) | 48 (62) | 158 (313)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 12 (14) | 44 (72) | 138 (200)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 4 (4) | 30 (33) | 53 (57)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (13) | 17 (18) | 57 (84)
Platelet count decreased (Investigations) | 3 (3) | 25 (57) | 114 (349) | 229 (695)
Neutrophil count decreased (Investigations) | 3 (4) | 29 (56) | 82 (228) | 181 (499)
Alanine aminotransferase increased (Investigations) | 3 (7) | 12 (23) | 46 (102) | 122 (257)
Weight decreased (Investigations) | 2 (2) | 21 (29) | 49 (68) | 110 (178)
Aspartate aminotransferase increased (Investigations) | 2 (5) | 10 (17) | 49 (87) | 117 (254)
White blood cell count decreased (Investigations) | 6 (6) | 12 (25) | 37 (69) | 94 (284)
Blood creatinine increased (Investigations) | 3 (3) | 4 (5) | 38 (76) | 97 (216)
Amylase increased (Investigations) | 1 (2) | 7 (13) | 20 (33) | 60 (117)
Blood alkaline phosphatase increased (Investigations) | 1 (3) | 3 (3) | 10 (13) | 59 (137)
Blood thyroid stimulating hormone increased (Investigations) | 0 (0) | 9 (11) | 19 (24) | 36 (48)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 64 (132) | 155 (291) | 293 (527)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 30 (39) | 88 (151) | 163 (252)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 26 (34) | 59 (81) | 123 (163)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 19 (24) | 47 (71) | 82 (96)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (9) | 33 (44) | 47 (64)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 7 (9) | 25 (34) | 50 (69)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 10 (10) | 26 (32) | 43 (52)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 7 (7) | 22 (34) | 28 (34)
Decreased appetite (Metabolism and nutrition disorders) | 8 (8) | 31 (40) | 100 (140) | 233 (388)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (2) | 30 (46) | 91 (180) | 172 (313)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (6) | 16 (27) | 47 (73) | 109 (247)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4) | 10 (24) | 20 (49) | 61 (144)
Hyperglycaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (15) | 32 (49) | 51 (95)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 9 (11) | 24 (26) | 40 (49)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 7 (7) | 7 (14) | 11 (16) | 39 (104)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (2) | 9 (9) | 12 (21) | 19 (28)
Urinary tract infection (Infections and infestations) | 4 (4) | 27 (54) | 83 (140) | 143 (234)
COVID-19 (Infections and infestations) | 1 (1) | 5 (5) | 50 (55) | 96 (108)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 20 (24) | 87 (127) | 183 (275)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 21 (26) | 58 (64) | 121 (164)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 21 (26) | 60 (79) | 120 (166)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 20 (20) | 41 (45)
Hypertension (Vascular disorders) | 3 (3) | 41 (81) | 126 (262) | 236 (509)
Hot flush (Vascular disorders) | 0 (0) | 17 (22) | 46 (59) | 69 (78)
Insomnia (Psychiatric disorders) | 0 (0) | 25 (31) | 84 (106) | 143 (176)
Anxiety (Psychiatric disorders) | 2 (2) | 18 (21) | 45 (55) | 70 (83)
Depression (Psychiatric disorders) | 2 (3) | 9 (9) | 21 (26) | 40 (51)
Infusion related reaction (Injury, poisoning and procedural complications) | 3 (4) | 15 (24) | 40 (48) | 49 (61)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 21 (26) | 42 (47)
Proteinuria (Renal and urinary disorders) | 0 (0) | 10 (15) | 36 (78) | 60 (106)
Dysuria (Renal and urinary disorders) | 0 (0) | 9 (9) | 15 (19) | 27 (34)
Hypothyroidism (Endocrine disorders) | 0 (0) | 9 (10) | 27 (32) | 150 (189)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 5 (5) | 12 (15) | 42 (47)
Palpitations (Cardiac disorders) | 0 (0) | 6 (7) | 26 (37) | 52 (62)
Tachycardia (Cardiac disorders) | 1 (1) | 4 (6) | 15 (20) | 43 (60)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 0 (0) | 4 (4) | 9 (10)
Vision blurred (Eye disorders) | 1 (1) | 9 (10) | 12 (12) | 44 (47)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 6 (6) | 21 (32) | 20 (25)
Hypersensitivity (Immune system disorders) | 0 (0) | 11 (12) | 10 (13) | 18 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2025-08-08): https://cdn.clinicaltrials.gov/large-docs/59/NCT03602859/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-06): https://cdn.clinicaltrials.gov/large-docs/59/NCT03602859/SAP_001.pdf